## Statistical Analysis Plan

**Study ID: 213362** 

**Official Title of Study:** An Open-Label, Randomized-Sequence, Multicenter, Single-Crossover Study to Assess the Relative Bioavailability and Bioequivalence of Niraparib Tablet Formulation Compared to Niraparib Capsule Formulation in Patients With Advanced Solid Tumors

**NCT ID:** NCT03329001

Date of Document (version 7): 12-July-2023

Date of Document (version 6): 21-December-2021

# Statistical Analysis Plan

AN OPEN-LABEL, RANDOMIZED-SEQUENCE, MULTICENTER, SINGLE-CROSSOVER STUDY TO ASSESS THE RELATIVE BIOAVAILABILITY AND BIOEQUIVALENCE OF NIRAPARIB TABLET FORMULATION COMPARED TO NIRAPARIB CAPSULE FORMULATION IN PATIENTS WITH ADVANCED SOLID TUMORS

GSK/TESARO Protocol 213362/3000-01-004

Number:

Protocol Version: 6.0 (Amendment 5)

Compound Number: GSK 3985771, MK-4827

Study Drug Name: Niraparib

Phase: Phase 1

Methodology: Open-Label, Cross-Over

Sponsor: TESARO, GSK Company

Analysis Plan Date: 12 July 2023

Analysis Plan Version: Version 7.0

#### **Confidentiality Statement**

All information contained in this document is privileged and confidential to TESARO, a wholly owned subsidiary of GSK. Any distribution, copying, or disclosure is strictly prohibited without prior written approval by TESARO.

#### SPONSOR SIGNATURE PAGE

Protocol Title: AN OPEN-LABEL, RANDOMIZED-SEQUENCE,

MULTICENTER, SINGLE-CROSSOVER STUDY TO ASSESS THE RELATIVE BIOAVAILABILITY AND

BIOEQUIVALENCE OF NIRAPARIB TABLET

FORMULATION COMPARED TO NIRAPARIB CAPSULE FORMULATION IN PATIENTS WITH ADVANCED SOLID

Protocol No: 3000-01-004

**TUMORS** 

Protocol Number: 3000-01-004

Sponsor: TESARO, a GSK Company

980 Great West Road

Brentford

Middlesex, TW8 9GS

UK

By signing this document, I acknowledge that I have read the document and approve of the planned statistical analyses described herein. I agree that the planned statistical analyses are appropriate for this study, are in accordance with the study objectives, and are consistent with the statistical methodology described in the protocol, clinical development plan, and all applicable regulatory guidance and guidelines.

| Author: Alina Striha Principal Statistician Plus-Project Ltd. | Signature: |
|---------------------------------------------------------------|------------|
| | Date: |
| Approver: Wenlei Liu Statistics Director GSK Company | Signature: |
| | Date: |

# TABLE OF CONTENTS

| SPONSO | OR SIGNATURE PAGE | 2 |
|---------|------------------------------------------------------|----|
| TABLE | OF CONTENTS | 3 |
| TABLE | S INCLUDED IN THE TEXT | 5 |
| FIGURE | ES INCLUDED IN THE TEXT | 5 |
| LIST OF | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 6 |
| 1. Info | formation from the Study Protocol | 8 |
| 1.1. | Introduction and Objectives | 8 |
| 1.1 | .1. Introduction | 8 |
| 1.1 | .2. Study Objectives | 8 |
| 1.1 | .3. Scope and Revision History | 9 |
| 1.2. | Study Design | 14 |
| 1.2 | .1. Synopsis of Study Design | 14 |
| 1.2 | .2. Randomization Methodology | 18 |
| 1.2 | .3. Unblinding | 18 |
| 1.2 | .4. Study Procedures | 18 |
| 1.2 | .5. Efficacy, Safety, and Pharmacokinetic parameters | 18 |
| 2. Pat | ient Population | 19 |
| 2.1. | Population Definitions | 19 |
| 2.2. | Protocol Deviations | 19 |
| 3. Gei | neral Statistical Methods | 19 |
| 3.1. | Sample Size Justification | 19 |
| 3.2. | General Methods | 21 |
| 3.3. | Baseline Definitions | 22 |
| 3.4. | Methods of Pooling Data | 22 |
| 3.5. | Adjustments for Covariates | 22 |
| 3.6. | Multiplicity Adjustment | 22 |
| 3.7. | Subpopulations | 22 |
| 3.8. | Withdrawals, Drop-outs, Loss to Follow-up | 22 |
| 3.9. | Missing Data | 22 |
| 3.10. | Visit Windows | 23 |
| 3.11. | Interim Analysis | 23 |
| 3.12. | COVID-19 | 23 |

| 4. | Stu | dy Analyses | 24 |
|----|------|------------------------------------------------------------|----|
| | 4.1. | Patient Disposition | 24 |
| | 4.2. | Demographics, Baseline Characteristics and Medical History | 24 |
| | 4.3. | Investigator Assessment of Response | 25 |
| | 4.4. | Safety Evaluation | 25 |
| | 4.4. | .1. Treatment Exposure and Compliance | 25 |
| | 4.4. | .2. Adverse Events | 26 |
| | 4.4. | .3. Laboratory Data | 29 |
| | 4.4. | .4. Vital Signs and Physical Examination | 29 |
| | 4.4. | .5. Electrocardiogram | 30 |
| | 4.4. | .6. Prior and Concomitant Mediations | 30 |
| | 4.4. | .7. Prior and Concomitant Transfusions and Growth Factors | 31 |
| | 4.4. | .8. COVID-19 | 31 |
| 5. | Cha | anges to Planned Analyses | 31 |
| | 4.5. | Changes in v5.0 of the SAP | 31 |
| | 4.6. | Changes in v6.0 of the SAP | 32 |
| | 4.7. | Changes in v7.0 of the SAP | 32 |
| 6. | App | pendix | 33 |
| | 6.1. | Planned Statistical Tables, Listings, and Figures | |

| TABLES INCLUDED IN THE TEXT | |
|---|---|
| TABLE 1 REVISION HISTORY | 13 |
| TABLE 2 NCI COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS V4.03 (CTCAE) | 29 |
| FIGURES INCLUDED IN THE TEXT | |

Statistical Analysis Plan


Niraparib

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|---|---|
| AE(s) | adverse event(s) |
| AESI | Adverse Events of Special Interest |
| ALT | alanine aminotransferase |
| ALP | alkaline phosphatase |
| AML | Acute Myeloid Leukemia |
| AST | aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| AUC | area under the plasma concentration-time curve |
| BA | bioavailability |
| BE | bioequivalence |
| BMI | body mass index |
| CI | confidence interval |
| CL/F | apparent total body clearance |
| C <sub>max</sub> | Maximum observed plasma concentration |
| CSR | clinical study report |
| CV | coefficient of variation |
| ECG | electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic case report form |
| ЕОТ | end-of-treatment |
| FE | food effect |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| LLN | lower limit of normal |
| LS mean | least-squares mean |
| CCI | |
| MDRP | Medical Data Review Plan |
| MDS | Myelodysplastic Syndromes |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCI CTCAE | National Cancer Institute Common Terminology Criteria for Adverse Events |
| PI | Package Insert |
| PK | pharmacokinetics |
| PT | preferred term |

| Abbreviation | Definition |
|------------------|------------------------------------------|
| $Q_1$ | first quartile |
| Q <sub>3</sub> | third quartile |
| QD | one time per day |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SOC | system organ class |
| t <sub>1/2</sub> | termination elimination half-life |
| TEAE | treatment-emergent adverse event |
| t <sub>max</sub> | Time to reach C <sub>max</sub> |
| US | United States |
| ULN | upper limit of normal |
| Vz/F | apparent terminal volume of distribution |
| WHO | World Health Organization |

## 1. Information from the Study Protocol

#### 1.1. Introduction and Objectives

#### 1.1.1. Introduction

The approved niraparib drug product is an immediate release hard gelatin capsule dosage form that contains 100 mg of niraparib per capsule. The labelled starting dose for niraparib is 300 mg. Facilitating this dose requires the administration of three 100 mg capsules.

It is the Sponsor's intent to introduce a tablet dosage form that provides the 100 mg, 200 mg and 300 mg dose in single dose strength tablets to reduce the pill burden on the patients.

To this end, the Sponsor has developed a tablet dosage form with the specific intent to provide comparable performance to the approved capsule dosage form. The formulation and manufacturing process of the tablet were selected to produce a tablet with comparable in-vitro performance to the capsule.

This study is an open-label Phase 1 study to evaluate the relative bioavailability (BA) and bioequivalence (BE) of niraparib administered as a tablet formulation compared to the reference capsule formulation manufactured by the same process as currently marketed in the United States. Specifically, a 300 mg niraparib tablet will be compared to three (3) niraparib capsules (3 × 100 mg). In addition, this study will evaluate the effect of a high-fat meal on the pharmacokinetics (PK) of the niraparib 300 mg tablet formulation (Stage 3). The Extension Phase of this study is to enable patients enrolled in the study to continue to receive treatment with niraparib if they are tolerating it and, in the Investigator's opinion, may receive benefit.

#### 1.1.2. Study Objectives

The primary objectives of this study are as follows:

- Stage 1: To obtain preliminary assessment of the relative bioavailability of 300 mg niraparib administered as a tablet versus capsule formulation and to estimate the intra-subject variability of niraparib PK
- Stage 2: To evaluate if the tablet formulation ( $1 \times 300 \text{ mg}$ ) of niraparib is bioequivalent to the capsule formulation ( $3 \times 100 \text{ mg}$ )
- Stage 3: To assess the effect of a high-fat meal on niraparib PK following a single 300 mg dose of the tablet formulation.

The secondary objectives of this study are as follows:

- Stage 1, Stage 2, and Stage 3: To evaluate the safety of single dose niraparib when administered as a tablet or capsule formulation in patients with advanced solid tumors
- Extension Phase: To evaluate the safety of continuously dosed niraparib in patients with advanced solid tumors.

The exploratory objectives of this study are as follows:

CCI

#### 1.1.3. Scope and Revision History

A separate PK analysis plan will be written to address the PK objectives and data for this study.

This statistical analysis plan (SAP) is designed to outline the methods to be used in the analyses of non-pharmacokinetic study data. Patient populations to be used for analyses, data handling rules, statistical methods, and formats for data presentation are identified and provided. The statistical analyses and summary tabulations described in this SAP will provide the basis for the results sections of the clinical study report (CSR) for this trial.

The SAP will outline any differences in the currently planned analytical objectives relative to those planned in the study protocol.

The SAP is a living document that will be created during the trial conduct. It will be maintained throughout the lifecycle of the trial. Important changes following approval of SAP v1.0 will be tracked in this section.

The following changes have been implemented in the Appendix containing shells of the Planned Statistical Tables, Listings and Figures.

| Table/Listing | | |
|---|---|---|
| Number | Correction | Reason for Correction |
| Table 14.1.1d | Footnotes [2] and [3] added to the table and in the footer. | Clarification why two patients have been double counted in Screening. |
| Table 14.1.3.1c | Footnote added to the shell. | Clarification added to the output for Extension Phase reporting effort. |
| Table 14.1.4d | Added "Missing" category to Cancer stage and Number of prior lines of therapy. | Data collected has missing information on the eCRF. |
| Table 14.3.1.1.2d | Removed "Any COVID-19 related TEAE". | Removing a duplicate entry row. |
| Table 14.3.1.14d | Removed "System Organ Class" from the table. | Line not required for the table in question as summary by Preferred Term is of interest. |
| Table 14.3.1.16.1c | Table shell added. | Table added for final study disclosure purposes of Extension Phase data. |
| Table 14.3.1.16d | Added footnote: "NOTE: Deaths due to progressive disease were not collected as adverse events." | Added to reflect data collection and management process and align with Stage 1 and Stage 2 programming practice. |
| Table 14.3.1.2.1.1d | Note: COVID-19 Case Diagnosis is based on WHO Definition as of DDMMMYYYY. | |
| Table 14.3.1.20d<br>Table 14.3.1.21d<br>Table 14.3.1.22d | Footnote [1] updated to: "Note: Extension Phase for all Stages of TABLET study overlapped with COVID-19 pandemic, with all Stage 3 patients commencing treatment for the Extension Phase on or after 02JUN2021 placing the AE onset during the pandemic, while last patient commenced treatment for Stages 1 and 2 on 14MAY2018 and 05DEC2019, respectively, placing their first Extension Phase treatment dose administration prior to the start of the pandemic, as defined by WHO as of 20MAR2020, with | Clarification of footnote explaining calendar placement of the Stages 1-3 during COVID-19 pandemic. |

| Table/Listing | | |
|---|---|---|
| Number | Correction | Reason for Correction |
| | patients across all Stages ongoing until DDMMMYYYY." | |
| | Table titles updated to: Table 14.3.1.20d Summary of Incidence of COVID-19 Related Adverse Events Over Time (Safety Population in the Stage 3 PK Phase) Table 14.3.1.21d Summary of Incidence of COVID-19 Related Adverse Events Over Time by Gender (Safety Population in the Stage 3 PK Phase) Table 14.3.1.22d Summary of Incidence of COVID-19 Related Adverse Events Over Time by Age Group (Safety Population in the Stage 3 PK Phase) | Clarification of titles to reflect the reporting effort of COVID-19 related AE incidence rates. |
| Table 14.4.1c | Summary table of Important Protocol Deviations for Open-Label Extension Phase added. | Added upon request from study team for CSR reporting purposes. |
| Table 14.4.1d | Summary table of Important Protocol Deviations for the PK Phase Occurring Through End of Treatment (Safety Population in the Stage 3 PK Phase). | Added upon request from study team for CSR reporting purposes. |
| | Footnotes and corresponding references added to the table. | Added upon request for clarification. |
| Listing 16.2.2.2c | Footnote [1] updated to: "Note: Extension Phase for all Stages of TABLET study overlapped with COVID-19 pandemic, with all Stage 3 patients commencing treatment for the Extension Phase on or after 02JUN2021 placing the AE onset during the pandemic, while last patient commenced treatment for Stages 1 and 2 on 14MAY2018 and 05DEC2019, respectively, placing their first Extension Phase treatment dose administration prior to the start of the pandemic, as defined by WHO as of 20MAR2020, with patients across all Stages ongoing until DDMMMYYYY. Added "PK Dose 1" and "PK Dose 2" date | Clarification of footnote explaining calendar placement of the Stages 1-3 during COVID-19 pandemic. Added columns to the shells to align |
| Listing 16.2.5.1d | columns to the listing. | Stage 3 reported outputs with those reported in Stages 1 and 2. |
| Listing 16.2.5.3d | Moved "Patient Number" into header row. Added "Rel Day [1]" column and [1] footnote: "[1] Relative to first dose during the PK Phase." For readability purposes. Added to the shells to align Stag reported outputs with those repo in Stages 1 and 2. | |
| Listing 16.2.5.5d | Columns "Full Dose Taken?", "If N, how much consumed?", "Reason for Change", "Nausea within specified time of dose?" removed from the listing. | Columns removed from Stage 3 listing as not applicable, as per study design. |
| Listing 16.2.8.1.1d Programming note added regarding location of and associated "Patient Number" in the outputs. | | Depending on spacing/information<br>displayed, "Patient Number" may be<br>displayed in the header row after |

| Table/Listing | | |
|---|---|---|
| Number Correction | | Reason for Correction |
| | | "Treatment Sequence" in order to aid |
| | | readability of the listing. |
| Listing 16.2.8.2d | Removed "Heart Rate" column. | Data collected under "Pulse" in |
| | | Stage 3, added "Heart Rate" to the |
| | | shells in error. |
| Listing 16.2.8.5d | Added text to footnote: "in the PK Phase" | Previously missing in error. |
| Listing 16.2.9.2c | Footnote [1] updated to: | Clarification of footnote explaining |
| | "Note: Extension Phase for all Stages of TABLET | calendar placement of the Stages 1-3 |
| | study overlapped with COVID-19 pandemic, with | during COVID-19 pandemic. |
| | all Stage 3 patients commencing treatment for the | |
| | Extension Phase on or after 02JUN2021 placing | |
| | the AE onset during the pandemic, while last | |
| | patient commenced treatment for Stages 1 and 2 | |
| | on 14MAY2018 and 05DEC2019, respectively, | |
| | placing their first Extension Phase treatment dose administration prior to the start of the pandemic, | |
| | as defined by WHO as of 20MAR2020, with | |
| | patients across all Stages ongoing until | |
| | DDMMMYYYY. | |
| Listing 16.2.2c | Listing updated to include only "Important" | Updated upon request from study |
| C | protocol deviations; title updated to reflect | team for CSR reporting purposes. |
| | change. | |
| | "Protocol Deviation Severity" column dropped. | Obsolete field. |
| Listing 16.2.2.1d | Listing updated to include only "Important" | Updated upon request from study |
| | protocol deviations; title updated to reflect | team for CSR reporting purposes. |
| Section 1.2 | change. Definition of data cut has been amended. | D.C. 22 1 14 Cl. 4 4 1 |
| Section 1.2 | Definition of data cut has been amended. | Definition changed to reflect study reporting requirements upon request |
| | | from study team. |
| Table 14.1.1c | Table has been updated to include Starting Dose | Updated upon request from study |
| 1 4 6 7 1 1 1 1 1 2 | (100 mg, 200 mg and 300 mg) and categorization | team for CSR reporting purposes. |
| | by Stage (TABLET Stages 1, 2 and 3). | |
| Table 14.1.10c | Table added for Extension Phase. | Added upon request from study team |
| | | for CSR reporting purposes. |
| Extension Phase | Treatment arm labels updated to be TABLET, | Updated for consistency. |
| tables | CAPSULE and OVERALL, for consistency, | |
| | throughout the shells | |
| Table 14.3.1.1.1c | Table shell spelled out for Extension Phase | Updated upon request from study |
| | reporting effort, including COVID-19 summary | team for CSR reporting purposes. |
| т.1.1. | categories. | A 11-1 |
| Table | New repeat table added for Extension Phase. | Added upon request from study team for CSR reporting purposes. |
| 14.3.1.1.1c<br>Table 14.3.1.11.1a | New table added for DV Ct 1 | Required for plain text summary |
| 14.3.1.11.18 | New table added for PK Stage 1. | reporting effort. |
| Table 14.3.1.11.1b | | |
| 10010 17.3.1.111.10 | reporting effort. | |
| Table 14.3.1.11.1c | New table added for Extension Phase. | Required for plain text summary |
| | The state added to Enterior Financial | reporting effort. |
| Table 14.3.1.11.1d | | |
| | | reporting effort. |
| Table 14.3.1.23.1a | New table added for PK Stage 1. | Required for disclosure reporting |
| | | effort. |

| Table/Listing | | |
|---|---|---|
| Number Correction | | Reason for Correction |
| Table 14.3.1.23.1b | New table added for PK Stage 2. | Required for disclosure reporting effort. |
| Table 14.3.1.23.1c | New table added for Extension Phase. | Required for disclosure reporting effort. |
| Table 14.3.1.23.1d | New table added for PK Stage 3. | Required for disclosure reporting effort. |
| Table 14.3.1.23.2a | New table added for PK Stage 1. | Required for plain text summary reporting effort. |
| Table 14.3.1.23.2b | New table added for PK Stage 2. | Required for plain text summary reporting effort. |
| Table 14.3.1.23.2c | New table added for Extension. | Required for plain text summary reporting effort. |
| Table 14.3.1.23.2d | New table added for PK Stage 3. | Required for plain text summary reporting effort. |
| Table 14.3.1.14c | Footnotes omitted as not applicable for Extension phase reporting. | Updated for clarification. |
| Table 14.3.1.20c | Footnote updated to reflect reporting period for overall study population in Extension Phase. | Updated for clarification. |
| Table 14.3.1.21c | Table added for Extension Phase reporting. | Updated upon request from study team for CSR reporting purposes. |
| Table 14.3.1.22c Table added for Extension Phase reporting. | | Updated upon request from study team for CSR reporting purposes. |
| Table 14.3.4.1c 'Number of Cycles' changed to 'Maximum number of cycles'. Labels for dose interruptions/reductions/re-escalations modified for clarity. 'Median number of cycles started', 'Exposure duration (months)' and 'Dose intensity' added to output. | | Updated to reflect changes requested by study team. |
| Table 14.3.4.5.1c Table added for Extension Phase reporting. | | Updated upon request from study team for CSR reporting purposes. |
| Listing 16.2.2.2c Listing added for Extension Phase reporting. | | Updated upon request from study team for CSR reporting purposes. |
| Listing 16.2.5.1.1c Listing added for Extension Phase reporting. | | Updated upon request from study team for CSR reporting purposes. |
| Listing 16.2.5.5c | "Tablets remaining" and "Was Full Dose Taken?" column dropped. | Data not collected consistently for study reporting purposes. |
| Listing 16.2.6.1c "Visit" column dropped. "Tumor Type" column added. | | Visit data not collected, only date of assessment. Added upon request from study team for CSR reporting purposes. |
| Listing 16.2.7.1c Listing shell spelled out for Extension Phase reporting effort. 'Dose at onset of AE' variable dropped from listing. | | Updated upon request from study team for CSR reporting purposes. Data not collected consistently for production of reliable results. |
| Listing 16.2.7.2c | Listing added for Extension Phase reporting. | Added upon request from study team for CSR reporting purposes |
| Listing 16.2.9.2c | | |
| Figure 14.3.4.3.1c Figure shell added for Extension Phase reporting effort. | | Updated upon request from study team for CSR reporting purposes. |

Table 1 Revision History

| SAP<br>version | Protocol version | eCRF<br>version | Changes from previous version |
|---|---|---|---|
| 1.0 | 2.0 | 5.0 (26FEB2018) | First Draft |
| 2.0 | 4.0 | 8.0 (12FEB2019) | Major changes to this draft of the SAP include the following: |
| | | | Incorporate changes based on amended protocol. |
| | | | Modify Stage 2 analysis of AEs to accommodate the increase in washout time between Period 1 and Period 2 for Stage 2. |
| | | | For the Extension Phase, specify that analysis will be performed by formulation and overall to accommodate allowance of both tablet and capsule formulation in the Extension Phase. |
| | | | Define the BA/BE evaluable population and add demographic and baseline characteristic summaries for this population. |
| | | | Clarify definition of concomitant medications and add additional table for Stage 2 to analyze only medications taken during the PK collection period. |
| | | | Clarifications to mock table and listing shells (e.g., numbering, footnotes). |
| 3.0 | 5.0 | 10.0 (31JUL2019) | Major changes to this draft of the SAP include the following: |
| | | | <ul> <li>Incorporate changes based on amended protocol, including:</li> </ul> |
| | | | <ul> <li>Updated numbers of patients enrolled to account<br/>for non-evaluability.</li> </ul> |
| | | | <ul> <li>Specification of reasons for non-evaluability for<br/>the analysis of bioequivalence.</li> </ul> |
| | | | <ul> <li>Focus Extension Phase laboratory summaries on select<br/>laboratory assessments hemoglobin, neutrophils, platelets,<br/>bilirubin, creatinine, AST, and ALT).</li> </ul> |
| 4.0 | 6.0 | 11.0 (16APR2020) | Major changes to this draft of the SAP include the following: |
| | | | <ul> <li>Incorporate changes based on amended protocol, to<br/>address the objectives for Stage 3 of the study.</li> </ul> |
| | | | Addition of sections relating to COVID-19 reporting. |
| 5.0 | 6.0 | 13.0 (17MAR2021) | Primary changes to this draft associated with addition of Important Protocol Deviation table and updates to the associated listing to reporting effort. |
| | | | Minor updates to align Stage 1, 2 and 3 TLFs with shells, and associated update to Protocol Deviation reporting, as per the SAP. |

| SAP<br>version | Protocol version | eCRF<br>version | Changes from previous version |
|---|---|---|---|
| 6.0 | 6.0 | 13.0 (17MAR2021) | Primary change to this draft of the SAP is change of the data cut for reporting of final Stage 3 analysis. |
| | | | Minor update to footnotes of Important Protocol Deviation summary table. |
| | | | Minor update to Section 5 formatting. |
| 7.0 | 6.0 | 14.0 (17NOV2021) | Minor updates to template output/column header and title formatting to align with produced output header and title formatting. |
| | | | CRF versions updated to align with CRF booklet version upgrades starting from SAP version 4.0 onwards. |
| | | | COVID-19 related output shell added for Extension phase. |
| | | | Definitions of exposure and compliance derivations expanded to include dose intensity. |
| | | | Additional tables and listings have been added/modified for Extension Phase; disclosure and plain language summary reporting tables have been added across all study stages. |
| | | | Section 3.2 'Dose at onset of AE' has been removed from AE listings; output shells added for adverse event reporting in the Extension Phase/to cover time between end of PK Phase and start of Extension Phase. |
| | | | Section 2 updated to include definition for dose intensity in exposure table for Extension Phase. |
| | | | Section 4.4.2 updated AE classification for PK Period 1 for Stage 3. |

#### 1.2. Study Design

#### 1.2.1. Synopsis of Study Design

This is a multicenter, open-label study in patients with advanced solid tumors. This is a 3-stage, randomized-sequence, single-crossover study to assess the relative BA and BE of niraparib tablet formulation relative to the capsule formulation. In addition, Stage 3 of the protocol is a single cohort, randomized-sequence, 2 period, single dose, crossover study to assess effect of food on the PK of the niraparib tablet formulation.

Pharmacokinetics (PK) Phase: In Stages 1 and 2, patients will be randomized 1:1 to receive tablet formulation followed by capsule formulation or capsule formulation followed by tablet formulation. In Stage 3, patients will be randomized 1:1 to receive tablet formulation in a fasted state followed by tablet taken with a high-fat meal, or by tablet taken with a high-fat meal followed by tablet formulation taken in a fasted state.

Stage 1: Following an 8-hour fast on Day 1, patients will receive a single dose of the formulation (tablet  $[1 \times 300 \text{ mg}]$  or capsule  $[3 \times 100 \text{ mg}]$ ) followed by a 7-day (+1 day) Washout/PK period, followed by a dose of the alternate formulation also in a fasted state, followed by a 7-day (+1 day) Washout/PK period for Stage 1 of the study followed by a dose of the alternate formulation also in a fasted state, followed by a 7-day Washout/PK period. Patients receiving the tablet in the first treatment period will receive the capsules in the second treatment period and vice versa (Figure 1). Extensive PK sampling will be carried out after niraparib dosing.

Stage 2: Following an 8-hour fast on Day 1, patients will receive a single dose of the formulation (tablet  $[1 \times 300 \text{ mg}]$  or capsule  $[3 \times 100 \text{ mg}]$ ) followed by a 14-day (+/- 4 days) Washout/PK period followed by a dose of the alternate formulation also in a fasted state, followed by a 7-day Washout/PK period. Patients receiving the tablet in the first treatment period will receive the capsules in the second treatment period and vice versa (Figure 1). Extensive PK sampling will be carried out after niraparib dosing.

Stage 3: In Period 1, patients will receive a single 300 mg niraparib tablet either following a 10-hour fast or directly following consumption of a high-fat meal, followed by a 14-day (+4 days) PK sampling and Washout period. In Period 2, patients will be crossed over to receive a single 300 mg niraparib tablet in a fasted state or with a high-fat meal, followed by a 7-day PK sampling period. All patients will fast for a minimum of 4 hours post-dose in both periods. Patients receiving the tablet in the fasted state in the first treatment period will receive the tablet with a high-fat meal in the second treatment period and vice versa.

In the rare instance where a delay of the entire PK Period 2 is needed for any reason beyond the 4 day window specified above the site must contact the Sponsor's medical monitor to discuss the patient circumstances, the Sponsor will decide if the patient can continue with PK Period 2 with a delay. Similarly, should the laboratory results on Day 15 (D15) (the day of niraparib administration in PK Period 2) show changes in organ function such that the original inclusion criteria for laboratory values are no longer met, or in the event of a significant change of patient's clinical status as judged by the Investigator, the site must consult with the Sponsor to discuss the patient's continued participation in PK Period 2. Note that sites need not wait for the pre-dose laboratory results to begin PK Period 2, but rather consult the Sponsor once the results are available as needed. In Stage 2, patients who experience emesis within 9 hours of dosing or who miss a critical PK sample (such as the last PK sample on Day 8 in each period) will be discontinued from the PK Phase and will be allowed to be screened for the Extension Phase. In Stage 3, patients who experience emesis within 10 hours of dosing will be discontinued from the PK Phase and will be allowed to be screened for the Extension Phase. Patients who miss sufficient samples to render calculation of AUC unreliable will be discontinued from the PK Phase; those that meet other criteria for continued niraparib therapy will be eligible to be screened for the Extension Phase.

For Stage 1, the PK parameters that will be estimated include area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration ( $AUC_{0-t}$ ), area under the plasma concentration-time curve from time 0 extrapolated to infinity ( $AUC_{0-\infty}$ ), apparent total body clearance (CL/F), maximum observed plasma concentration ( $C_{max}$ ), time to reach  $C_{max}$  ( $t_{max}$ ), termination elimination half-life ( $t_{1/2}$ ), apparent terminal volume of distribution (Vz/F) and BA of tablet formulation relative to the capsule formulation based on  $AUC_{0-t}$ ,  $AUC_{0-\infty}$ , and  $C_{max}$ . Relative bioavailability will be assessed based on the ratio of geometric least-squares (LS) means of the test (tablet) to reference

(capsule). Additionally, the pharmacokinetics of **CC** will be determined (Stage 1 only).

For Stage 2, the same PK parameters as above will be estimated. To conclude bioequivalence, the 90% confidence interval (CI) of the ratio of geometric LS means of the test (tablet) to reference (capsule) product should be within 0.800 - 1.250 (80% - 125%) for  $AUC_{0-x}$ ,  $AUC_{0-t}$ , and  $C_{max}$ .

For Stage 3, the same PK parameters as above will be estimated. In addition,  $t_{lag}$ , the time from administration of the dose to the first quantifiable concentration, will be determined, and  $t_{max}$  will be compared between the fed and fasted states. The relative bioavailability of the 300 mg niraparib tablet administered with a high-fat meal relative to fasted dosing will be based on the ratio of geometric LS means of  $AUC_{0-t}$ ,  $AUC_{0-\infty}$ , and  $C_{max}$ .

Additional PK parameters may be estimated (e.g., residual area), if deemed appropriate.

Extension Phase: When patients complete the PK Phase of the study (at least 7-days from the beginning of PK Period 2), they may be eligible to participate in the Extension Phase following review of the Extension Phase inclusion criteria and completion of the required Extension Phase screening assessments. The starting dose of niraparib in the Extension Phase will be based on the patient's baseline actual body weight or platelet count. Patients with a baseline actual body weight of >77 kg and screening platelet count of ≥150,000/μL (obtained after completion of the PK Phase, as part of Extension Phase screening) will take one 300 mg strength tablet or 3 × 100 mg tablet/capsules at each dose administration (once a day [QD]). Patients with a baseline actual body weight of <77 kg or screening platelet count of <150,000/μL will take one 200 mg strength tablet or  $2 \times 100$  mg tablet/capsules at each dose administration (QD). For patients whose initial starting dose is 200 mg QD, escalation to 300 mg QD is permitted after 2 cycles of therapy if no treatment interruption or discontinuation was required during the first 2 cycles of Extension Phase therapy and after approval from the Sponsor. Additional dose modifications will not be based upon changes in the patient's actual body weight during study participation. If laboratory values at the beginning of Extension Phase are outside of the range specified in the inclusion criteria, the patient may continue to participate in the study only upon Sponsor approval with consideration for an appropriately reduced dose. Should a patient start the Extension Phase at 100 mg, consideration may be given to escalate to 200 mg after 2 cycles of therapy if no treatment interruption or discontinuation was required during the first 2 cycles of Extension Phase therapy and after approval from the Sponsor.

Patients have up to 28 days (21 days for Stage 3 only; up to 28 days may be acceptable following discussion between the Sponsor and Investigator) after completion of the PK Phase to complete the screening assessments and the Extension Phase Screening Visit.

A tumor assessment is to be performed prior to the first dose of the Extension Phase (pre-Extension Phase). The pre-Extension Phase tumor assessment need not be completed if the baseline tumor assessment was performed  $\leq$  56 days before the first dose of the Extension Phase.

The Cycle 1/Day 1 Visit can occur on the same day as the Extension Phase Screening Visit, dependent upon availability of radiographic results obtained  $\leq$  56 days of the first planned dose in the Extension Phase. If the Extension Phase Screening Visit and the Cycle 1/Day 1 Visit occur on the same day, the clinical laboratory results will be reviewed by the study personnel prior to study drug administration to

ensure eligibility. At the Cycle 1/Day 1 Visit, patients will undergo safety assessments and will receive study drug supply for the duration of 1 cycle (300 mg or 200 mg tablets of niraparib for QD dosing or 3 × 100 mg or 2 × 100 mg tablet/capsules of niraparib for QD dosing, depending on availability). It is preferred that patients remain on the same formulation (tablet versus capsule) throughout the Extension Phase. Patients will return on the first day of every treatment cycle (28 ± 7 days) to receive study drug and for safety assessments. Visits will continue approximately every 4 weeks until treatment discontinuation. In line with the niraparib United States Package Insert (US PI), dose interruption (no longer than 28 days) will be allowed based on adverse events (AEs). In addition, dose reductions to 200 mg QD and subsequently to 100 mg QD will be allowed based on AEs (please refer to US PI). Any dose reductions differing from this must be discussed with the medical monitor. Patients can continue in the Extension Phase until the patient meets 1 of the withdrawal criteria.

End-of-treatment (EOT) and Safety Follow-up Visits: The EOT visit will occur within 7 days of the decision to discontinue study drug, for any reason, or completion of the PK Phase for patients who participate in the Extension Phase (Stage 3 only), whichever occurs first. Should the first dose of a new anti-cancer therapy occur within 14 days of the decision to discontinue study drug, all assessments required for the Safety Follow-up visit should occur at the EOT visit and this visit will be considered the Safety Follow-up visit. If the first dose of the new anti-cancer therapy occurs >14 days of the decision to discontinue study, the Safety Follow-up visit will occur 30 +7 days after the last dose of the study drug, or at the start of any new anti-cancer therapy, whichever occur first.

For Stage 3 of the PK Phase only, the data cut will occur when all patients have completed the PK Phase. Data collected up to and including PK EOT visit prior to the data cut will be presented in the FE Stage 3 PK CSR for all randomized and treated patients. Additionally, the Sponsor will include safety data related to the PK Phase, as identified up to Cycle 1/Day 1 of the Extension Phase.





Abbreviations: PK = pharmacokinetics.

#### 1.2.2. Randomization Methodology

Randomization will occur centrally using an interactive voice response system/integrated web response system. In Stage 1 and Stage 2, patients will be assigned randomly in a 1:1 ratio to a dosing sequence: capsule formulation followed by tablet formulation, or vice versa. In Stage 3, patients will be assigned randomly in a 1:1 ratio to a dosing sequence: dosing after receiving a high-fat meal (fed) followed by dosing after fasting, or vice versa. The period between randomization and Cycle 1/Day 1 should be no longer than 5 calendar days.

#### 1.2.3. Unblinding

Unblinding is not applicable as this is an open-label study.

#### 1.2.4. Study Procedures

Refer to the latest protocol for the schedule of assessments.

#### 1.2.5. Efficacy, Safety, and Pharmacokinetic parameters

#### 1.2.5.1. Efficacy parameters

Investigator assessment of response will occur every 3-cycles while on study or per the Institution's standard practice.

#### 1.2.5.2. Safety parameters

Safety parameters to be assessed include:

- Treatment emergent adverse events (TEAE)
- Discontinuations due to AEs
- Physical examination (PE) findings
- Vital signs
- Clinical laboratory results (hematology, chemistry, urinalysis)
- Electrocardiograms (ECG)
- Use of concomitant medications.

#### 1.2.5.3. PK parameters

PK parameters and analysis methodology will be addressed in the PK analysis plan.

## 2. Patient Population

#### 2.1. Population Definitions

The following patient populations will be evaluated for analyses specified in this SAP. Additional populations, relevant to the PK analysis will be defined in the PK analysis plan.

- Safety Population in the Stage 1 PK Phase: All patients who receive any amount of niraparib during the Stage 1 PK Phase of the study.
- Safety Population in the Stage 2 PK Phase: All patients who receive any amount of niraparib during the Stage 2 PK Phase of the study.
- Safety Population in the Stage 3 PK Phase: All patients who receive any amount of niraparib during the Stage 3 PK Phase of the study.
- Safety Population in the Extension Phase: All patients who receive any amount of niraparib in the Open-Label Extension Phase of the study.
- BA/BE Evaluable Population: All patients who complete both PK periods and have sufficient PK sample collection to accurately estimate PK parameters, without significant niraparib carryover (baseline concentration > 5% of  $C_{max}$ ), in both PK Periods. Patients who have significant niraparib carryover from Period 1 in Period 2 will be completely excluded from the BA/BE Evaluable Population. The terminology BA Evaluable Population will be used for Stage 1 and BE Evaluable Population will be used for Stage 2.
- Food effect (FE) Evaluable Population: All patients who complete both PK periods and have sufficient PK sample collection to accurately estimate PK parameters in both periods. Patients meeting non-evaluability criteria or having significant niraparib carryover (baseline concentration >5% of C<sub>max</sub>) will be completely excluded from the FE Population.

#### 2.2. Protocol Deviations

Protocol deviations will be assessed and classified as important and/or significant per Sponsor's SOP. The Medical Data Review Plan (MDRP) prospectively identifies classification criteria for important deviations. All protocol deviations will be identified, classified and finalized prior to database lock.

A listing of protocol deviations will be provided for the Stage 1 PK Phase, Stage 2 PK Phase; for Stage 3 PK Phase and the Open-Label Extension Phase a listing of only "Important" protocol deviations will be provided.

For Stage 3 PK Phase and Open-Label Extension Phase, tables summarizing "Important" protocol deviations will be provided.

#### 3. General Statistical Methods

# 3.1. Sample Size Justification Stage 1

No formal sample size calculation was performed for Stage 1. Approximately 24 patients will be enrolled in Stage 1. This sample size is considered adequate for preliminary assessment of the relative bioavailability of the tablet compared to the capsules and for estimating the intra-subject coefficient of variation, after accounting for patient drop-outs and potential carryover.

#### Stage 2

Based on estimates from Stage 1, 100 BA/BE evaluable patients are required in Stage 2. With 100 evaluable patients, assuming the intra-subject coefficient of variation (CV) is 25% and the true ratio of means is 0.89 (89%), there is at least 90% power to demonstrate the bioequivalence (bioequivalence range: 0.80 to 1.250 [80% – 125%], alpha=0.05). Power calculations were also performed under alternative assumptions for the CV and mean ratio. Assuming the CV is 30% and the true ratio of means is 0.89 (89%), with 100 evaluable patients, there is at least 82% power to demonstrate bioequivalence. Assuming the true ratio is 0.90 (90%), the power is 96% and 88% assuming CVs of 25% and 30%, respectively.

The final analysis of bioequivalence will be based on Stage 2 BA/BE evaluable patients only, with a target sample size of 100 evaluable patients. Patients may be identified as non-evaluable due to issues arising during the study conduct, such as:

- Emesis within 9 hours of dosing,
- Dosing errors,
- Patient did not fast prior to dosing,
- Missing critical PK sample on Day 8,
- Failure to complete both PK periods, and
- Significant changes to the patient medical status that would potentially affect the PK profile as determined by the Sponsor in consultation with the Investigator prior to PK data analysis.

In this patient population, approximately 170 total patients are targeted for enrollment, assuming a 35% non-evaluability rate during the study conduct, and an additional 10% non-evaluability rate during PK analysis. The non-evaluability rate arising during the study conduct will be continuously monitored by the Sponsor and the total number of enrolled patients may be adjusted accordingly with the aim to target the resulting sample size of 100 BA/BE evaluable patients.

#### Stage 3

Assuming the true ratio of means is 1 and the intra-subject CV is 20% for  $AUC_{0-t}$  and  $AUC_{0-\infty}$ , with 16 evaluable patients, there is approximately 83% probability that the 90% CI of the ratio of geometric means will be within 0.800 and 1.250 (80% - 125%). Based on the results of a FE study conducted using the capsule formulation, an effect of a high-fat meal on  $C_{max}$  is possible. The sample size of 16 patients is deemed adequate to characterize this effect.  $AUC_{0-t}$  and  $AUC_{0-\infty}$  will be the primary parameters for analysis.

The primary analysis will be based on the FE Evaluable Population as it is the most conservative approach, which maximizes the benefits of the crossover design, where each patient serves as their own control. Results for the PK Evaluable Population will also be summarized and reported for this study.

To account for non-evaluable patients, approximately 20 total patients are targeted for enrollment. The final analysis will be based on Stage 3 FE evaluable patients only. Patients may be identified as non-evaluable due to issues arising during the study conduct, such as:

• Emesis within 10 hours of dosing,

- Dosing errors,
- Patient did not follow dietary requirements prior to dose and post-dose,
- Failure to complete both PK periods, and
- Significant changes to the patient medical status that would potentially affect the PK profile as determined by the Sponsor in consultation with the Investigator prior to PK data analysis.

Patients who miss critical PK samples or miss sufficient samples to render calculation of AUC unreliable will be discontinued from the PK Phase; those that meet other criteria for continued niraparib therapy will be eligible to be screened for the Extension Phase. The non-evaluability rate arising during the study conduct will be continuously monitored by the Sponsor and the total number of enrolled patients may be adjusted accordingly with the aim to target the resulting sample size of 16 evaluable patients.

#### 3.2. General Methods

All statistical analyses will be performed using SAS statistical software v9.4 or later, unless otherwise noted. All output will be incorporated into Microsoft Word or Excel files, or Adobe Acrobat PDF files, sorted and labeled according to the International Council for Harmonisation (ICH) recommendations, and formatted to the appropriate page size(s).

For categorical variables, summary tabulations of the number and percentage of patients within each category of the parameter will be presented. Percentages will be based on the patients with a non-missing parameter unless missing category is presented. Percentages will be reported to one decimal place. Percentages will not be presented for zero counts.

For continuous variables, the number of patients, mean, standard deviation (SD), median, first quartile  $(Q_1)$ , third quartile  $(Q_3)$ , minimum, and maximum values will be presented. Mean, median,  $Q_1$ , and  $Q_3$  will be reported to 1 more decimal place than the raw data, while the SD will be reported to 2 more decimal places than the raw data.

All data listings that contain an evaluation date will also contain a relative study day. A unique relative study day will be calculated for the PK Phase and Extension Phase based on the first date of dosing within the respective study phase. Pre-treatment and on-treatment study days are numbered relative to the day of the first dose of study drug which is designated as Day 1. The preceding day is Day -1, the day before that is Day -2, etc. Post-treatment study days are numbered relative to the first dose and are designated as Day +1, Day +2, etc.

#### In addition:

- Medical history and AEs will be coded using the most up-to-date version of Medical Dictionary for Regulatory Activities (MedDRA).
- Laboratory parameter changes during the Extension Phase for selected laboratory tests will be described using shift tables, relative to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
- Concomitant medications will be coded using the latest version of the World Health Organization's (WHO) Anatomical Therapeutic Chemical (ATC) classification.
- CIs will be presented to one more decimal place than the raw data.

Summaries in the Extension Phase will be performed by formulation and overall, regardless of starting dose, unless otherwise specified. The niraparib formulation will be included in the listing for the Extension Phase.

All tables, figures, and listings will include footers at the bottom of the page reflecting the programs used to generate the tables, figures, and listings, and date and time of the generation of the output.

Some minor modifications may be necessary to the planned design of tables, figures, and listings to accommodate data collected during the actual study conduct.

#### 3.3. Baseline Definitions

For all analyses unless otherwise noted, baseline is defined as the most recent measurement prior to the first administration of study drug, for each phase of the study. Baseline can be the same date as first dose, given the measurement is expected prior to first dose when only date information is available.

## 3.4. Methods of Pooling Data

Data will be pooled across study sites.

#### 3.5. Adjustments for Covariates

No formal statistical analyses that adjust for possible covariate effects are planned for the safety endpoints.

#### 3.6. Multiplicity Adjustment

Multiplicity is not adjusted in this study.

### 3.7. Subpopulations

Not applicable.

## 3.8. Withdrawals, Drop-outs, Loss to Follow-up

Patients will not be replaced during Stage 1. During Stage 2 and Stage 3, patients who do not complete Period 1 or Period 2, or who are missing PK samples which render the determination of the primary PK parameters not possible, will be replaced. After evaluation, patients receiving concomitant medications which may affect the final analysis may be replaced.

#### 3.9. Missing Data

In general, there will be no imputations made to accommodate missing data points. All data recorded on the eCRF will be included in data listings for the CSR.

When tabulating AE data, partial dates will be handled as follows:

- If the day of the month is missing, the onset day will be set to the first day of the month unless it is the same month and year as first study treatment. In this case, in order to conservatively report the event as treatment-emergent, the onset date will be assumed to be the date of first study treatment.
- If the onset day and month are both missing, the day and month will be assumed to be January 1, unless the event occurred in the same year as the first study treatment. In this case, the event onset will be coded to the day of first study treatment in order to conservatively report the event as treatment-emergent.

• A missing onset date will be coded as the first day of study treatment. If the resulting onset date is after a reported date of resolution, the onset date will be set equal to the date of resolution, after considering any required imputation.

Imputation of partial dates is used only to determine whether an event is treatment-emergent; data listings will present the partial date as recorded in the eCRF.

Partial start dates for prior/concomitant medication, growth factor and transfusion data will be handled in the same way as described above for adverse events. Stop dates will be imputed as follows:

- If only day of the month is missing, the end day will be set to the last day of the month.
- If end day and end month are missing, and the year is not missing, then the day and month will be set to December 31 (or date of study discontinuation/completion if earlier than December 31).
- If the stop date is completely missing, it will be set to the date of study discontinuation/completion.
- If the imputed stop date is greater than the date of study discontinuation/completion then the date will be set to the date of study discontinuation/completion.

#### 3.10. Visit Windows

By-visit summaries and analyses will be performed by nominal visit. All data will be tabulated per the evaluation visit as recorded on the eCRF even if the assessment is outside of the visit window for analysis.

#### 3.11. Interim Analysis

There will be no interim analysis for this study.

#### 3.12. COVID-19

COVID-19 pandemic may impact the conduct of clinical studies. Challenges may arise from quarantines, site closures, travel limitations interruptions to the supply chain for the investigational product or other considerations if site personnel or patients become infected with COVID-19. These challenges may lead to difficulties in meeting protocol specified procedures, including administering or using the investigational product or adhering to protocol-mandated visits and laboratory/diagnostic testing.

This study was initiated by TESARO, which was subsequently acquired by GSK. Prior to the acquisition, protocol deviations were classified using TESARO definitions. The TESARO protocol deviation system was decommissioned in May 2020, and thereafter, protocol deviations were classified using GSK definitions.

All protocol deviations collected during the study will be reviewed by the TESARO (for Stage 1 and Stage 2) or GSK (for Stage 3 only) study team, as appropriate, in order to identify TESARO "Significant"/"Important" protocol deviations and GSK "Important" protocol deviations, respectively. Consistent with ICH E3 guidance, only protocol deviations identified as "Important" (GSK) are evaluated in the CSR for impact on the Stage 3 primary endpoint.

## 4. Study Analyses

#### 4.1. Patient Disposition

A by-patient data listing of patient disposition information will be presented for each phase.

For the PK Phase (Stage 1, Stage 2, and Stage 3 separately), patient disposition will be tabulated and will include the number of patients in each of the following categories:

- Patients screened
- Patients randomized
- Patients treated with each formulation (Stage 1 and 2)
- Patients treated in fed and fasted state (Stage 3)
- Patients in the Safety Population
- Patients completing the PK Phase
- Primary reason for discontinuation from the PK Phase
- Primary reason for discontinuation from the study, for patients who do not continue to the Extension Phase.

For the Open-Label Extension Phase, patient disposition will be tabulated and will include the number of patients in each of the following categories:

- Patients treated with at least one dose
- Patients who discontinue treatment and the reason(s) for withdrawal
- Patients who discontinue the study and the reason(s) for withdrawal.

#### 4.2. Demographics, Baseline Characteristics and Medical History

Demographics, baseline characteristics, primary cancer history, and medical history information will be summarized for the PK Safety Population by sequence and overall (Stage 1, Stage 2 and Stage 3 separately) and for the Open-Label Extension Phase, using descriptive statistics for the Safety Population. No formal statistical comparisons will be performed. Demographics and baseline characteristics will also be summarized for the BA for Stage 1, BE Evaluable Population for Stage 2 and FE Evaluable Population for Stage 3.

The demographic and baseline characteristics tables will include the following variables:

- Age at time of screening (years)
- Age categories (18 to <65, 65 to  $<75, \ge 75$ ; and  $\ge 65$ )
- Sex
- Race (White, Black, Asian, American Indian/Alaska Native, Native Hawaiian or other Pacific Islander, Other and Not Reported)
- Ethnicity (Hispanic or Latino, not-Hispanic or Latino, Not Reported and Unknown)
- Baseline weight (in kilograms)
- Baseline height (in centimeters)
- Baseline body mass index (BMI) (kg/m<sup>2</sup>), calculated using the patient's height and weight at screening [BMI (kg/m<sup>2</sup>) = weight (kg) / height (m)<sup>2</sup>]
- Eastern Cooperative Oncology Group (ECOG) performance status at baseline.

Primary cancer history will be summarized for the safety population and will include the following variables:

- Tumor type
- Time from first diagnosis to informed consent (years)
- Cancer stage (most recent) (Locally advanced, Metastatic)
- Number of prior lines of therapy
- Any prior radiotherapy.

Prior anti-cancer treatments will be coded using the most current version of the WHO Drug Dictionary. The number and percentage of patients reporting the use of at least one preferred term will be reported for the Safety Population in the PK Phase (Stage 1, Stage 2 and Stage 3 separately) and the Safety Population in the Extension Phase.

Medical history will be coded using the most current version of MedDRA, and the number and percentage of patients experiencing at least one such diagnosis by MedDRA System Organ Class (SOC) and preferred term (PT) will be reported for the Safety Population in the PK Phase (Stage 1, Stage 2 and Stage 3 separately) and the Safety Population in the Extension Phase.

Demographics, baseline characteristics, primary cancer history, and medical history information for each patient will be provided in data listings.

#### 4.3. Investigator Assessment of Response

Investigator assessment of response will be provided in data listings for the Extension Phase. Additional descriptive summaries of response may be performed by tumor type.

#### 4.4. Safety Evaluation

#### 4.4.1. Treatment Exposure and Compliance

#### PK Phase

The number and percentage of patients receiving capsules and tablets during the PK Phase (Stage 1 and Stage 2, separately) will be summarized. For Stage 3, the number of tablets received will be summarized by fed/fasted state.

A by-patient listing of the niraparib treatment data will be produced for the PK Safety Population.

#### **Extension Phase**

Study treatment exposure and compliance will be summarized by formulation (Capsule; Tablet) and overall, including:

- Number and percentage of patients who initiated 1, 2, 3, 4, 5,  $\geq$ 6 treated cycles (Maximum Number of Cycles).
- Median number of cycles started.
- Duration of treatment (months), defined as: [last dose date first dose date in the Extension Phase + 1] / 30.4375.
- Duration on study (months), defined as:

[last contact date - first dose date in the Extension Phase + 1] / 30.4375, where last contact date is the last visit date or date of death.


- Dose intensity (mg/day), defined as:
  - Sum of daily doses consumed / [last dose date first dose date in Extension Phase + 1]
- Number of patients with at least one dose interruption.
- Number of patients with at least one dose reduction.
- Number of patients with at least one dose re-escalation.

In addition, the starting niraparib dose for each cycle will be summarized.

A by-patient listing of the niraparib treatment data will be produced for the Open-Label Extension Phase safety population.

#### 4.4.2. Adverse Events

All AEs will be classified by SOC and PT using the most up-to-date version of MedDRA.

Per protocol, all SAEs will be collected from the signing of the ICF for this study through 90 days after the last dose of study drug (or until the start of alternate anticancer therapy, whichever occurs first, and recorded in the eCRF.

All AEs, regardless of the source of identification (e.g., physical examination, laboratory assessment, ECG, or reported by patient), will be collected and recorded in the eCRF for each patient from the time of randomization and/or treatment assignment until 30 days after the last dose of study drug.

All AEs experienced by a patient, regardless of the suspected causality, will be monitored until the AE or SAE has resolved, until AE(s) or SAE(s) have returned to baseline or normal levels, until stabilized with a satisfactory explanation for the changes observed, until the patient is lost to follow-up, or until the patient has died, starts alternate anti-cancer therapy, or until the patient withdraws consent.

For analysis, TEAEs will be defined as any AEs collected with a start date on or after the first dose of study drug. Any AEs recorded in the database that occur from the time of ICF to first dose will be listed only and not included in safety analyses. Pre-existing conditions will be recorded in the eCRF on the Medical History or appropriate page.

The severity of the toxicities will be graded according to the NCI CTCAE v4.03. Within the same MedDRA PT, only the most severe AE for each patient will be counted in tabulations by severity. Within a MedDRA SOC, patients with more than 1 MedDRA PT will be counted only once for the most severe AE reported.

The Investigator must provide a causality assessment (related or not related) regarding the relationship of the event with the study drug and/or study procedure for all AEs. In Stage 1, for analysis of the PK Phase, AEs considered related to either tablet or capsule will be considered to be related to study drug. Any AEs for which the relationship is missing (for either tablet or capsule during the Stage 1 PK Phase) will be considered related to study treatment. During Stage 2 PK Phase, Stage 3 PK Phase and Extension Phase, relationship relative to niraparib will be considered. Within the same MedDRA PT, only the AE with the highest ranked relationship to treatment for each patient will be counted in tabulations by relationship to treatment. Within a MedDRA SOC, patients with more than 1 MedDRA PT will be counted only once for

the AE that is most related to treatment. The imputation for a missing relationship will take place prior to determining the most related AE within a SOC or PT for a given patient.

If the start date is missing for an AE and the actual start date cannot be determined from a partial date, the AE will be considered treatment-emergent.

Adverse Events of Special Interest (AESI) for niraparib are the following:

- Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML)
- Secondary cancers (new malignancies [other than MDS or AML])
- Pneumonitis (for Stage 1 and Stage 2 only)
- Embryo-fetal toxicity (for Stage 1 and Stage 2 only).

AEs will be classified into the following time periods for analysis.

- PK Phase (for Stage 1, Stage 2, and Stage 3 separately):
  - o Period 1: Any AE that begins on or after Dose 1 but prior to Dose 2.
    - For Stage 1, Period 1 will be defined as 7-days post Dose 1 for patients who do not receive Dose 2.
    - For Stage 2 and Stage 3, Period 1 will be defined as 14-days post Dose 1 for patients who do not receive Dose 2.
  - o Period 2: Any AEs that begins on or after Dose 2 but prior to the end of the PK Phase as defined by 7-days post Dose 2.
  - o Safety Follow-Up/Extension Screening Period:
    - For patients not participating in the Extension Phase, AEs that begin after the end of the PK Phase.
    - For patients participating in the Extension Phase, AEs that begin after the end of the PK Phase until the date of first dose in the Extension Phase.
- Open-Label Extension Phase:
  - o Any AEs that start on or after the first dose in the Extension Phase.
- Any AEs with onset during the PK Phase/Safety Follow-Up/Extension Screening Period and ongoing/ resolved during the Extension Phase will be listed separately.

The analyses indicated below will be performed for each of the above-mentioned phases.

A high-level overview of TEAEs will be presented in a summary table. This table will include the number and percentage of patients for the following categories:

- Any TEAE
- Any related TEAEs
- Any serious TEAEs
- Any related serious TEAEs
- Any TEAEs with CTCAE toxicity grade 3 or above
- Any related TEAEs with CTCAE toxicity grade 3 or above
- Any TEAEs leading to treatment discontinuation
- Any related TEAEs leading to treatment discontinuation

- Any TEAEs leading to dose interruption
- Any TEAEs leading to dose reduction
- Any TEAEs leading to death.

The number and percentage of patients reporting a TEAE will be summarized in the following additional AE tables. AE tabulations will be ordered in terms of decreasing frequency for SOC (alphabetically for SOCs with the same number of AEs reported), and decreasing frequency for PT within SOC (alphabetically for PTs with the same number of AEs reported within a SOC) considering the overall rate.

- TEAE by SOC and PT
- Related TEAE by SOC and PT
- Treatment emergent SAEs by SOC and PT
- Related treatment emergent SAEs by SOC and PT
- TEAE with toxicity grade 3 or above by SOC and PT
- Related TEAE with toxicity grade 3 or above by SOC and PT
- TEAEs leading to treatment discontinuation by SOC and PT
- TEAEs leading to dose interruption by SOC and PT (Extension Phase Only)
- TEAEs leading to dose reduction by SOC and PT
- TEAEs leading to death by SOC and PT
- TEAE by PT (sorted by frequency)
- TEAE by SOC, PT, and maximum toxicity grade
- Treatment emergent AESI.

For Stage 1 and Stage 2 PK Phase, primary tabulations for the PK Phase data will be provided by formulation (regardless of period), those occurring during the Follow-up/Extension Screening, and overall. In addition, the high-level overview of TEAEs and summary of TEAEs by SOC and PT will be summarized by sequence and formulation. For Stage 3 PK Phase, primary tabulations for the PK Phase data will be provided by fed/fasted state (regardless of period), and overall. In addition, the high-level overview of TEAEs and summary of TEAEs by SOC and PT will be summarized by sequence and fed/fasted state. For the Open-Label Extension Phase, data will be summarized by formulation and for all patients overall.

The following by-patient listings will be produced for the PK Phase (Stage 1, Stage 2, and Stage 3 separately) and the Open-Label Extension Phase:

- All TEAEs
- Treatment emergent SAEs
- All Deaths
- TEAEs leading to dose interruption (Extension Phase Only)
- TEAEs leading to dose reduction
- TEAEs leading to treatment discontinuation
- Any TEAEs with onset during PK Phase (including Safety Follow-Up/Extension Screening Period) and ongoing/resolved during Extension Phase.

#### 4.4.3. Laboratory Data

Laboratory assessments for safety oversight are performed locally at each center's laboratory by means of their established methods. All laboratory values will be converted to SI units and classified as normal, low, or high based on normal ranges supplied by the local laboratories and upon employing standardization.

A by-patient listing of all laboratory data will be provided, with laboratory reference ranges and abnormal values highlighted, and including center, patient identifier, and visit for the PK Phase and the Extension Phase of the study.

For the Extension Phase, select hematology (hemoglobin, neutrophils and platelets) and chemistry (bilirubin, creatinine, aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) will be analyzed using change from baseline by visit.

For the Extension Phase, select hematology (hemoglobin, neutrophils and platelets) and chemistry tests (bilirubin, creatinine, ALT, and AST), baseline and post-baseline results will be categorized by NCI CTCAE v4.03 grade (Table 2). Shift tables will be produced by maximum post-baseline grade. Results that are considered 'normal' will be assigned a Grade 0.

Table 2 NCI Common Terminology Criteria for Adverse Events v4.03 (CTCAE)



#### 4.4.4. Vital Signs and Physical Examination

Vital sign measurements will be presented for each patient in a data listing.

Baseline physical examination findings will be presented in a data listing. Any new or changed condition will be captured as an adverse event and will be summarized in the AE tables and listings.

#### 4.4.5. Electrocardiogram

Standard 12-lead ECGs will be performed locally for patients in the study. Any ECG findings that are assessed as clinically significant and are reported as an AE or SAE will be summarized in the AE tables and listings.

All ECG results (i.e., interpretations) for each patient will be provided in a data listing.

#### 4.4.6. Prior and Concomitant Mediations

Medications collected at Screening and during the study will be coded using the current version of the WHO Drug dictionary. Study treatment, prior anti-cancer treatments for primary cancer, transfusions and growth factors are collected and summarized separately. For each of the study phases (Stage 1 PK, Stage 2 PK, Stage 3 PK and Extension Phase), medications will be categorized as prior or concomitant using the following definitions:

- Prior medications during the PK Phase: any medications which started prior to the first dose date of study treatment during the PK Phase.
- Concomitant medications during the PK Phase: any medications being taken on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase.
  - o For Stage 2 PK Phase, concomitant medications will be further identified as those taken during the PK collection period, defined by dates of the first PK-draw to last PK-draw.
- Prior medications during the Extension Phase: any medications which started prior to the first dose date of study treatment during the Extension Phase.
- Concomitant medications during the Extension Phase: any medications on or after the first treatment dosing date in the Extension Phase through 30 days after the last dose of treatment.
- Any concomitant medication taken during PK Phase that were ongoing during the Extension Phase will be classified as Both, i.e., concomitant and prior, for the purposes of the Extension Phase.

Note: medications can be classified as both prior and concomitant.

Both prior medications and concomitant medications will be summarized by ATC classification drug class and WHO preferred name using the number and percentage of patients for each cohort. A patient reporting the same medication more than once will be counted only once when calculating the number and percentage of patients who received that medication in a given time category (prior or concomitant). The summary of concomitant medications will be ordered alphabetically by drug class and then by descending frequency of preferred name in total within the drug class. For drugs with the same frequency, sorting will be done alphabetically. Summaries will be based on the safety population.

For PK Stage 2, an additional summary of concomitant medications used during the PK collection period will be provided for the BE Evaluable Population.

For each phase of the study, all prior and concomitant medications will be provided in a by-patient listing sorted by patient ID number and administration date in chronological order.

#### 4.4.7. Prior and Concomitant Transfusions and Growth Factors

The number and percentage of patients receiving prior and concomitant growth factors during the PK Phase and Extension Phase will be summarized. The data will be classified as prior or concomitant using similar logic as provided in Section 4.4.6.

For each phase of the study, all prior and concomitant transfusions and growth factor use will be provided in a by-patient listing sorted by patient ID number and administration date in chronological order.

#### 4.4.8. COVID-19

The PK Phase Stage 3 of the trial takes place during COVID-19 pandemic, as a result, some of the trial procedures could be impacted in terms of missing visits and/or assessments. Missing protocol required data/visits due to COVID-19 must be noted in participant notes and recorded as COVID-19-related protocol deviations.

A summary of the following COVID-19 assessments will be produced: case diagnosis, COVID-19 test performed, and results of the COVID-19 test.

The incidence of COVID-19 related AEs and SAEs will be summarized as part of the safety reporting summaries along with COVID-19-related as reasons for treatment discontinuation.

A listing of all patients with COVID-19 assessments and symptom assessments will be produced and will include the following:

- Treatment sequence
- Patient number
- COVID-19 case diagnosis
- COVID-19 test performed
- Result of the COVID-19 test
- Assessments and symptom assessments performed
- Results of the assessments and symptom assessments.

For PK Phase Stage 3, a separate listing defining "Important" GSK protocol deviations related to COVID-19 will be presented.

For protocol deviation reporting during the Extension Phase, a listing will be produced to present TESARO Classification of protocol deviations for patients continuing from Stage 1 and Stage 2, and GSK Classification of protocol deviations for patients continuing from Stage 3.

## 5. Changes to Planned Analyses

There is no change between the protocol-defined statistical analyses and those planned in this SAP.

#### 4.5. Changes in v5.0 of the SAP

Section 2.2 updated to include a summary tables of Important protocol deviations for Stage 3 PK Phase and Open-Label Extension Phases, as well as clarification of associated deviation listings presenting only protocol deviations classified as "Important".

#### 4.6. Changes in v6.0 of the SAP

Section 1.2 updated to reflect the change in PK data cut requirements for final Stage 3 analysis.

#### 4.7. Changes in v7.0 of the SAP

Case record form (CRF) versions updated to align with CRF booklet version upgrades starting from SAP version 4.0 onwards.

Section 2 updated to include definition for dose intensity in exposure table for Extension Phase.

Section 3.2 'Dose at onset of AE' column removed from AE listings.

Section 4.4.2 updated AE classification for PK Period 1 for Stage 3.

Table 2 header row labels updated to correct CTCAE version.

Table numbering and output header formatting updated to reflect the produced outputs.

Header row labels for Extension Phase updated to TABLET, CAPSULE and OVERALL for consistency.

Additional tables and listings have been added/modified for Extension Phase; disclosure and plain language summary reporting tables added across all study stages.

All-Cause Mortality table added for final study disclosure reporting purposes of the Extension Phase.

# 6. Appendix

# 6.1. Planned Statistical Tables, Listings, and Figures

| TABLE 14.1.2.1B DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) |
|---|
| Table 14.1.1c Subject Disposition in the Extension Phase (All Patients in the Extension Phase)45Table 14.1.1d Subject Disposition in the PK Phase (All Patients in the Stage 3 PK Phase)46Table 14.1.2a Demographics (Safety Population in the Stage 1 PK Phase)47Table 14.1.2.1a Demographics (BA Evaluable Population in the Stage 1 PK Phase)47Table 14.1.2.1b Demographics (Safety Population in the Stage 2 PK Phase)47Table 14.1.2.2b Demographics (BE Evaluable Population in the Stage 2 PK Phase)48Table 14.1.2c Demographics (Safety Population in the Extension Phase)48Table 14.1.2.1d Demographics (Safety Population in the Stage 3 PK Phase)48Table 14.1.2.2d Demographics (FE Evaluable Population in the Stage 3 PK Phase)48Table 14.1.3a Baseline Characteristics (Safety Population in the Stage 1 PK Phase)49Table 14.1.3.1b Baseline Characteristics (BA Evaluable Population in the Stage 1 PK Phase)49Table 14.1.3.2b Baseline Characteristics (Safety Population in the Stage 2 PK Phase)50Table 14.1.3.2b Baseline Characteristics (BE Evaluable Population in the Stage 2 PK Phase)50Table 14.1.3c Baseline Characteristics (Safety Population in the Extension Phase)50 |
| TABLE 14.1.1D SUBJECT DISPOSITION IN THE PK PHASE (ALL PATIENTS IN THE STAGE 3 PK PHASE) |
| TABLE 14.1.2A DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 1 PK PHASE)47TABLE 14.1.2.1B DEMOGRAPHICS (BA EVALUABLE POPULATION IN THE STAGE 1 PK PHASE)47TABLE 14.1.2.1B DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 2 PK PHASE)47TABLE 14.1.2.2B DEMOGRAPHICS (BE EVALUABLE POPULATION IN THE STAGE 2 PK PHASE)48TABLE 14.1.2C DEMOGRAPHICS (SAFETY POPULATION IN THE EXTENSION PHASE)48TABLE 14.1.2.1D DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 3 PK PHASE)48TABLE 14.1.2.2D DEMOGRAPHICS (FE EVALUABLE POPULATION IN THE STAGE 3 PK PHASE)48TABLE 14.1.3 BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE STAGE 1 PK PHASE)49TABLE 14.1.3.1B BASELINE CHARACTERISTICS (BA EVALUABLE POPULATION IN THE STAGE 2 PK PHASE)50TABLE 14.1.3.2B BASELINE CHARACTERISTICS (BE EVALUABLE POPULATION IN THE STAGE 2 PK PHASE)50TABLE 14.1.3.2B BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE STAGE 2 PK PHASE)50TABLE 14.1.3.2B BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE EXTENSION PHASE)50 |
| Table 14.1.2.1a Demographics (BA Evaluable Population in the Stage 1 PK Phase)47Table 14.1.2.1b Demographics (Safety Population in the Stage 2 PK Phase)47Table 14.1.2.2b Demographics (BE Evaluable Population in the Stage 2 PK Phase)48Table 14.1.2c Demographics (Safety Population in the Extension Phase)48Table 14.1.2.1d Demographics (Safety Population in the Stage 3 PK Phase)48Table 14.1.2.2d Demographics (FE Evaluable Population in the Stage 3 PK Phase)48Table 14.1.3a Baseline Characteristics (Safety Population in the Stage 1 PK Phase)49Table 14.1.3.1a Baseline Characteristics (BA Evaluable Population in the Stage 1 PK Phase)49Table 14.1.3.1b Baseline Characteristics (Safety Population in the Stage 2 PK Phase)50Table 14.1.3.2b Baseline Characteristics (BE Evaluable Population in the Stage 2 PK Phase)50Table 14.1.3c Baseline Characteristics (Safety Population in the Extension Phase)50Table 14.1.3c Baseline Characteristics (Safety Population in the Extension Phase)50 |
| TABLE 14.1.2.1B DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) |
| TABLE 14.1.2.2B DEMOGRAPHICS (BE EVALUABLE POPULATION IN THE STAGE 2 PK PHASE) |
| TABLE 14.1.2C DEMOGRAPHICS (SAFETY POPULATION IN THE EXTENSION PHASE)48TABLE 14.1.2.1D DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 3 PK PHASE)48TABLE 14.1.2.2D DEMOGRAPHICS (FE EVALUABLE POPULATION IN THE STAGE 3 PK PHASE)48TABLE 14.1.3A BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE STAGE 1 PK PHASE)49TABLE 14.1.3.1A BASELINE CHARACTERISTICS (BA EVALUABLE POPULATION IN THE STAGE 1 PK PHASE)49TABLE 14.1.3.1B BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE STAGE 2 PK PHASE)50TABLE 14.1.3.2B BASELINE CHARACTERISTICS (BE EVALUABLE POPULATION IN THE STAGE 2 PK PHASE)50TABLE 14.1.3C BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE EXTENSION PHASE)50 |
| TABLE 14.1.2.1D DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) |
| TABLE 14.1.2.2D DEMOGRAPHICS (FE EVALUABLE POPULATION IN THE STAGE 3 PK PHASE) |
| TABLE 14.1.3A BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) |
| Cable 14.1.3.1a Baseline Characteristics (BA Evaluable Population in the Stage 1 PK Phase) |
| Table 14.1.3.1b Baseline Characteristics (Safety Population in the Stage 2 PK Phase)50Table 14.1.3.2b Baseline Characteristics (BE Evaluable Population in the Stage 2 PK Phase)50Table 14.1.3c Baseline Characteristics (Safety Population in the Extension Phase)50 |
| Table 14.1.3.2b Baseline Characteristics (BE Evaluable Population in the Stage 2 PK Phase) 50 Table 14.1.3c Baseline Characteristics (Safety Population in the Extension Phase) 50 |
| Table 14.1.3c Baseline Characteristics (Safety Population in the Extension Phase) 50 |
| FADLE 1/1/2/1D DAGELINE CHAD ACTEDISTICS (SAFETY DODLH ATION IN THE STACE 2 DV DHASE) 50 |
| TABLE 14.1.3.1D BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) 50 TABLE 14.1.3.2D BASELINE CHARACTERISTICS (FE EVALUABLE POPULATION IN THE STAGE 3 PK PHASE) 50 |
| Table 14.1.3.2D Baseline Characteristics (FE Evaluable Population in the Stage 3 PK Phase)51 |
| Table 14.1.48 Primary Cancer History (Safety Population in the Stage 1 PK Phase) |
| Table 14.1.4c Primary Cancer History (Safety Population in the Extension Phase) 51 51 51 |
| Table 14.1.4d Primary Cancer History (Safety Population in the Stage 3 PK Phase) |
| Table 14.1.5a Prior Anti-Cancer Treatment (Safety Population in the Stage 1 PK Phase) |
| Table 14.1.5B Prior Anti-Cancer Treatment (Safety Population in the Stage 2 PK Phase) |
| Table 14.1.5c Prior Anti-Cancer Treatment (Safety Population in the Extension Phase) |
| Table 14.1.5D Prior Anti-Cancer Treatment (Safety Population in the Stage 3 PK Phase) |
| Table 14.1.6A Medical History (Safety Population in the Stage 1 PK Phase) |
| TABLE 14.1.6B MEDICAL HISTORY (SAFETY POPULATION IN THE STAGE 1 PK PHASE) |
| Table 14.1.6c Medical History and Prior Blood Disorders (Safety Population in the Extension Phase) |
| ABLE 14.1.0C MEDICAL HISTORY AND PRIOR BLOOD DISORDERS (SAFETY POPULATION IN THE EXTENSION PHASE) |
| Fable 14.1.6D Medical History (Safety Population in the Stage 3 PK Phase) |
| Fable 14.1.7a Prior Medications by ATC and PT (Safety Population in the Stage 1 PK Phase)54 |
| Table 14.1.7B Prior Medications by ATC and PT (Safety Population in the Stage 2 PK Phase)54 |
| Table 14.1.7c Prior Medications by ATC and PT (Safety Population in the Extension Phase)54 |
| Table 14.1.7D Prior Medications by ATC and PT (Safety Population in the Extension Phase)54 |
| TABLE 14.1.8A CONCOMITANT MEDICATIONS BY ATC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE)55 |
| TABLE 14.1.8.1B CONCOMITANT MEDICATIONS BY ATC AND PT (SAFETY POPULATION IN THE STAGE 11 KT HASE)55 |
| TABLE 14.1.8.2B CONCOMITANT MEDICATIONS BY ATC AND TY (SAFETY FOR DEATHON IN THE STAGE 2 TRATIFIASE) 35 |
| EVALUABLE POPULATION IN THE STAGE 2 PK PHASE) |
| FABLE 14.1.8c Concomitant Medications by ATC and PT (Safety Population in the Extension Phase)55 |
| TABLE 14.1.8D CONCOMITANT MEDICATIONS BY ATC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE)55 |
| TABLE 14.1.9A CONCOMITANT MEDICATIONS BY ATC AND LY (SAFETY POPULATION IN THE STAGE 3 TK THASE)30 |
| PHASE) |
| TABLE 14.1.9B CONCOMITANT TRANSFUSIONS AND GROWTH FACTORS (SAFETY POPULATION IN THE STAGE 2 PK |
| PHASE) |

| TABLE 14.1.9C CONCOMITANT TRANSFUSIONS AND GROWTH FACTORS (SAFETY POPULATION IN THE EXTENSION | |
|---|---|
| Phase) | 57 |
| TABLE 14.1.9D CONCOMITANT TRANSFUSIONS AND GROWTH FACTORS (SAFETY POPULATION IN THE STAGE 3 PK | |
| Phase) | 57 |
| TABLE 14.1.10c SUMMARY OF INVESTIGATOR-ASSESSED BEST RESPONSE BY TUMOR TYPE (SAFETY POPULATION IN | N |
| THE EXTENSION PHASE) | 58 |
| TABLE 14.3.1.1.1A OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS (SAFETY POPULATION IN TH | |
| STAGE 1 PK PHASE) | |
| TABLE 14.3.1.1.1B OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS (SAFETY POPULATION IN TH | |
| STAGE 2 PK PHASE) | |
| TABLE 14.3.1.1.1c OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS (SAFETY POPULATION IN TH | |
| EXTENSION PHASE) | |
| TABLE 14.3.1.1.1.1c Overall Summary of Treatment Emergent Adverse Events Ongoing from PK Phasi | |
| (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| TABLE 14.3.1.1.1D OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS (SAFETY POPULATION IN TH | |
| STAGE 3 PK PHASE) | 61 |
| TABLE 14.3.1.1.2A OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SEQUENCE AND PERIOD | |
| (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 62 |
| TABLE 14.3.1.1.2B OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SEQUENCE AND PERIOD | |
| (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 62 |
| TABLE 14.3.1.1.2D OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SEQUENCE AND PERIOD | |
| (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 63 |
| TABLE 14.3.1.2.1A SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION | |
| IN THE STAGE 1 PK PHASE) | 64 |
| TABLE 14.3.1.2.1B SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION | N |
| IN THE STAGE 2 PK PHASE) | 64 |
| TABLE 14.3.1.2.1C SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION | N |
| IN THE EXTENSION PHASE) | 65 |
| TABLE 14.3.1.2.1D SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION | N |
| IN THE STAGE 3 PK PHASE) | |
| TABLE 14.3.1.2.1.1D SUMMARY OF COVID-19 RELATED ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION | |
| THE STAGE 3 PK PHASE) | |
| TABLE 14.3.1.2.2A SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION | |
| IN THE STAGE 1 PK PHASE) | |
| TABLE 14.3.1.2.2B SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION | |
| IN THE STAGE 2 PK PHASE) | |
| TABLE 14.3.1.2.2D SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION | |
| IN THE STAGE 3 PK PHASE) | |
| TABLE 14.3.1.3A SUMMARY OF RELATED TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| Town 142 122 Congress on Day and TEAE are COC and DT (Congress Days and Teae and DV Days and | |
| TABLE 14.3.1.3B SUMMARY OF RELATED TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| T 144.14. (3 | |
| TABLE 14.3.1.3C SUMMARY OF RELATED TEAE BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| TABLE 14.3.1.3D SUMMARY OF RELATED TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| TABLE 14.3.1.4A SUMMARY OF SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| TABLE 14.3.1.4B SUMMARY OF SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| TABLE 14.3.1.4C SUMMARY OF SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE). | |
| TABLE 14.3.1.4D SUMMARY OF SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 70 |

| TABLE 14.3.1.5A SUMMARY OF RELATED SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) |
|---|
| TABLE 14.3.1.5B SUMMARY OF RELATED SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 PK |
| PHASE) |
| TABLE 14.3.1.5C SUMMARY OF RELATED SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION |
| PHASE) |
| TABLE 14.3.1.5D SUMMARY OF RELATED SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 3 PK |
| PHASE) |
| TABLE 14.3.1.6A SUMMARY OF TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY POPULATION IN |
| THE STAGE 1 PK PHASE) |
| TABLE 14.3.1.6B SUMMARY OF TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY POPULATION IN |
| THE STAGE 2 PK PHASE) |
| THE EXTENSION PHASE) |
| TABLE 14.3.1.6D SUMMARY OF TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY POPULATION IN |
| THE STAGE 3 PK PHASE) |
| TABLE 14.3.1.7A SUMMARY OF RELATED TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY |
| POPULATION IN THE STAGE 1 PK PHASE) |
| TABLE 14.3.1.7B SUMMARY OF RELATED TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY |
| POPULATION IN THE STAGE 2 PK PHASE) |
| TABLE 14.3.1.7C SUMMARY OF RELATED TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY |
| POPULATION IN THE EXTENSION PHASE)70 |
| TABLE 14.3.1.7D SUMMARY OF RELATED TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY |
| POPULATION IN THE STAGE 3 PK PHASE)70 |
| TABLE 14.3.1.8A SUMMARY OF TEAE LEADING TO TREATMENT DISCONTINUATION BY SOC AND PT (SAFETY |
| POPULATION IN THE STAGE 1 PK PHASE) |
| TABLE 14.3.1.8B SUMMARY OF TEAE LEADING TO TREATMENT DISCONTINUATION BY SOC AND PT (SAFETY |
| POPULATION IN THE STAGE 2 PK PHASE) |
| TABLE 14.3.1.8C SUMMARY OF TEAE LEADING TO TREATMENT DISCONTINUATION BY SOC AND PT (SAFETY |
| POPULATION IN THE EXTENSION PHASE) |
| TABLE 14.3.1.8D SUMMARY OF TEAE LEADING TO TREATMENT DISCONTINUATION BY SOC AND PT (SAFETY |
| POPULATION IN THE STAGE 3 PK PHASE) |
| TABLE 14.3.1.9C SUMMARY OF TEAE LEADING TO TREATMENT DOSE INTERRUPTION BY SOC AND PT (SAFETY |
| POPULATION IN THE EXTENSION PHASE) |
| POPULATION IN THE STAGE 1 PK PHASE) |
| TABLE 14.3.1.10B SUMMARY OF TEAE LEADING TO TREATMENT DOSE REDUCTION BY SOC AND PT (SAFETY |
| POPULATION IN THE STAGE 2 PK PHASE) |
| TABLE 14.3.1.10C SUMMARY OF TEAE LEADING TO TREATMENT DOSE REDUCTION BY SOC AND PT (SAFETY |
| POPULATION IN THE EXTENSION PHASE) 71 |
| TABLE 14.3.1.10D SUMMARY OF TEAE LEADING TO TREATMENT DOSE REDUCTION BY SOC AND PT (SAFETY |
| POPULATION IN THE STAGE 3 PK PHASE) |
| TABLE 14.3.1.11A SUMMARY OF TEAE LEADING TO DEATH BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 |
| PK PHASE)71 |
| TABLE 14.3.1.11B SUMMARY OF TEAE LEADING TO DEATH BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 |
| PK PHASE)71 |
| TABLE 14.3.1.11C SUMMARY OF TEAE LEADING TO DEATH BY SOC AND PT (SAFETY POPULATION IN THE |
| EXTENSION PHASE)71 |
Niraparib

| TABLE 14.3.1.14D SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY P1 (SAFETY F STAGE 3 PK PHASE) | |
|---|---|
| TABLE 14.3.1.15a LISTING OF SERIOUS TEAES DURING PK PHASE (SAFETY POPULATION IN 1 | |
| T 140 145 1 0 | |
| TABLE 14.3.1.15B LISTING OF SERIOUS TEAES DURING THE PK PHASE (SAFETY POPULATION PHASE) | |
| TABLE 14.3.1.15C LISTING OF SERIOUS TEAES DURING THE EXTENSION PHASE (SAFETY POP | ULATION IN THE |
| EXTENSION PHASE) | |
| TABLE 14.3.1.15D LISTING OF SERIOUS TEAES DURING THE PK PHASE (SAFETY POPULATION PHASE) | |
| TABLE 14.3.1.16a LISTING OF DEATHS DURING THE PK PHASE (SAFETY POPULATION IN THE | |
| TABLE 14.3.1.16B LISTING OF DEATHS DURING THE PK PHASE (SAFETY POPULATION IN THE STABLE 14.3.1.16B LISTING THE PK PHASE (SAFETY POPULATION IN THE STABLE 14.3.1.16B LISTING THE STABLE 14.3.1.16B LI | |
| TABLE 14.3.1.16c LISTING OF DEATHS DURING THE EXTENSION PHASE (SAFETY POPULATION | |
| PHASE) | |
| TABLE 14.3.1.16D LISTING OF DEATHS DURING THE PK PHASE (SAFETY POPULATION IN THE | |
| TABLE 14.3.1.17C LISTING OF TEAE LEADING TO DOSE INTERRUPTION DURING THE EXTENSI | |
| POPULATION IN THE EXTENSION PHASE) | |
| TABLE 14.3.1.17D LISTING OF TEAE LEADING TO DOSE INTERRUPTION DURING THE PK PHASE | |
| POPULATION IN THE STAGE 3 PK PHASE) | 78 |
| TABLE 14.3.1.18A LISTING OF TEAE LEADING TO DOSE REDUCTION DURING THE PK PHASE ( | (SAFETY POPULATION IN |
| THE STAGE 1 PK PHASE) | 78 |
| TABLE 14.3.1.18B LISTING OF TEAE LEADING TO DOSE REDUCTION DURING THE PK PHASE ( | (SAFETY POPULATION IN |
| THE STAGE 2 PK PHASE) | 78 |
| TABLE 14.3.1.18c LISTING OF TEAE LEADING TO DOSE REDUCTION DURING THE EXTENSION | PHASE (SAFETY |
| POPULATION IN THE EXTENSION PHASE) | |
| TABLE 14.3.1.18d LISTING OF TEAE LEADING TO DOSE REDUCTION DURING THE PK PHASE ( | |
| THE STAGE 3 PK PHASE) | |
| TABLE 14.3.1.19A LISTING OF TEAE LEADING TO TREATMENT DISCONTINUATION DURING THE | · |
| POPULATION IN THE STAGE 1 PK PHASE) | |
| TABLE 14.3.1.19B LISTING OF TEAE LEADING TO TREATMENT DISCONTINUATION DURING THE | |
| POPULATION IN THE STAGE 2 PK PHASE) | |
| TABLE 14.3.1.19C LISTING OF TEAE LEADING TO TREATMENT DISCONTINUATION DURING THE | |
| (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| TABLE 14.3.1.19d LISTING OF TEAE LEADING TO TREATMENT DISCONTINUATION DURING THE | * |
| POPULATION IN THE STAGE 3 PK PHASE) | |
| TABLE 14.3.1.16.1c ALL-CAUSE MORTALITY (SAFETY POPULATION IN THE EXTENSION PHASE | |
| TABLE 14.3.1.20D SUMMARY OF INCIDENCE OF COVID-19 RELATED ADVERSE EVENTS OVER | No. of the contract of the con |
| POPULATION IN THE STAGE 3 PK PHASE) | |
| TABLE 14.3.1.20c SUMMARY OF INCIDENCE OF COVID-19 RELATED ADVERSE EVENTS OVER | |
| POPULATION IN THE EXTENSION PHASE) | |
| TABLE 14.3.1.21D SUMMARY OF INCIDENCE OF COVID-19 RELATED ADVERSE EVENTS OVER | |
| (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| TABLE 14.3.1.22D SUMMARY OF INCIDENCE OF ADVERSE EVENTS OVER TIME BY AGE GROUP | |
| IN THE STAGE 3 PK PHASE) | |
| (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| TABLE 14.3.1.22c Summary of Incidence of Adverse Events Over Time by Age Group | |
| IN THE EXTENSION PHASE) | |
| · —, ····· | |

| LISTING 16.2.4.1B DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 106 |
|---|---|
| LISTING 16.2.4.1c DEMOGRAPHICS (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.4.1D DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.4.2A MEDICAL HISTORY (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.4.2B MEDICAL HISTORY (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.4.2c MEDICAL HISTORY (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.4.2D MEDICAL HISTORY (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.4.3A PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.4.3B PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.4.3C PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.4.3D PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.4.4a PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.4.4B PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.4.4c PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.4.4D PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.4.5A PRIOR/CONCOMITANT RADIOTHERAPY (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.4.5B PRIOR/CONCOMITANT RADIOTHERAPY (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.4.5c PRIOR/CONCOMITANT RADIOTHERAPY (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.4.5D PRIOR/CONCOMITANT RADIOTHERAPY (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.5.1B PRIOR AND CONCOMITANT MEDICATIONS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.5.1c PRIOR AND CONCOMITANT MEDICATIONS (SAFETY POPULATION IN THE EXTENSION PHASE). | |
| LISTING 16.2.5.10 PRIOR AND CONCOMITANT MEDICATIONS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.5.1.1c Treatment Exposure and Duration (Safety Population in the Extension Phase). | |
| LISTING 16.2.5.1.1C TREATMENT EXPOSORE AND DURATION (SAFETY FOR LATION IN THE EXTENSION FIRSE). LISTING 16.2.5.2A PRIOR/CONCOMITANT PROCEDURES DURING PK PHASE (SAFETY POPULATION IN THE STAGE | |
| PHASE) | |
| LISTING 16.2.5.2B PRIOR/CONCOMITANT PROCEDURES DURING THE PK PHASE (SAFETY POPULATION IN THE ST | |
| PK PHASE) | |
| LISTING 16.2.5.2c PRIOR/CONCOMITANT PROCEDURES DURING THE EXTENSION PHASE (SAFETY POPULATION IN | |
| EXTENSION PHASE) | |
| LISTING 16.2.5.2D PRIOR/CONCOMITANT PROCEDURES DURING THE PK PHASE (SAFETY POPULATION IN THE ST | |
| PK PHASE) | |
| LISTING 16.2.5.3A PRIOR AND CONCOMITANT TRANSFUSIONS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.5.3B PRIOR AND CONCOMITANT TRANSFUSIONS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.5.3C PRIOR AND CONCOMITANT TRANSFUSIONS (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.5.3D PRIOR AND CONCOMITANT TRANSFUSIONS (SAFETY POPULATION IN THE EXTENSION THASE) | |
| LISTING 16.2.5.4A PRIOR AND CONCOMITANT TRANSPOSIONS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 10.2.3.4AT RIOR AND CONCOMITANT GROWTH PACTORS (SAFETY TOPULATION IN THE STAGE LT & LE | 100 |
| LISTING 16.2.5.4B PRIOR AND CONCOMITANT GROWTH FACTORS (SAFETY POPULATION IN THE STAGE 2 PK PHA | |
| LISTING 10.2.3.461 RIOR AND CONCOMITANT GROWTH PACTORS (SAFETY I OPULATION IN THE STAGE 21 K I HA | |
| LISTING 16.2.5.4c PRIOR AND CONCOMITANT GROWTH FACTORS (SAFETY POPULATION IN THE EXTENSION PHA | |
| LISTING 10.2.5.7CT KIOK AND CONCOMITANT GROWTH PACTORS (SAFETT FOFULATION IN THE EXTENSION THA | |
| LISTING 16.2.5.4D PRIOR AND CONCOMITANT GROWTH FACTORS (SAFETY POPULATION IN THE STAGE 3 PK PHA | |
| LISTING 10.2.5.4D I KIOK AND CONCOMITANT GROWTH FACTORS (SAFETT FOR CLATION IN THE STAGE STREET | |
| LISTING 16.2.5.5A STUDY TREATMENT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.5.5A STUDY TREATMENT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.5.5C STUDY TREATMENT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.5.5C STUDY TREATMENT (SAFETY POPULATION IN THE EXTENSION PHASE) LISTING 16.2.5.5D STUDY TREATMENT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.5.6B SUBSEQUENT ANTI-CANCER THERAPY (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.5.6C SUBSEQUENT ANTI-CANCER THERAPY (SAFETY POPULATION IN THE EXTENSION PHASE) | 120 |

| LISTING 16.2.5.6D MEAL STATUS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 121 |
|---|---|
| $LISTING\ 16.2.6.1c\ Investigator\ Assessment\ of\ Response\ (Safety\ Population\ in\ the\ Extension\ Phase)$ | 122 |
| LISTING 16.2.7.1A ADVERSE EVENTS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 123 |
| LISTING 16.2.7.1B ADVERSE EVENTS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 123 |
| LISTING 16.2.7.1D ADVERSE EVENTS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 123 |
| LISTING 16.2.7.1C ADVERSE EVENTS (SAFETY POPULATION IN THE EXTENSION PHASE) | 124 |
| LISTING 16.2.7.2C ADVERSE EVENTS ONGOING FROM PK PHASE (SAFETY POPULATION IN THE EXTENSION PHASE) | SE)125 |
| LISTING 16.2.8.1.1A HEMATOLOGY RESULTS IN THE PK PHASE (SAFETY POPULATION IN THE STAGE 1 PK PHASE | E).126 |
| LISTING 16.2.8.1.1B HEMATOLOGY RESULTS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 126 |
| LISTING 16.2.8.1.1C HEMATOLOGY RESULTS (SAFETY POPULATION IN THE EXTENSION PHASE) | 126 |
| LISTING 16.2.8.1.1D HEMATOLOGY RESULTS THROUGH THE PK END OF TREATMENT VISIT (SAFETY POPULATION | N IN |
| THE STAGE 3 PK PHASE) | 126 |
| LISTING 16.2.8.1.2A CHEMISTRY RESULTS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 126 |
| LISTING 16.2.8.1.2B CHEMISTRY RESULTS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 126 |
| LISTING 16.2.8.1.2C CHEMISTRY RESULTS (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.8.1.2D CHEMISTRY RESULTS THROUGH THE PK END OF TREATMENT VISIT (SAFETY POPULATION | IN THE |
| STAGE 3 PK PHASE) | |
| LISTING 16.2.8.1.3A URINALYSIS RESULTS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.8.1.3B URINALYSIS RESULTS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.8.1.3C URINALYSIS RESULTS (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.8.1.3D URINALYSIS RESULTS THROUGH THE PK END OF TREATMENT VISIT (SAFETY POPULATION | |
| THE STAGE 3 PK PHASE) | |
| LISTING 16.2.8.1.4c LIVER FUNCTION TESTS – POTENTIAL HY'S LAW CASES (SAFETY POPULATION IN THE | |
| EXTENSION PHASE) | 128 |
| LISTING 16.2.8.2A VITAL SIGNS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.8.2B VITAL SIGNS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 129 |
| LISTING 16.2.8.2c VITAL SIGNS (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.8.2D VITAL SIGNS THROUGH THE PK END OF TREATMENT VISIT (SAFETY POPULATION IN THE STA | |
| PK Phase) | 129 |
| LISTING 16.2.8.3A ECG RESULTS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 130 |
| LISTING 16.2.8.3B ECG RESULTS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 130 |
| LISTING 16.2.8.3C ECG RESULTS (SAFETY POPULATION IN THE EXTENSION PHASE) | 130 |
| LISTING 16.2.8.3D ECG RESULTS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.8.4A ECOG PERFORMANCE STATUS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.8.4B ECOG PERFORMANCE STATUS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 131 |
| LISTING 16.2.8.4C ECOG PERFORMANCE STATUS (SAFETY POPULATION IN THE EXTENSION PHASE) | 131 |
| LISTING 16.2.8.4D ECOG PERFORMANCE STATUS THROUGH THE PK END OF TREATMENT VISIT (SAFETY | |
| POPULATION IN THE STAGE 3 PK PHASE) | 131 |
| LISTING 16.2.8.5A BASELINE PHYSICAL EXAMINATION FINDINGS (SAFETY POPULATION IN THE STAGE 1 PK PHA | |
| | 132 |
| LISTING 16.2.8.5B BASELINE PHYSICAL EXAMINATION FINDINGS (SAFETY POPULATION IN THE STAGE 2 PK PHA | ASE) |
| LISTING 16.2.8.5C BASELINE PHYSICAL EXAMINATION FINDINGS (SAFETY POPULATION IN THE EXTENSION PHA | SE) |
| LISTING 16.2.8.5D BASELINE PHYSICAL EXAMINATION FINDINGS (SAFETY POPULATION IN THE STAGE 3 PK PHA | |
| LISTING 16.2.8.6a PREGNANCY TEST (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 133 |
| LISTING 16.2.8.6B PREGNANCY TEST (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 133 |
| LISTING 16.2.8.6C PREGNANCY TEST (SAFETY POPULATION IN THE EXTENSION PHASE) | |

| • | | • • • | |
|---|------|-------|---|
| Ν | ıraı | oari | b |

# Statistical Analysis Plan

| LISTING 16.2.8.6D PREGNANCY TEST (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 133 |
|---|---|
| LISTING 16.2.9.2D LISTING OF COVID-19 ASSESSMENTS AND SYMPTOM ASSESSMENTS FOR PATIE | NTS WITH COVID- |
| 19 ADVERSE EVENTS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 134 |
| LISTING 16.2.9.2c LISTING OF COVID-19 ASSESSMENTS AND SYMPTOM ASSESSMENTS FOR PATIE | NTS WITH COVID- |
| 19 Adverse Events (Safety Population in the Extension Phase) | 135 |

# **TABLES**

# General guidelines:

Tables will be provided for the Stage 1 PK Phase, Stage 2 PK Phase, Stage 3 PK Phase and the Open-Label Extension Phase. For the PK Phase (Stage 1, Stage 2 and Stage 3):

- Treatment=Sequence and Overall, in general. For PK and AE data, please see mock tables.
- Population=Safety Population in Stage 1 PK (Stage 2 PK or Stage 3 PK) Phase, unless otherwise specified.
- PK Phase Data:
  - o For patients who do not continue to Extension Phase, PK Phase is any data collected.
  - o For patients who do continue to Extension Phase,
    - AEs prior to first dose in Extension Phase
    - Prior meds/procedures/etc. prior to first dose in PK Phase
    - Concomitant meds meds prior to first dose in Extension Phase.
- Assessments (Labs, ECGs, Vitals, ECOG, PE, etc.) use visit to identify data.

# For the Extension Phase:

- Treatment=Niraparib Tablet or Capsule (regardless of starting dose); Summarize by Tablet; Capsule; Overall, unless otherwise specified.
- Population=Safety Population in the Open-Label Extension Phase (i.e., those who receive at least 1 dose), unless otherwise specified.
- Extension Phase Data:
  - o For patients who do not continue to Extension Phase, there is no Extension Phase data.
  - o For patients who do continue to Extension Phase,
    - AEs on or after first dose in Extension Phase
    - Prior meds/procedures/etc. prior to first dose in Extension Phase
    - Concomitant meds meds on or after the first dose in Extension Phase
    - Assessments (Labs, ECGs, Vitals, ECOG, PE, etc.) use visit to identify data.

Sort order: All AE tabulations, unless otherwise specified, will be ordered in terms of decreasing frequency for SOC (alphabetically for SOCs with the same number of AEs reported), and decreasing frequency for PT within SOC (alphabetically for PTs with the same number of AEs reported within a SOC) considering the overall rate.


TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Table 14.1.1a

Subject Disposition in the PK Phase (All Patients in the Stage 1 PK Phase)

| Parameter | Statistic | Sequence<br>TABLET/CAPSULE | Sequence<br>CAPSULE/TABLET | Overall |
|---|---|---|---|---|
| Number of Patients | | | | |
| Screened | n | | | xx |
| Randomized | n | Х | Х | х |
| Received Tablet | n | Х | х | х |
| Received Capsule | n | Х | Х | х |
| Received Both Tablet and Capsule | n | Х | х | х |
| PK Phase Safety Population | n | Х | Х | Х |
| Completed PK Phase | n | X | Х | X |
| Discontinuation from PK Phase | n | Х | X | X |
| Reason1 | n | Х | X | Х |
| Reason2 | n | Х | Х | Х |
| Participate in Extension Phase | n | X | X | X |
| rareterpace in Execusion rhase | 11 | Λ | Α | A |
| Discontinuation from Study Prior to Entering the Extension Phase | | | | |
| Reason1 | n | XX | XX | XX |
| Reason2 | n | XX | XX | XX |

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# [Programming Notes]

Only include DC from study for those patients who do not enter the Extension Phase.

Protocol: XXXXX

Table 14.1.1b

Subject Disposition in the PK Phase (All Patients in the Stage 2 PK Phase)

| Parameter | Statistic | Sequence<br>TABLET/CAPSULE | Sequence<br>CAPSULE/TABLET | Overall |
|---|---|---|---|---|
| Number of Patients | | | | |
| Screened | n | | | XX |
| Randomized | n | Х | Х | Х |
| Not Treated | n | Х | Х | Х |
| Received Tablet | n | Х | Х | Х |
| Received Capsule | n | Х | Х | Х |
| Received Both Tablet and Capsule | n | Х | Х | Х |
| PK Phase Safety Population | n | Х | Х | Х |
| Completed PK Phase | n | Х | Х | Х |
| Discontinuation from PK Phase [1] | n | Х | Х | X |
| Reason 1 | n | Х | Х | X |
| Reason 2 | n | Х | Х | X |
| Participate in Extension Phase | n | Х | Х | X |
| Discontinuation from Study Prior to Entering the Extension Phase | | | | |
| Reason 1 | n | XX | XX | XX |
| Reason 2 | n | XX | XX | XX |

[1] Includes patients in the Safety Population (i.e., treated patients) only.

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

[Programming Notes]

Only include DC from study for those patients who do not enter the Extension Phase.

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

#### Table 14.1.1c

Subject Disposition in the Extension Phase (All Patients in the Extension Phase)

| Parameter | Statistic | TABLET | CAPSULE | OVERALL |
|---|---|---|---|---|
| Number of Patients | | | | |
| Dosed | n | xx | xx | XX |
| By Stage: | | | | |
| Dosed in Stage 1 | n (%) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Dosed in Stage 2 | n (%) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Dosed in Stage 3 | n (%) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| By Starting Dose: | | | | |
| 100mg/d | n (%) | xx (xx.x) | xx ( xx.x) | xx ( xx.x) |
| 200mg/d | n (%) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| 300mg/d | n (%) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Discontinued Treatment After Receiving at Least 1 Dose | n | XX | XX | XX |
| Reason 1 | n | xx | xx | xx |
| Reason 2 | n | XX | XX | XX |
| Discontinued Study | n | XX | XX | XX |
| Reason 1 | n | XX | XX | XX |
| Reason 2 | n | xx | XX | XX |

NOTE: The starting dose of 100 mg/day was selected based on Investigator decision.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


Protocol: XXXXX

### Table 14.1.1d

Subject Disposition in the PK Phase (All Patients in the Stage 3 PK Phase)

| Parameter | Statistic | Sequence<br>NIRAPARIB TABLET<br>FASTED/FED | Sequence<br>NIRAPARIB TABLET<br>FED/FASTED | OVERALL |
|---|---|---|---|---|
| Number of Patients | | | | |
| Screened [1] | n | | | XX |
| Randomized | n | Х | Х | Х |
| Not Treated | n | Х | Х | Х |
| Received Tablet in Fasted State | n | Х | Х | Х |
| Received Tablet in Fed State | n | X | X | Х |
| Received Tablet in Both Fasted and Fed State | n | Х | X | X |
| PK Phase Safety Population | n | Х | х | X |
| Completed PK Phase | n | х | Х | Х |
| Discontinuation from PK Phase [2] | n | Х | Х | X |
| Reason 1 | n | Х | х | X |
| Reason 2 | n | Х | х | X |
| Participate in Extension Phase | n | Х | Х | Х |
| Discontinuation from Study Prior to Entering the Extension Phase | | | | |
| Reason 1 | n | XX | XX | XX |
| Reason 2 | n | xx | xx | XX |

<sup>[1]</sup> Patient xxxxxx-xxxx (Screen Failure ID: XXi) and xxxxxx-xxxx (Screen Failure ID: YYi) re-screened and reconsented after screen failure are counted twice in Screening.

# [Programming Note]

XXi/YYi is ID that was SF.

Programming, please note footnote references changed order in the shell and footer.

<sup>[2]</sup> Includes patients in the Safety Population (i.e., treated patients) only.

Protocol: XXXXX

#### Table 14.1.2a

Demographics (Safety Population in the Stage 1 PK Phase)

| Parameter | Statistic | Sequence | Sequence | |
|---|---|---|---|---|
| | | TABLET/CAPSULE | CAPSULE/TABLET | OVERALL |
| | | (N=xx) | (N=xx) | (N=xx) |
| Age (yrs) | n | XX | XX | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| 2 | | | | |
| Age Group | (0) | | | , , |
| 18 -< 65 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 65 -< 75 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ≥ 75 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sex | | | | |
| Male | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race | | | | |
| White | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| African American | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| American Indian or Alaska Native | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Native Hawaiian or other Pacific Islander | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity | | | | 1 |
| Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | · · · · · | , , |
| Not Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# Repeat for:

Table 14.1.2.1a Demographics (BA Evaluable Population in the Stage 1 PK Phase)

Table 14.1.2.1b Demographics (Safety Population in the Stage 2 PK Phase)

Table 14.1.2.2b Demographics (BE Evaluable Population in the Stage 2 PK Phase)

Table 14.1.2c Demographics (Safety Population in the Extension Phase)

- Summarize Extension Phase Data with columns for TABLET; CAPSULE; OVERALL.
- Add footnote: "Note: Age was collected at PK Phase entry only."

Table 14.1.2.1d Demographics (Safety Population in the Stage 3 PK Phase)

Table 14.1.2.2d Demographics (FE Evaluable Population in the Stage 3 PK Phase)

• Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL.


Protocol: XXXXX

# Table 14.1.3a

Baseline Characteristics (Safety Population in the Stage 1 PK Phase)

| Parameter | Statistic | Sequence<br>TABLET/CAPSULE | Sequence<br>CAPSULE/TABLET | OVERALL |
|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) |
| Weight (kg) | n | xx | xx | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | XX.X |
| | Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Min, Max | XX, XX | XX, XX | xx, xx |
| Height (cm) | n | XX | XX | XX |
| neight (Chi) | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | 11111, 111111 | , | , | , |
| BMI (kg/m²) | n | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| ECOG Performance Status | | | | |
| 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

ECOG = Eastern Cooperative Oncology Group:

0=Fully active, able to carry on all pre-disease performance without restriction

1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature

2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours

3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours

4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Table 14.1.3.1a Baseline Characteristics (BA Evaluable Population in the Stage 1 PK Phase)


Table 14.1.3.1b Baseline Characteristics (Safety Population in the Stage 2 PK Phase)

Table 14.1.3.2b Baseline Characteristics (BE Evaluable Population in the Stage 2 PK Phase)

Table 14.1.3c Baseline Characteristics (Safety Population in the Extension Phase)

- Summarize Extension Phase Data with columns for TABLET; CAPSULE; OVERALL.
- Add footnote for Extension Phase and relevant reference in the table:
- [1] Only weight and ECOG Performance Status were repeated at Extension Phase entry.

Table 14.1.3.1d Baseline Characteristics (Safety Population in the Stage 3 PK Phase)

- Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL Table 14.1.3.2d Baseline Characteristics (FE Evaluable Population in the Stage 3 PK Phase)
- Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Table 14.1.4a

### Primary Cancer History (Safety Population in the Stage 1 PK Phase)

| Parameter | Statistic | Sequence<br>TABLET/CAPSULE | Sequence<br>CAPSULE/TABLET | OVERALL |
|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) |
| Tumor Type | | | | |
| Xxxxxxx | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Xxxxxxx | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Xxxxxxx | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time from first diagnosis to informed consent (years) | n | XX | XX | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Cancer Stage (most recent) | | | | |
| Locally advanced | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Metastatic | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of prior lines of therapy | | | | |
| 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=6 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any prior radiotherapy | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# Repeat for:

Table 14.1.4b Primary Cancer History (Safety Population in the Stage 2 PK Phase)

Table 14.1.4c Primary Cancer History (Safety Population in the Extension Phase)

- Summarize Extension Phase Data with columns for TABLET; CAPSULE; OVERALL.
- Table 14.1.4d Primary Cancer History (Safety Population in the Stage 3 PK Phase)
- Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL

|-----------------|
| Protocol: XXXXX |

Table 14.1.5a

Prior Anti-Cancer Treatment (Safety Population in the Stage 1 PK Phase)

| Preferred Term | Statistic | Sequence<br>TABLET/CAPSULE<br>(N=xx) | Sequence<br>CAPSULE/TABLET<br>(N=xx) | OVERALL<br>(N=xx) |
|---|---|---|---|---|
| Agent 1 | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Agent 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Agent 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

Sort by decreasing frequency in the OVERALL column.

#### Repeat for:

Table 14.1.5b Prior Anti-Cancer Treatment (Safety Population in the Stage 2 PK Phase)

Table 14.1.5c Prior Anti-Cancer Treatment (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for TABLET; CAPSULE; OVERALL.

Table 14.1.5d Prior Anti-Cancer Treatment (Safety Population in the Stage 3 PK Phase)

Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED AND OVERALL.

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Table 14.1.6a

Medical History (Safety Population in the Stage 1 PK Phase)

| System Organ Class | Statistic | Sequence | Sequence | |
|--------------------|-----------|----------------|----------------|-----------|
| Preferred Term | | TABLET/CAPSULE | CAPSULE/TABLET | OVERALL |
| | | (N=xx) | (N=xx) | (N=xx) |
| Any condition | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

[Programming Notes]

Sort alphabetically by SOC/PT.

#### Repeat for:

Table 14.1.6b Medical History (Safety Population in the Stage 2 PK Phase)

Table 14.1.6c Medical History and Prior Blood Disorders (Safety Population in the Extension Phase)

- Summarize Extension Phase Data with columns for TABLET; CAPSULE; OVERALL.
- Add footnote: "Note: The table summarizes combined data from Medical History and Prior Blood Disorders eCRFs. Duplicate events reported across both eCRFs are counted only once per patient in this table."

Table 14.1.6d Medical History (Safety Population in the Stage 3 PK Phase)

• Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Table 14.1.7a

Prior Medications by ATC and PT (Safety Population in the Stage 1 PK Phase)

| ATC (Level 3) | Statistic | Sequence | Sequence | |
|---|---|---|---|---|
| Preferred Term | | TABLET/CAPSULE | CAPSULE/TABLET | OVERALL |
| | | (N=xx) | (N=xx) | (N=xx) |
| Any prior medication | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC1 | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Prior medications are any medications with a start date earlier than the first dose date of study treatment and are coded using WHO Drug Dictionary version YYYYMM. Study treatment, prior anti-cancer treatments for primary cancer, transfusions and growth factors are not included.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

Sort alphabetically by ATC3 and Preferred Term. If there are uncoded terms due to no ATC level 3 term not being available, add footnote for uncoded term: [1] ATC level 3 term is not available through WHO Drug Dictionary.

#### Repeat for:

Table 14.1.7b Prior Medications by ATC and PT (Safety Population in the Stage 2 PK Phase)

Table 14.1.7c Prior Medications by ATC and PT (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for TABLET; CAPSULE; OVERALL.

#### [Programming Notes]

- Footnote Extension Phase: Prior medications are any medications, other than study treatments and pre-medications for study treatment, with a start date earlier than the first dose date of study treatment during the Extension Phase and are coded using WHO Drug Dictionary version YYYYMM.
- Prior anti-cancer treatments for primary cancer are not included.

Table 14.1.7d Prior Medications by ATC and PT (Safety Population in the Stage 3 PK Phase)

Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL.

Protocol: XXXXX

#### Table 14.1.8a

Concomitant Medications by ATC and PT (Safety Population in the Stage 1 PK Phase)

| ATC (Level 3) | Statistic | Sequence | Sequence | |
|---|---|---|---|---|
| Preferred Term | | TABLET/CAPSULE | CAPSULE/TABLET | OVERALL |
| | | (N=xx) | (N=xx) | (N=xx) |
| Any concomitant medication | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Concomitant medications are any medications being taken on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase. They are coded using WHO Drug Dictionary version YYYYMM.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

Sort alphabetically by ATC3 and Preferred Term. If there are uncoded terms due to no ATC level 3 term not being available, add footnote for uncoded term: [1] ATC level 3 term is not available through WHO Drug Dictionary.

#### Repeat for:

Table 14.1.8.1b Concomitant Medications by ATC and PT (Safety Population in the Stage 2 PK Phase)

Table 14.1.8.2b Concomitant Medications During the PK Collection Period by ATC and PT (BE Evaluable Population in the Stage 2 PK Phase)

• Footnote: Concomitant medications during the PK collection period are any concomitant medications taken between the first PK-draw until the last PK-draw. They are coded using WHO Drug Dictionary version YYYYMM.

Table 14.1.8c Concomitant Medications by ATC and PT (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for TABLET; CAPSULE; OVERALL.

#### [Programming Notes]

- Footnote Extension Phase: Concomitant medications are any medications being taken on or after the initial study treatment dosing date during the Extension Phase through 30 days after the last dose. They are coded using WHO Drug Dictionary version YYYYMM.

  Table 14.1.8d Concomitant Medications by ATC and PT (Safety Population in the Stage 3 PK Phase)
- Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL
- Footnote Stage 3: Concomitant medications are any medications being taken on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase. They are coded using WHO Drug Dictionary version YYYYMM.

Protocol: XXXXX

Table 14.1.9a

Concomitant Transfusions and Growth Factors (Safety Population in the Stage 1 PK Phase)

| Parameter | Statistic | Sequence | Sequence | |
|---|---|---|---|---|
| | | TABLET/CAPSULE | CAPSULE/TABLET | OVERALL |
| | | (N=xx) | (N=xx) | (N=xx) |
| Any Concomitant Transfusions | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Red Blood Cells | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Platelet | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Concomitant Growth Factors | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| G-CSF | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GM-CSF | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Recombinant Erythropoietin | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Concomitant transfusions or growth factors are any transfusion or growth factor given on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose for those not continuing into the Extension Phase.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Table 14.1.9b Concomitant Transfusions and Growth Factors (Safety Population in the Stage 2 PK Phase)

Table 14.1.9c Concomitant Transfusions and Growth Factors (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for TABLET; CAPSULE; OVERALL.

#### [Programming Notes]

• Footnote - Extension Phase: Concomitant transfusions or growth factors are any transfusion or growth factor given on or after the initial study treatment dosing date during the Extension Phase through 30 days after the last dose.

Table 14.1.9d Concomitant Transfusions and Growth Factors (Safety Population in the Stage 3 PK Phase)

- Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL
- Footnote Stage 3: Concomitant transfusions or growth factors are any transfusion or growth factor given on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose for those not continuing into the Extension Phase.

Protocol: XXXXX

Table 14.1.10c

Summary of Investigator-Assessed Best Response by Tumor Type (Safety Population in the Extension Phase)

| Treatment: <tablet, capsule=""></tablet,> | (N=xx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Investigato | r Assessment | | |
| | Complete | Partial | Stable Disease | Progressive | Not Evaluable | |
| Tumor type [1] | Response (CR) | Response (PR) | (SD) | Disease (PD) | (NE) | Total [2] |
| Prostate Cancer | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mesothelioma Malignant | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Duodenal Adenocarcinoma | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Colon Cancer | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Malignant Melanoma | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| • • • | | | | | | |
| Other: xxx | | | | | | |
| Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N=Number of patients in Safety Population.

Note: 'Total' represents the number of patients with non-missing investigator assessment.

- [1] The percentages are based on row totals.
- [2] The percentages are based on overall response totals.

#### [Programming Notes]

Present by decreasing order of total frequency of tumor types observed, in the event of tie, sort in alphabetical order. If better fit requires taking Treatment out into the header row, split table across pages with each treatment on a new page.


Table 14.3.1.1.1a

Overall Summary of Treatment Emergent Adverse Events (Safety Population in the Stage 1 PK Phase)

| | TABLET [1] | CAPSULE [2] | FU/Ext Screening | Total [4] |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | [3] (N=xx) | (N=xx) |
| Any Treatment Emergent Adverse Event (TEAE) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Reduction | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib capsules.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

Repeat for:

TESARO, Inc.

Protocol: XXXXX

Table 14.3.1.1.1b Overall Summary of Treatment Emergent Adverse Events (Safety Population in the Stage 2 PK Phase)


Protocol: XXXXX

#### Table 14.3.1.1.1c

Overall Summary of Treatment Emergent Adverse Events (Safety Population in the Extension Phase)

| | TABLET | CAPSULE | OVERALL |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| Any Treatment Emergent Adverse Event (TEAE) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Reduction | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Death | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any COVID-19 related TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: This table reports Treatment Emergent Adverse Events (TEAEs) with onset during Extension Phase only.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### [Programming Notes]

• Sort order: All AE tabulations, unless otherwise specified, will be ordered in terms of decreasing frequency for SOC (alphabetically for SOCs with the same number of AEs reported), and decreasing frequency for PT within SOC (alphabetically for PTs with the same number of AEs reported within a SOC) considering the overall rate.

#### Repeat for:

Table 14.3.1.1.1.1c Overall Summary of Treatment Emergent Adverse Events Ongoing from PK Phase (Safety Population in the Extension Phase)

[Programming Notes for Table 14.3.1.1.1.1c]

Footnote: "Note: This table reports Treatment Emergent Adverse Events (TEAEs) with onset during PK Phase of the study.

This table summarizes data from Listing 16.2.7.2c, please use this listing as source reference in the footnote.


Protocol: XXXXX Table 14.3.1.1.1d

TESARO, Inc.

Overall Summary of Treatment Emergent Adverse Events (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB | NIRAPARIB | FU/Ext | |
|---|---|---|---|---|
| | | | - / - | |
| | TABLET FASTED [1] | TABLET FED [2] | Screening [3] | Total [4] |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any Treatment Emergent Adverse Event (TEAE) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Reduction | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any COVID-19 related TEAE Leading to Treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinuation | | | | |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


Protocol: XXXXX

#### Table 14.3.1.1.2a

Overall Summary of Treatment Emergent Adverse Events by Sequence and Period (Safety Population in the Stage 1 PK Phase)

| | | Sequence | | | Sequence | |
|---|---|---|---|---|---|---|
| | TABLET/CAPSULE | | | CAPSULE/TABLET | | |
| | | (N=xx) | | | (N=xx) | |
| | TABLET | CAPSULE | FU/Ext | CAPSULE | TABLET | FU/Ext |
| | Period 1 | Period 2 | Screening | Period 1 | Period 2 | Screening |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any Treatment Emergent Adverse Event (TEAE) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Reduction | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE Leading to Treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinuation | | | | | | |
| Any TEAE Leading to Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

 $\texttt{Source: Program: XXXXXXXXXXXXXXXXXXXXX}. \ \ \texttt{Output: xxxxxxxxxxxxxxxx.rtf.} \ \ \texttt{Generated on DDMMMYYYY:HH:MM:SS}$ 

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Table 14.3.1.1.2b Overall Summary of Treatment Emergent Adverse Events by Sequence and Period (Safety Population in the Stage 2 PK Phase)


TESARO, Inc. Protocol: XXXXX

Table 14.3.1.1.2d


Overall Summary of Treatment Emergent Adverse Events by Sequence and Period (Safety Population in the Stage 3 PK Phase)

| | Sequence | | | Sequence | | |
|---|---|---|---|---|---|---|
| | NIRAPARIB TABLET FASTED/FED | | | NIRAPARIB TABLET FED/FASTED | | |
| | (N=xx) | | | (N=xx) | | |
| | NIRAPARIB | NIRAPARIB | | NIRAPARIB | | |
| | TABLET | TABLET | | TABLET | NIRAPARIB | |
| | FASTED | FED | FU/Ext | FED | TABLET FASTED | FU/Ext |
| | Period 1 | Period 2 | Screening | Period 1 | Period 2 | Screening |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any Treatment Emergent Adverse Event (TEAE) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE with CTCAE Toxicity Grade ≥ | | | | | | |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Reduction | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE Leading to Treatment | | | | | | |
| Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any COVID-19 related TEAE Leading to | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment Discontinuation | | | | | | |

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Table 14.3.1.2.1a

Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 1 PK Phase)

| System Organ Class<br>Preferred Term | TABLET [1] (N=xx) | CAPSULE [2]<br>(N=xx) | FU/Ext Screening [3] (N=xx) | Total [4]<br>(N=xx) |
|---|---|---|---|---|
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib capsules.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

Niraparib

Protocol: XXXXX

For all tables of adverse events by SOC and PT, sort SOCs by descending overall frequency of events reported. Within each SOC, sort PTs by descending overall frequency of events reported.

Table 14.3.1.2.1b Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 2 PK Phase)

Protocol: XXXXX

#### Table 14.3.1.2.1c

Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Extension Phase)

| System Organ Class | TABLET | CAPSULE | OVERALL |
|--------------------|-----------|-----------|-----------|
| Preferred Term | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2021 | | ( ) | |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# [Programming Notes]

For all tables of adverse events by SOC and PT, sort SOCs by descending overall frequency of events reported. Within each SOC, sort PTs by descending overall frequency of events reported.


#### Table 14.3.1.2.1d

Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB | NIRAPARIB | FU/Ext | |
|---|---|---|---|---|
| System Organ Class | TABLET FASTED [1] | TABLET FED [2] | Screening [3] | Total [4] |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

Protocol: XXXXX

For all tables of adverse events by SOC and PT, sort SOCs by descending overall frequency of events reported. Within each SOC, sort PTs by descending overall frequency of events reported.

Protocol: XXXXX

# Table 14.3.1.2.1.1d

Summary of COVID-19 related Adverse Events by SOC and PT (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB | NIRAPARIB | FU/Ext | |
|---|---|---|---|---|
| System Organ Class | TABLET FASTED [1] | TABLET FED [2] | Screening [3] | Total [4] |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: COVID-19 Case Diagnosis is based on WHO Definition as of DDMMMYYYY.

- [1] Includes COVID-19 related TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes COVID-19 related TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes COVID-19 related TEAEs occurring at any time during the PK Phase.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

For all tables of adverse events by SOC and PT, sort SOCs by descending overall frequency of events reported. Within each SOC, sort PTs by descending overall frequency of events reported.

Select only COVID-19 related TEAEs.

Protocol: XXXXX

#### Table 14.3.1.2.2a

Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 1 PK Phase)

| | | Sequence<br>TABLET/CAPSULE<br>(N=xx) | | | Sequence<br>CAPSULE/TABLET<br>(N=xx) | |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | TABLET Period 1 (N=xx) | CAPSULE<br>Period 2<br>(N=xx) | FU/Ext<br>Screening<br>(N=xx) | CAPSULE<br>Period 1<br>(N=xx) | TABLET Period 2 (N=xx) | FU/Ext<br>Screening<br>(N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1<br>PT 1 | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2<br>PT 1 | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |

# [Programming Notes]

For tables of adverse events by SOC and PT by sequence and period, sort alphabetically by SOCs and PTs.

Table 14.3.1.2.2b Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 2 PK Phase)

Protocol: XXXXX

# Table 14.3.1.2.2d

Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 3 PK Phase)

| NIRAPARI NIRAPARIB BLET FASTED Period 1 (N=xx) xx (xx.x) | RIB TABLET FASTI<br>(N=xx)<br>NIRAPARIB<br>TABLET FED<br>Period 2<br>(N=xx) | ED/FED FU/Ext Screening (N=xx) | NIRAPARIB<br>TABLET FASTED<br>Period 1 | ARIB TABLET FED/F. (N=xx) NIRAPARIB TABLET FED Period 2 | ASTED FU/Ext Screening |
|---|---|---|---|---|---|
| BLET FASTED Period 1 (N=xx) | NIRAPARIB<br>TABLET FED<br>Period 2<br>(N=xx) | Screening | TABLET FASTED Period 1 | NIRAPARIB<br>TABLET FED | · · |
| BLET FASTED Period 1 (N=xx) | TABLET FED Period 2 (N=xx) | Screening | TABLET FASTED Period 1 | TABLET FED | · · |
| Period 1<br>(N=xx) | Period 2<br>(N=xx) | Screening | Period 1 | | · · |
| (N=xx) | (N=xx) | _ | | Period 2 | Screening |
| , , | · · · · · · | (N=xx) | (37) | | |
| xx (xx.x) | | 1 ' | (N=xx) | (N=xx) | (N=xx) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| / \ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | | (x (xx.x) | (xx (xx.x) | xx (xx.x) | (xx (xx.x) |

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# [Programming Notes]

For tables of adverse events by SOC and PT by sequence and period, sort alphabetically by SOCs and PTs.

```
Using Mock Shell (Table 14.3.1.2.1a, Table 14.3.1.2.1b, Table 14.3.1.2.1c, Table 14.3.1.2.1d)
Repeat for:
Table 14.3.1.3a Summary of Related TEAE by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.3b Summary of Related TEAE by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.3c Summary of Related TEAE by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.3d Summary of Related TEAE by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.4a Summary of Serious TEAE by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.4b Summary of Serious TEAE by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.4c Summary of Serious TEAE by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.4d Summary of Serious TEAE by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.5a Summary of Related Serious TEAE by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.5b Summary of Related Serious TEAE by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.5c Summary of Related Serious TEAE by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.5d Summary of Related Serious TEAE by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.6a Summary of TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.6b Summary of TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.6c Summary of TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.6d Summary of TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.7a Summary of Related TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.7b Summary of Related TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.7c Summary of Related TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.7d Summary of Related TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.8a Summary of TEAE Leading to Treatment Discontinuation by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.8b Summary of TEAE Leading to Treatment Discontinuation by SOC and PT (Safety Population in the Stage 2 PK Phase)
```


```
Table 14.3.1.8c Summary of TEAE Leading to Treatment Discontinuation by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.8d Summary of TEAE Leading to Treatment Discontinuation by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.9c Summary of TEAE Leading to Treatment Dose Interruption by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.10a Summary of TEAE Leading to Treatment Dose Reduction by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.10b Summary of TEAE Leading to Treatment Dose Reduction by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.10c Summary of TEAE Leading to Treatment Dose Reduction by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.10d Summary of TEAE Leading to Treatment Dose Reduction by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.11a Summary of TEAE Leading to Death by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.11b Summary of TEAE Leading to Death by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.11c Summary of TEAE Leading to Death by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.11d Summary of TEAE Leading to Death by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.11.1a Summary of Related TEAE Leading to Death by SOC and PT (Safety Population in the Stage 1 PK Phase)
   [Programming notes] - TABLE FOR PLAIN TEXT SUMMARY PURPOSES ONLY.
Table 14.3.1.11.1b Summary of Related TEAE Leading to Death by SOC and PT (Safety Population in the Stage 2 PK Phase)
  [Programming notes] - TABLE FOR PLAIN TEXT SUMMARY PURPOSES ONLY.
Table 14.3.1.11.1c Summary of Related TEAE Leading to Death by SOC and PT (Safety Population in the Extension Phase)
   [Programming notes] - TABLE FOR PLAIN TEXT SUMMARY PURPOSES ONLY.
```

Table 14.3.1.11.1d Summary of Related TEAE Leading to Death by SOC and PT (Safety Population in the Stage 3 PK Phase)

[Programming notes] - TABLE FOR PLAIN TEXT SUMMARY PURPOSES ONLY.

Table 14.3.1.12a Summary of Treatment Emergent AESI by SOC and PT (Safety Population in the Stage 1 PK Phase)

Table 14.3.1.12b Summary of Treatment Emergent AESI by SOC and PT (Safety Population in the Stage 2 PK Phase)

Table 14.3.1.12c Summary of Treatment Emergent AESI by SOC and PT (Safety Population in the Extension Phase)

Table 14.3.1.12d Summary of Treatment Emergent AESI by SOC and PT (Safety Population in the Stage 3 PK Phase)


- Table 14.3.1.23.1a Summary of Non-Serious TEAE (≥5%) by SOC and PT (Safety Population in the Stage 1 PK Phase)

  [Programming notes] TABLE FOR DISCLOSURE PURPOSES ONLY.
- Table 14.3.1.23.1b Summary of Non-Serious TEAE (≥5%) by SOC and PT (Safety Population in the Stage 2 PK Phase)

  [Programming notes] TABLE FOR DISCLOSURE PURPOSES ONLY.
- Table 14.3.1.23.1c Summary of Non-Serious TEAE (≥5%) by SOC and PT (Safety Population in the Extension Phase)

  [Programming notes] TABLE FOR DISCLOSURE PURPOSES ONLY.
- Table 14.3.1.23.1d Summary of Non-Serious TEAE (≥5%) by SOC and PT (Safety Population in the Stage 3 PK Phase)

  [Programming notes] TABLE FOR DISCLOSURE PURPOSES ONLY.
- Table 14.3.1.23.2a Summary of Related Non-Serious TEAE by SOC and PT (Safety Population in the Stage 1 PK Phase)

  [Programming notes] TABLE FOR PLAIN TEXT SUMMARY PURPOSES ONLY.
- Table 14.3.1.23.2b Summary of Related Non-Serious TEAE by SOC and PT (Safety Population in the Stage 2 PK Phase)

  [Programming notes] TABLE FOR PLAIN TEXT SUMMARY PURPOSES ONLY.
- Table 14.3.1.23.2c Summary of Related Non-Serious TEAE by SOC and PT (Safety Population in the Extension Phase)

  [Programming notes] TABLE FOR PLAIN TEXT SUMMARY PURPOSES ONLY.
- Table 14.3.1.23.2d Summary of Related Non-Serious TEAE by SOC and PT (Safety Population in the Stage 3 PK Phase)

  [Programming notes] TABLE FOR PLAIN TEXT SUMMARY PURPOSES ONLY.

Protocol: XXXX

Table 14.3.1.13a

Summary of Treatment Emergent Adverse Events by SOC and PT and CTCAE Toxicity Grade (Safety Population in the Stage 1 PK Phase)

| | | | FU/Ext | |
|--------------------|------------|-------------|---------------|-----------|
| System Organ Class | TABLET [1] | CAPSULE [2] | Screening [3] | Total [4] |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Grade 1 | | | | |
| ••• | | | | |
| Grade 5 | | | | |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Grade 1 | | | | |
| • • • | | | | |
| Grade 5 | | | | |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Grade 1 | | | | |
| • • • | | | | |
| Grade 5 | | | | |
| ••• | | | | |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib capsules.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Table 14.3.1.13b Summary of Treatment Emergent Adverse Events by SOC and PT and Maximum Toxicity (Safety Population in the Stage 2 PK Phase)

Table 14.3.1.13c Summary of Treatment Emergent Adverse Events by SOC and PT and Maximum Toxicity (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for TABLET; CAPSULE; OVERALL.

### [Programming Notes]

For all tables of adverse events by SOC and PT, sort SOCs by descending overall frequency of events reported. Within each SOC, sort PTs by descending overall frequency of events reported. Within each PT, sort by presented maximum toxicity grade.

# Confidential

Protocol: XXXX Table 14.3.1.13d

TESARO, Inc.

Summary of Treatment Emergent Adverse Events by SOC and PT and CTCAE Toxicity Grade (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB | NIRAPARIB | FU/Ext | |
|---|---|---|---|---|
| System Organ Class | TABLET FASTED [1] | TABLET FED [2] | Screening [3] | Total [4] |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| • • • | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| Grade 5 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| Grade 5 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| ••• | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| Grade 5 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


Protocol: XXXXX

Table 14.3.1.14a

Summary of Treatment Emergent Adverse Events by PT (Safety Population in the Stage 1 PK Phase)

| | TABLET [1] | CAPSULE [2] | FU/Ext Screening [3] | Total [4] |
|----------------|------------|-------------|----------------------|-----------|
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib capsules.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Repeat for:

Table 14.3.1.14b Summary of Treatment Emergent Adverse Events by PT (Safety Population in the Stage 2 PK Phase)

Table 14.3.1.14c Summary of Treatment Emergent Adverse Events by PT (Safety Population in the Extension Phase)

- Summarize Extension Phase Data with columns for TABLET; CAPSULE; OVERALL.
- [1], [2], [3] and [4] are not applicable.

[Programming Notes]

Sort PTs by descending overall frequency of events reported.

Protocol: XXXXX

Table 14.3.1.14d

Summary of Treatment Emergent Adverse Events by PT (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB | NIRAPARIB | FU/Ext | |
|---|---|---|---|---|
| Preferred Term | TABLET FASTED [1] | TABLET FED [2] | Screening [3] | Total [4] |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | | | | |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxxrtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

Protocol: XXXXX

Table 14.3.1.15a

Listing of Serious TEAEs During PK Phase (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| | | | Start | Stop | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Date | Date | | | | | | | |
| | | | Time/ | Time | | | | | | | |
| | Dosing Period/ | Adverse Event | (Rel | (Rel | | SAE/ | | Action Taken | Other | | |
| Patient | Niraparib | [P]MedDRA Preferred Term | Day | Day | | Reason | | on Study | Action | Relationship | |
| Number | Treatment | [S]System Organ Class | [1]) | [1]) | TEAE? | [2] | Severity | Treatment[3] | Taken | [3] | Outcome |
| | Period 1/ | XXXXXXXXXXXXX | уууу- | уууу- | Y | N | Grade 1 | T: NA | | T: NA | Recovered/ |
| | Capsule | [P]XXXXXXXXXXXXXXXXXX | mm-dd | mm-dd | | | | C: Dose Not | | C: Related | Resolved |
| | | [S]XXXXXXXXXXXXXXXXXX | hh:mm | [x] | | | | Changed | | | |
| | | | [x] | | | | | | | | |
| | Period 2/ | XXXXXXXXXXXXX | уууу- | уууу- | Y | N | Grade 1 | T: Dose Not | | T: Related | Recovered/ |
| | Tablet | [P]XXXXXXXXXXXXXXXXXX | mm-dd | mm-dd | | | | Changed | | C: NA | Resolved |
| | | [S]XXXXXXXXXXXXXXXXXX | hh:mm | [x] | | | | C: NA | | | |
| | | | [x] | | | | | | | | |
| | PK Safety FU | | | | | | | | | | |

- [1] Relative to the date of first dose in PK Phase.
- [2] Reason for SAE: 1 = Result in death; 2 = Life threatening; 3 = Result in persistent or significant disability/incapacity;
- 4 = Requires or prolongs hospitalization; 5 = Congenital abnormality/birth defect; 6 = Other medically important event.
- [3] T=Tablet; C=Capsule.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### [Programming notes]

Please add time to Start Date column for PK Phase Stage 2 and Extension Phase.

### Repeat for:

Table 14.3.1.15b Listing of Serious TEAEs During the PK Phase (Safety Population in the Stage 2 PK Phase)

Table 14.3.1.15c Listing of Serious TEAEs During the Extension Phase (Safety Population in the Extension Phase)

Table 14.3.1.15d Listing of Serious TEAEs During the PK Phase (Safety Population in the Stage 3 PK Phase)

Table 14.3.1.16a Listing of Deaths During the PK Phase (Safety Population in the Stage 1 PK Phase)

Table 14.3.1.16b Listing of Deaths During the PK Phase (Safety Population in the Stage 2 PK Phase)


Table 14.3.1.16c Listing of Deaths During the Extension Phase (Safety Population in the Extension Phase)

Table 14.3.1.16d Listing of Deaths During the PK Phase (Safety Population in the Stage 3 PK Phase)

- Footnote: 'NOTE: Deaths due to progressive disease were not collected as adverse events.'
- Table 14.3.1.17c Listing of TEAE Leading to Dose Interruption During the Extension Phase (Safety Population in the Extension Phase)
- Table 14.3.1.17d Listing of TEAE Leading to Dose Interruption During the PK Phase (Safety Population in the Stage 3 PK Phase)
- Table 14.3.1.18a Listing of TEAE Leading to Dose Reduction During the PK Phase (Safety Population in the Stage 1 PK Phase)
- Table 14.3.1.18b Listing of TEAE Leading to Dose Reduction During the PK Phase (Safety Population in the Stage 2 PK Phase)
- Table 14.3.1.18c Listing of TEAE Leading to Dose Reduction During the Extension Phase (Safety Population in the Extension Phase)
- Table 14.3.1.18d Listing of TEAE Leading to Dose Reduction During the PK Phase (Safety Population in the Stage 3 PK Phase)
- Table 14.3.1.19a Listing of TEAE Leading to Treatment Discontinuation During the PK Phase (Safety Population in the Stage 1 PK Phase)
- Table 14.3.1.19b Listing of TEAE Leading to Treatment Discontinuation During the PK Phase (Safety Population in the Stage 2 PK Phase)
- Table 14.3.1.19c Listing of TEAE Leading to Treatment Discontinuation During the Extension Phase (Safety Population in the Extension Phase)

Table 14.3.1.19d Listing of TEAE Leading to Treatment Discontinuation During the PK Phase (Safety Population in the Stage 3 PK Phase)

### [Programming Notes]

- Stage 3: Treatment Sequence will be NIRAPARIB TABLET FASTED/FED and NIRAPARIB TABLET FED/FASTED.
- Stage 3: Column 2: Dosing Period/Treatment Treatment should be NIRAPARIB FASTED or NIRAPARIB FED.
- Stage 3: Treatment discontinuation during PK Phase add column to record if discontinuation was due to COVID-19 ["COVID-19 Reason" with Options "COVID-19 infection" or "Issues rel. to COVID-19 pandemic"].
- Extension Phase: Replace column for Dosing Period/Treatment with Treatment (TABLET, CAPSULE) and Starting Dose.
- Extension Phase: Do not need time with start/stop dates.
- Extension Phase: Footnote: [1] Relative to first dose during the Extension Phase.

Niraparib


TESARO, Inc. Confidential

Protocol: XXXXX

Table 14.3.1.16.1c

All-Cause Mortality (Safety Population in the Extension Phase)

| | TABLET | CAPSULE | OVERALL |
|------------------------|------------|------------|------------|
| | (N=xx) | (N=xx) | (N=xx) |
| Death due to any cause | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

NOTE: Deaths occurring outside 30-day window following end of Extension Phase treatment are included in the counts.

Source: Listing 16.2.1c. Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

[Programming Notes]

This table is for final disclosure reporting purposes ONLY. All deaths reported/recorded in the database should be included.

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Table 14.3.1.20d

Summary of Incidence of COVID-19 Related Adverse Events Over Time (Safety Population in the Stage 3 PK Phase)

| | | NIRAPARIB | NIRAPARIB |
|---|---|---|---|
| | | TABLET FASTED | TABLET FED |
| | Period during COVID-19 | (N=xx) | (N=xx) |
| | Pandemic [1] | n/Patients at Risk (%) | n/Patients at Risk (%) |
| Any COVID-19 Related AE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| my covid is notaced in | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | | | , |
| Any COVID-19 Related SAE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Any COVID-19 Related Grade ≥3 AE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |

<sup>[1]</sup> TABLET PK Phase Stage 3 opened to recruitment on DDMMMYYYY, with first patient consented on DDMMMYYYY, placing the start of the recruitment during the COVID-19 pandemic.

Source: Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

Protocol: XXXXX

### Table 14.3.1.20c

Summary of Incidence of COVID-19 Related Adverse Events Over Time (Safety Population in the Extension Phase)

| | TABLET (N=xx) | CAPSULE<br>(N=xx) | OVERALL<br>(N=xx) |
|---|---|---|---|
| | n/Patients at Risk (%) | n/Patients at Risk (%) | n/Patients at Risk (%) |
| Any COVID-19 Related AE | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Im, covid is netaced in | () | , ( | (1111) |
| Any COVID-19 Related SAE | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Any COVID-19 Related Grade ≥3 AE | xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |

Note: Extension Phase for all Stages of TABLET study overlapped with COVID-19 pandemic, with all Stage 3 patients commencing treatment for the Extension Phase on or after 02JUN2021 placing the AE onset during the pandemic, while last patient commenced treatment for Stages 1 and 2 on 14MAY2018 and 05DEC2019, respectively, placing their first Extension Phase treatment dose administration prior to the start of the pandemic, as defined by WHO as of 20MAR2020, with patients across all Stages ongoing until DDMMMYYYY.

### [Programming Notes]

N accounts for all patients in Safety Population of the Extension Phase.

 ${\tt n}$  - number of patients with an event related to COVID-19.

Patients at Risk (%) - number of patients who were ongoing on Extension Phase treatment on or after 20MAR2020.


Protocol: XXXXX

Table 14.3.1.21d

Summary of Incidence of COVID-19 Related Adverse Events Over Time by Gender (Safety Population in the Stage 3 PK Phase)

Report on separate page for each: <Gender: Male, Female>

| | | NIRAPARIB<br>TABLET FASTED | NIRAPARIB<br>TABLET FED |
|---|---|---|---|
| | Period during COVID-19 | (N=xx) | (N=xx) |
| | Pandemic [1] | n/Patients at Risk (%) | n/Patients at Risk (%) |
| Any COVID-19 Related AE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Any COVID-19 Related SAE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Any COVID-19 Related Grade ≥3 AE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | | , ( | , (, |

[1] TABLET PK Phase Stage 3 opened to recruitment on DDMMMYYYY, with first patient consented on DDMMMYYYY, placing the start of the recruitment during the COVID-19 pandemic.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### Repeat for:

Table 14.3.1.22d Summary of Incidence of Adverse Events Over Time by Age Group (Safety Population in the Stage 3 PK Phase)

• Use the FDAAA age groups  $\leq$ =18, 18-64,  $\geq$ =65.

Protocol: XXXXX

Table 14.3.1.21c

Summary of Incidence of COVID-19 Related Adverse Events Over Time by Gender (Safety Population in the Extension Phase)

Report on separate page for each: <Gender: Male, Female>

| (N=xx) | (N=xx) | (N=xx) |
|---|---|---|
| n/Patients at Risk (%) | n/Patients at Risk (%) | n/Patients at Risk (%) |
| xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| xx/xxx (xx.x%) | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | n/Patients at Risk (%) xx/xxx (xx.x%) xx/xxx (xx.x%) | n/Patients at Risk (%) n/Patients at Risk (%) xx/xxx (xx.x%) xx/xxx (xx.x%) xx/xxx (xx.x%) xx/xxx (xx.x%) |

Note: Extension Phase for all Stages of TABLET study overlapped with COVID-19 pandemic, with all Stage 3 patients commencing treatment for the Extension Phase on or after 02JUN2021 placing the AE onset during the pandemic, while last patient commenced treatment for Stages 1 and 2 on 14MAY2018 and 05DEC2019, respectively, placing their first Extension Phase treatment dose administration prior to the start of the pandemic, as defined by WHO as of 20MAR2020, with patients across all Stages ongoing until DDMMMYYYY.

## Repeat for:

Table 14.3.1.22c Summary of Incidence of Adverse Events Over Time by Age Group (Safety Population in the Extension Phase)

• Use the FDAAA age groups  $\leq 18, 18-64, \geq 65$ .

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

### Table 14.3.4.1a

Summary of Study Treatment Exposure During the PK Phase (Safety Population in the Stage 1 PK Phase)

| | Statistic | Sequence<br>TABLET/CAPSULE<br>(N=xx) | Sequence<br>CAPSULE/TABLET<br>(N=xx) | OVERALL<br>(N=xx) |
|---|---|---|---|---|
| # of 100 mg Capsules Received | | | | |
| 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| # of 300 mg Tablets Received | | | | |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### Repeat for:

Table 14.3.4.1b Summary of Study Treatment Exposure During the PK Phase (Safety Population in the Stage 2 PK Phase)


# stical Analysis Plan Protocol No: 3000-01-004

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Table 14.3.4.1c

Summary of Study Treatment Exposure During the Extension Phase (Safety Population in the Extension Phase)

| | | TABLET | CAPSULE | OVERALL |
|---|---|---|---|---|
| Parameters | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Maximum Number of Cycles | Deacibeic | (IV ZIZI) | (IV AA) | (IV AA) |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | | |
| ≥ 6 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median number of cycles started | n | xx | xx | XX |
| Duration of Treatment (months) | n | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | xx.x |
| | Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Min, Max | XX, XX | XX, XX | xx, xx |
| Duration on Study (months) | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | xx.x |
| | Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Exposure duration (Months) | n | xx | xx | xx |
| <1 Month | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 - <2 Months | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 - <3 Months | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 3 Months | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 6 Months | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 12 Months | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total Number of Patients with at least 1 dose interruption | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total Number of Patients with at least 1 dose reduction | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total Number of Patients with at least 1 dose re-escalation | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dose intensity (mg/day) [1] | n | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> Dose intensity was calculated as sum of daily doses consumed divided by overall treatment exposure, in days.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Table 14.3.4.1d

Summary of Study Treatment Exposure During the PK Phase (Safety Population in the Stage 3 PK Phase)

| | Statistic | NIRAPARIB | NIRAPARIB | |
|------------------------------|-----------|-----------|-----------|-----------|
| | | FASTED | FED | OVERALL |
| | | (N=XX) | (N=XX) | (N=xx) |
| # of 300 mg Tablets Received | | | | |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Table 14.3.4.2c

Summary of Niraparib Dose by Cycle (Safety Population in the Extension Phase)

| Cycle | Starting<br>Niraparib<br>Dose (mg) | Statistic | TABLET | CAPSULE | OVERALL |
|---|---|---|---|---|---|
| 1 | 300<br>200<br>100 | N<br>n (%)<br>n (%)<br>n (%) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| 2 | 300<br>200<br>100 | N<br>n (%)<br>n (%)<br>n (%) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| 3 | 300<br>200<br>100 | N<br>n (%)<br>n (%)<br>n (%) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| • | | | | | |

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


TESARO, Inc. Protocol: XXXXX

# Confidential Table 14.3.4.3.1c

Summary and Change from Baseline of Select Hematology Parameters by Visit During the Extension Phase (Safety Population in the Extension Phase)

| | | | TABLET (N=xx) | | CAPSULE (N=xx) | | OVERALL (N=xx) | |
|---|---|---|---|---|---|---|---|---|
| arameter | Visit | Statistic | Actual | Change | Actual | Change | Actual | Change |
| arameter | Baseline | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | |
| | Cycle 1<br>- Day 8 | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| | Cycle 1<br>- Day 15 | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| | Cycle 1<br>- Day 22 | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| | Cycle 2<br>- Day 1 | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| | | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| | EOT | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x |

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:State Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY



## Programming Notes:

• Report hemoglobin, neutrophils and platelets only.

Protocol: XXXXX

### Table 14.3.4.3.2c

Shift Summary of Select Hematology Parameters During the Extension Phase (Safety Population in the Extension Phase)

| reatment Group | ment Group Post-Baseline Maximum CTCAE Grade | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| TABLET | Laboratory<br>Test | Baseline<br>CTCAE Grade | Statistic | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Missing |
| | xxxxx | Grade 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Grade 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Grade 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Grade 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Grade 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Missing | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xxxxx | | | | | | | | |

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

Include TABLET, CAPSULE and OVERALL.

### Repeat for:

Table 14.3.4.4.1c Summary and Change from Baseline of Select Chemistry Parameters by Visit During the Extension Phase (Safety Population in the Extension Phase)

Table 14.3.4.4.2c Shift Summary of Select Chemistry Parameters in Maximum Toxicity Grade During the Extension Phase (Safety Population in the Extension Phase)

Protocol: XXXXX

### Table 14.3.4.4.1d

Summary of COVID-19 Assessments for Patients with Suspected, Probable or Confirmed COVID-19 Case Diagnosis (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB TABLET | NIRAPARIB TABLET |
|-------------------------------|------------------|------------------|
| | FASTED | FED |
| Assessment | (N=XX) | (N=XX) |
| COVID-19 Case Diagnosis [1] | xx (xx.x%) | xx (xx.x%) |
| Confirmed | xx (xx.x%) | xx (xx.x%) |
| Probable | xx (xx.x%) | xx (xx.x%) |
| Suspected | xx (xx.x%) | xx (xx.x%) |
| COVID-19 Test Performed [2] | | |
| n | XX | XX |
| No | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Yes | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Result from the COVID-19 Test | | |
| n | XX | XX |
| Negative | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Positive | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Indeterminate | xx/xx (xx.x%) | xx/xx (xx.x%) |

- [1] COVID-19 Case Diagnosis is based on WHO Definition as of DDMMMYYYY.
- [2] COVID-19 Test Performed is only captured for patients with a COVID-19 Case Diagnosis.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### [Programming Notes]

For COVID-19 Test Performed, the small n is based on the number of subjects with a COVID-19 Case Diagnosis. For Result of the COVID-19 Test, the small n is based on the COVID-19 Test Performed=Yes.

IDSL standard shell PAN1.

Protocol: XXXXX

## TESARO, Inc. Confidential Page 1 of x

### Table 14.3.4.5.1c

Summary of COVID-19 Assessments for Patients with Suspected, Probable or Confirmed COVID-19 Case Diagnosis (Safety Population in the Extension Phase)

| | TABLET | CAPSULE | OVERALL |
|---|---|---|---|
| Assessment | (N=XX) | (N=XX) | (N=XX) |
| COVID-19 Case Diagnosis [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Confirmed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Probable | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Suspected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| COVID-19 Test Performed [2] | | | |
| n | xx | xx | XX |
| No | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Yes | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Result from the COVID-19 Test | | | |
| n | XX | xx | XX |
| Negative | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Positive | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Indeterminate | xx/xx (xx.x%) | xx/xx (xx.x%) | xx/xx (xx.x%) |

<sup>[1]</sup> COVID-19 Case Diagnosis is based on WHO Definition as of 20MAR2020.

Note: Extension Phase for all Stages of TABLET study overlapped with COVID-19 pandemic, with all Stage 3 patients commencing treatment for the Extension Phase on or after 02JUN2021 placing the AE onset during the pandemic, while last patient commenced treatment for Stages 1 and 2 on 14MAY2018 and 05DEC2019, respectively, placing their first Extension Phase treatment dose administration prior to the start of the pandemic, as defined by WHO as of 20MAR2020, with patients across all Stages ongoing until DDMMMYYYY.

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

<sup>[2]</sup> COVID-19 Test Performed is only captured for patients with a COVID-19 Case Diagnosis.

|-----------------|
| Protocol: XXXXX |

### Table 14.4.1c

Summary of Important Protocol Deviations (Safety Population in the Extension Phase)

| Category/Coded Term | TABLET (N=XX) | CAPSULE<br>(N=XX) | TOTAL<br>(N=XX) |
|---|---|---|---|
| Any important protocol deviations | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| CATEGORY 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| SUBCATEGORY 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| SUBCATEGORY 2 | xx (xx%) | xx (xx%) | xx (xx%) |
| CATEGORY 2 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| SUBCATEGORY 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| SUBCATEGORY 2 | xx (xx%) | xx (xx%) | xx (xx%) |

Source: Listing XXXXXXXXX. Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### [Programming Notes]:

- Include only IMPORTANT protocol deviations.
- <Category 1...> represents ADDV.DVCAT. <Subcategory 1...> represents ADDV.DVDECOD.
- Sort Categories in descending order according to overall counts, if ties are present, present alphabetically.

Table 14.4.1d

Summary of Important Protocol Deviations for the PK Phase Occurring Through End of Treatment (Safety Population in the Stage 3 PK Phase)

| Category/Coded Term | NIRAPARIB TABLET<br>FASTED [1]<br>(N=XX) | NIRAPARIB TABLET<br>FED [2]<br>(N=XX) | TOTAL [3]<br>(N=XX) |
|---|---|---|---|
| Any important protocol deviations | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| CATEGORY 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| SUBCATEGORY 1 SUBCATEGORY 2 | xx (xx%) | xx (xx%)<br>xx (xx%) | xx (xx%) |
| CATEGORY 2 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| SUBCATEGORY 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| SUBCATEGORY 2 | xx (xx%) | xx (xx%) | xx (xx%) |

- [1] Includes protocol deviations with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes protocol deviations with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.
- [3] Includes protocol deviations occurring at any time during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### [Programming Notes]:

Protocol: XXXXX

- Include only IMPORTANT protocol deviations.
- <Category 1...> represents ADDV.DVCAT. <Subcategory 1...> represents ADDV.DVDECOD.
- Sort Categories in descending order according to overall counts, if ties are present, present alphabetically.

# **LISTINGS**

# General guidelines:

Listings are separated for the PK Phase (Stage 1, Stage 2 and Stage 3 separately) and the Open-Label Extension Phase.

### For the PK Phase:

- Treatment=Sequence (for Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET; for Stage 3: NIRAPARIB TABLET FASTED/FED or NIRAPARIB TABLET FED/FASTED).
- Population=Safety Population in the PK Phase (i.e., those who receive at least 1 dose), unless otherwise specified.
- Include all data assessments relative to the PK Phase.
  - o For patients who do not continue to the Extension Phase, include all EOT/Safety FU data. Also include Extension Phase Screening for those patients who DO not proceed to the Extension Phase.
- Relative day: With respect to first date of dosing in PK period.

### For the Extension Phase:

- Treatment=TABLET; CAPSULE.
- Population=Safety Population in the Open-Label Extension Phase (i.e., those who receive at least 1 dose), unless otherwise specified.
- Include all assessments relative to the Extension Phase.
  - $\circ\quad$  Any assessment specific to Extension Phase, including Screening Data.
- Relative day: With respect to first date of dosing in Extension Phase.
  - o "-" event taking place prior to first dose in Extension Phase.
  - o "\*" event taking place after EOT in Extension Phase.


# TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

# Listing 16.2.1a

Disposition for PK Phase (All Patients Enrolled in the Stage 1 PK Phase)

Treatment: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| Patient | Date of Last | Date of | Reason for | Date of | Reason for | Date of | Date of | Protocol |
|---|---|---|---|---|---|---|---|---|
| Number | Niraparib Dose | Discontinuation | Discontinuation | Discontinuation | Discontinuation | Death | Progression | Version |
| | During PK Phase | From PK Phase | from PK Phase | from Study (Rel | from Study | (Rel | (Rel Day) | |
| | (Rel Day) | (Rel Day) | | Day) | | Day) | | |
| | | | Other: specify | | | | | |
| | | | Completion | | | | | |

Relative Day calculated relative to first dose in PK Phase.

Only study discontinuations, disease progressions and deaths that occur during PK Phase (i.e., before 1st dose of extension or prior to discontinuing the study for patients not entering the Extension Phase) are listed.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### [Programming Notes - PK Phase]

• Include only data that falls before first-dose Open-Label Extension Phase, i.e., for those patients who DC study and do not continue in the Open-Label Extension Phase.

#### Repeat for:

Listing 16.2.1b Disposition for PK Phase (Safety Population in the Stage 2 PK Phase)

Listing 16.2.1c Disposition for Open-Label Extension Phase (All Patients Enrolled for the Extension Phase)

Listing 16.2.1d Disposition for PK Phase (Safety Population in the Stage 3 PK Phase)

### [Programming Notes - Extension Phase]

- Change 'PK Phase' to 'Extension' Phase in respective columns.
- Treatment: Niraparib Tablet or Niraparib Capsule.
- Footnote: Relative Day calculated relative to first dose in Extension Phase. '-' Rel day before first Dose during Extension Phase, '\*' Rel day post 30-day safety window from EOT .

# Niraparib Statistical Analysis Plan Protocol No: 3000-01-004

| TESARO, Inc. | | Page 1 of x |
|---|---|---|
| Protocol: XXXXX | | |
| | | Listing 16.2.1.2a |
| | Reasons for Screen Fa | illure (Patients who Failed Screening in the Stage 1 PK Phase) |
| Treatment Sequence: <sc< td=""><td>REEN FAILURE&gt;</td><td></td><td></td></sc<> | REEN FAILURE> | |
| Patient | | |
| Number | Protocol Version | Inclusion/Exclusion Criteria Not Met |
| xxxxx-xxxx | Version 1.0 (original) | INPXX: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | • | |
| xxxxxx-xxxx | Version 1.0 (original) | EXPXX: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| <u> </u> | XXXXXXXXXXXXX. Output:<br>MMYYYY, Data Cutoff Dat | xxxxxxxxxxxxxrtf. Generated on DDMMMYYYY:HH:MM:SS |

# Repeat for:

Listing 16.2.1.2b Reasons for Screen Failure (Patients who Failed Screening in the Stage 2 PK Phase)

Listing 16.2.1.2d Reasons for Screen Failure (Patients who Failed Screening in the Stage 3 PK Phase)

| TESARO, Inc. | | Confi | Page 1 of x | |
|---|---|---|---|---|
| Protocol: XXX | XXX | | | |
| | | Listing | g 16.2.2a | |
| | Protocol Deviations for the PK Phase (Safety Population in the Stage 1 PK Phase) | | | |
| Treatment: < | Stage 1 & 2 | : TABLET/CAPSULE or CAPSULE/TABLET> | | |
| Patient<br>Number | Visit | Protocol Deviation Category | Protocol Deviation Severity | Description of Protocol Deviation |
| Number | VIDIC | Trococor Beviation Category | riceded peviation beverity | Descripcion of Freedom Deviation |
| Source: Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxxxrtf. Generated on DDMMMYYYY:HH:MM:SS | | | | |

### [Programming Notes]

• Include only data that falls before first-dose Open-Label Extension Phase (i.e., for those patients who DC study and do not continue in the Open-Label Extension Phase)

### Repeat for:

Listing 16.2.2b Protocol Deviation for the PK Phase (Safety Population in the Stage 2 PK Phase)


Protocol: XXXXX

Listing 16.2.2c

Important Protocol Deviations for the Open-Label Extension Phase (Safety Population in the Extension Phase)

Treatment: <TABLET, CAPSULE>

| Patient | | | | | |
|---|---|---|---|---|---|
| Number | | Protocol Deviation | Description of Protocol | | GSK |
| | Visit | Category | Deviation | TESARO Classification [1] | Classification [2] |
| | | | | < <significant important="">&gt;</significant> | < <important non-<="" td=""></important> |
| | | | | | IMPORTANT>> |

<sup>[1]</sup> For Stages 1 & 2, protocol deviation classification is done based on TESARO Protocol Deviation Management System only. GSK Classification will remain blank.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### [Programming notes]

For Stage 3 Extension Phase, patients will receive NIRAPARIB TABLET formulation only.

For Stages 1 and 2 reporting, only TESARO Classifications will be populated, for Stage 3 - only GSK Classification will be populated.

Only include protocol deviation classified as Important.


<sup>[2]</sup> For Stage 3, protocol deviation classification is done based on GSK Protocol Deviation Management System only. TESARO Classification will remain blank.

| TESARO, Inc. Confidential Page | | | | | |
|---|---|---|---|---|---|
| Protocol: XX | XXXX | | | | |
| Importa | ant Protoco | l Deviations for the PK Phase | Listing 16.2.2.1d Occurring Through End of Trea | tment (Safety Population for Stage 3 PK | Phase) |
| Treatment: < | NIRAPARIB 1 | FASTED or NIRAPARIB FED> | | | |
| Patient<br>Number | Visit | Protocol Deviation Category | Protocol Deviation Severity | Description of Protocol Deviation | |
| _ | | XXXXXXXXXXXXXXX Output: xxxxx<br>MMMYYYY, Data Cutoff Date: D | | MMMYYYY:HH:MM:SS | |

# [Programming notes]:

Only include protocol deviation classed as Important.

TESARO, Inc. Confidential


Protocol: XXXXX

Listing 16.2.2.2d

GSK Protocol Deviations related to COVID-19 (Safety Population for Stage 3 PK Phase)

Treatment: <NIRAPARIB FASTED or NIRAPARIB FED>

| Patient<br>Number | Deviation Category | Description of Deviation | GSK Classification | Date |
|---|---|---|---|---|
| | | - | <pre><important not-important=""></important></pre> | |

Note: \* Patients with probable, suspected or confirmed COVID-19.

Note: This listing only includes COVID-19 related protocol deviations.

Source: Program: XXXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

Protocol: XXXXX

Listing 16.2.2.2c

GSK Protocol Deviations related to COVID-19 (Safety Population in the Extension Phase)

Treatment: <TABLET, CAPSULE>

| Patient<br>Number | Deviation Category | Description of Deviation | GSK Classification | Date |
|---|---|---|---|---|
| | | | <pre><important not-important=""></important></pre> | |

Note: \* Patients with probable, suspected or confirmed COVID-19.

Note: This listing only includes COVID-19 related protocol deviations.

Note: Extension Phase for all Stages of TABLET study overlapped with COVID-19 pandemic, with all Stage 3 patients commencing treatment for the Extension Phase on or after 02JUN2021 placing the AE onset during the pandemic, while last patient commenced treatment for Stages 1 and 2 on 14MAY2018 and 05DEC2019, respectively, placing their first Extension Phase treatment dose administration prior to the start of the pandemic, as defined by WHO as of 20MAR2020, with patients across all Stages ongoing until DDMMMYYYY.

Source: Program: XXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY: HH: MM: SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

|---|---|---|---|
| Protocol: XXX | XX | | |
| | | Listing 16.2.3a | |
| | Study Populations : | for the PK Phase (All Patients Enrolled in | the Stage 1 PK Phase) |
| Treatment: <t< td=""><td>ABLET/CAPSULE or CAPSULE/TABLET</td><td>or SCREEN FAILURE&gt;</td><td></td><td></td></t<> | ABLET/CAPSULE or CAPSULE/TABLET | or SCREEN FAILURE> | |
| Patient<br>Number | PK Phase Safety<br>(SAF) Population | Informed Consent Date | Randomization Date |
| | Y | | |
| _ | am: XXXXXXXXXXXXXXXXXX Outpu<br>Date: DDMMMYYYY, Data Cutoff | at: xxxxxxxxxxxx.rtf. Generated on DDMMMY Date: DDMMMYYYY | YYY:HH:MM:SS |

### Repeat for:

Listing 16.2.3b Study Populations for the PK Phase (All Patients Screened in the Stage 2 PK Phase)

• For Stage 2 PK, add column for BE Evaluable Population (Y/N).

# Niraparib Statistical Analysis Plan Protocol No: 3000-01-004

| TESARO, Inc. | | Confidential | | | | Page 1 o | fх |
|---|---|---|---|---|---|---|---|
| Protocol: XXXXX | Study Populations for t | Listing 16.2.3c<br>sion Phase (All Patier | nts Enrolled in the E | xtension Phas | se) | | |
| Treatment: <tabl< td=""><td>ET or CAPSULE&gt;</td><td></td><td></td><td></td><td></td><td></td><td></td></tabl<> | ET or CAPSULE> | | | | | | |
| Patient<br>Number | Extension Phase<br>Safety (SAF)<br>Population<br>Y | | | | | | |
| | XXXXXXXXXXXXXXXXXXX O<br>e: DDMMMYYYY, Data Cut | | MMMYYYY:HH:MM:SS | | | | |

Listing 16.2.3d

Study Populations for the PK Phase (All Patients Enrolled in the Stage 3 PK Phase)

Treatment: <FASTED/FED or FED/FASTED or SCREEN FAILURE>

Protocol: XXXXX

| Patient | PK Phase | FE Population | Informed Consent Date | Randomization Date |
|---|---|---|---|---|
| Number | Safety (SAF) Population | | | |
| | Y | Y | | |
| | | N | | |

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


Protocol: XXXXX

### Listing 16.2.4.1a

Demographics (Safety Population in the Stage 1 PK Phase)

Study Treatment: <Stage 1 & 2: NOT DOSED or TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: NOT DOSED or FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| 1211001101 | Enconstant industry as approach | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Patient | Age | Sex | Child-Bearing | Ethnicity | Race | Height | Weight | BMI | ECOG Performance |
| Number | (yrs) | | Potential | | | (cm) | (kg) | (kg/m²) | Status |
| | | | | | Other: specify | | | | |

ECOG = Eastern Cooperative Oncology Group:

0=Fully active, able to carry on all pre-disease performance without restriction

1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature

2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours

3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours

4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair

Source: Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxxrtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### Repeat for:

Listing 16.2.4.1b Demographics (Safety Population in the Stage 2 PK Phase)

Listing 16.2.4.1c Demographics (Safety Population in the Extension Phase)

Add footnote for Extension Phase and relevant reference in the listing:

[1] Only weight and ECOG Performance Status were repeated at Extension Phase entry.

Listing 16.2.4.1d Demographics (Safety Population in the Stage 3 PK Phase)

Protocol: XXXXX

Listing 16.2.4.2a

Medical History (Safety Population in the Stage 1 PK Phase)

PK Phase Treatment: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| | System Organ Class | | | |
|---------|----------------------------|-------|--------------|-----------|
| Patient | Preferred Term | Start | Ongoing at | |
| Number | Medical Condition or Event | Date | Study Start? | Stop Date |

Includes only patients with major medical conditions.

Note: MedDRA version XX.X.

Source: Program: XXXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### Repeat for:

Listing 16.2.4.2b Medical History (Safety Population in the Stage 2 PK Phase)

Listing 16.2.4.2c Medical History (Safety Population in the Extension Phase)

Listing 16.2.4.2d Medical History (Safety Population in the Stage 3 PK Phase)

### [Programming notes]

For Stage 3, the latest available MedDRA version is to be used.
Protocol: XXXXX

Listing 16.2.4.3a

Prior Anti-Cancer Treatment (Safety Population in the Stage 1 PK Phase)

Treatment: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| Patient | Regimen | -Verbatim Term | | |
|---|---|---|---|---|
| Number | Number | Preferred Term | Reason for Administration | Best Response |
| | | | Other: specify | |

#### Repeat for:

Listing 16.2.4.3b Prior Anti-Cancer Treatment (Safety Population in the Stage 2 PK Phase)

Listing 16.2.4.3c Prior Anti-Cancer Treatment (Safety Population in the Extension Phase)

Listing 16.2.4.3d Prior Anti-Cancer Treatment (Safety Population in the Stage 3 PK Phase)

Protocol: XXXXX

Listing 16.2.4.4a

Primary Cancer History (Safety Population in the Stage 1 PK Phase)

Treatment: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| Patient<br>Number | Tumor Type | Date of First<br>Diagnosis | Cancer Stage (Most Recent) | Number of Prior Lines of Therapy |
|---|---|---|---|---|
| | <pre>&lt;0ther: specify&gt;</pre> | | | |

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Listing 16.2.4.4b Primary Cancer History (Safety Population in the Stage 2 PK Phase)

Listing 16.2.4.4c Primary Cancer History (Safety Population in the Extension Phase)

Listing 16.2.4.4d Primary Cancer History (Safety Population in the Stage 3 PK Phase)

| TESARO, Inc. Conf | fidential P | Page 1 o | fх |
|-------------------|-------------|----------|----|
|-------------------|-------------|----------|----|

Protocol: XXXXX

#### Listing 16.2.4.5a

Prior/Concomitant Radiotherapy (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| , and arr | ······································ | | | | |
|---|---|---|---|---|---|
| Patient | | | | | Prior/ |
| Number | Site or Region | Date Started | Date Stopped | Total Grays | Concomitant Flag |

Note: Includes patients with prior or concomitant radiotherapy with respect to the PK Phase.

P=Prior (radiotherapy with start date earlier than the first dose date of study treatment).

C=Concomitant (radiotherapy occurring on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase).

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Listing 16.2.4.5b Prior/Concomitant Radiotherapy (Safety Population in the Stage 2 PK Phase)

Listing 16.2.4.5c Prior/Concomitant Radiotherapy (Safety Population in the Extension Phase)

#### [Programming Notes for Extension Phase]

Note: Includes patients with prior or concomitant radiotherapy with respect to the Extension Phase.

P=Prior (radiotherapy with start date earlier than the first dose date of Extension Phase treatment).

C=Concomitant (radiotherapy occurring on or after the initial Extension Phase treatment dosing date through EOT in Extension Phase).

Listing 16.2.4.5d Prior/Concomitant Radiotherapy (Safety Population in the Stage 3 PK Phase)

Protocol: XXXXX

Listing 16.2.5.1a

Prior and Concomitant Medications (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

Patient Number = xxxxxx-xxxx

| ATC/<br>Preferred<br>Term/<br>Verbatim | Dose per | Dose | Frequenc | Indica | Route of<br>Administr | Start/ | | Prior/<br>Concomitant | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Term | Administration | Unit | У | tion | ation | Stop Date | Ongoing | Flag | PK Dose 1 | PK Dose 2 |
| | | | | | | | | | YYYY-MM-DD | YYYY-MM-DD |

Note: Includes patients with prior or concomitant medications taken during the PK Phase. P=Prior medication only; C=Concomitant medication only; B=Both prior and concomitant medications.

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

- For the Prior/Concomitant Flag, list all that apply.
- If ATC3 not available, use a footnote [1] ATC level 3 term is not available through WHO Drug Dictionary.

#### Repeat for:

Listing 16.2.5.1b Prior and Concomitant Medications (Safety Population in the Stage 2 PK Phase)

Listing 16.2.5.1c Prior and Concomitant Medications (Safety Population in the Extension Phase)

#### [Programming Notes for Extension Phase]

Note: Includes patients with prior or concomitant medications during the Extension Phase.

P=Prior (any medication taken earlier than the first dose date of Extension Phase treatment).

C=Concomitant (any medication on or after the initial Extension Phase treatment dosing date through EOT in Extension Phase).

Prior and concomitant medications taken during PK Phase only are classified as Prior medications during Extension Phase.

Concomitant medications taken during PK Phase and ongoing during Extension Phase are classified as Both prior and concomitant medications during Extension Phase.

• Drop 'PK Dose 1' column and replace 'PK Dose 2' with 'Extension Phase'.

Listing 16.2.5.1d Prior and Concomitant Medications (Safety Population in the Stage 3 PK Phase)

Protocol: XXXXX

### Listing 16.2.5.1.1c

Treatment Exposure and Duration (Safety Population in the Extension Phase)

Study Stage/Formulation: <Stage 1: TABLET/CAPSULE/EXT, CAPSULE/TABLET/EXT> <Stage 2: TABLET/CAPSULE/EXT, CAPSULE/TABLET/EXT > <Stage 3: TABLET>, as applicable

| | | | | | | Extension | Time between PK |
|---|---|---|---|---|---|---|---|
| Patient | Randomization | | | PK Dose 1/ Rel | PK Dose 2/ Rel | Phase | and Extension |
| Number | Date | Stage | Treatment Sequence | Day [1] | Day [1] | Dose 1 | Phase doses [2] |
| xxxxxx-xxxx | YYYY-MM-DD | <stage 1="" 2=""></stage> | <pre><tablet capsule="" ext="" ext,="" tablet=""></tablet></pre> | YYYY-MM-DD/ -xx | YYYY-MM-DD/ -xx | YYYY-MM-DD | xx |
| xxxxxx-xxxx | YYYY-MM-DD | Stage 3 | <tablet ext=""></tablet> | YYYY-MM-DD/ -xx | YYYY-MM-DD/ -xx | YYYY-MM-DD | XX |

Note: Randomized patients who did not start PK Phase treatment and proceeded to Extension Phase treatment directly will have time between PK and Extension Phase dosing set to missing.

- [1] Relative to first dose during the Extension Phase. '-' Rel day before first Dose during Extension Phase.
- [2] The time between last non-missing PK dose and first Extension Phase dose (in days).

Source: Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

For treatment sequence use actual sequence labels, as displayed in ADaMs.

Randomized patients who did not start PK Phase treatment and proceeded to Extension Phase treatment directly will have time between PK and Extension Phase dosing set to '.'.

Treatment sequence displays actual treatment formulation received during Stages 1 and 2 (T/C, C/T), and for Stage 3 displays TABLET formulation irrespective of fasting (FED/FASTED) status.

Protocol: XXXXX

Listing 16.2.5.2a

Prior/Concomitant Procedures During PK Phase (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| Patient | Procedure | Rel Day | | | | | Prior/Concomitant |
|---|---|---|---|---|---|---|---|
| Number | Date | [1] | Procedure | Results/Findings | AE/SAE? | Indication | Flag |
| XXXXXX-XXXX | | | | | | | |

[1] Relative to first dose during the PK Phase.

Note: Includes patients with prior or concomitant procedures during the PK Phase.

P=Prior (any procedure earlier than the first dose date of study treatment).

C=Concomitant (any procedure on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase).

Source: Program: XXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY: HH: MM: SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for

Listing 16.2.5.2b Prior/Concomitant Procedures During the PK Phase (Safety Population in the Stage 2 PK Phase)

Listing 16.2.5.2c Prior/Concomitant Procedures During the Extension Phase (Safety Population in the Extension Phase)

[Programming Notes for Extension Phase]

• Footnote: [1] Relative to first dose during the Extension Phase. '-' Rel day before first Dose during Extension Phase, '\*' Rel day post 30-day safety window from EOT.

Note: Includes patients with prior or concomitant procedures during the Extension Phase.

P=Prior (any procedure undertaken earlier than the first dose date of Extension Phase treatment).

C=Concomitant (any procedure undertaken on or after the initial Extension Phase treatment dosing date through EOT in Extension Phase).

Prior and concomitant procedure undertaken during PK Phase only are classified as Prior procedure during Extension Phase. Concomitant procedures performed during PK Phase and ongoing during Extension Phase are classified as Both prior and concomitant procedure during Extension Phase.

Listing 16.2.5.2d Prior/Concomitant Procedures During the PK Phase (Safety Population in the Stage 3 PK Phase)

Protocol: XXXXX

Listing 16.2.5.3a

Prior and Concomitant Transfusions (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| | Received Transfusion | | | | | |
|---|---|---|---|---|---|---|
| Patient | within 14 days of first | Type of | | | | Prior/ |
| Number | dose or during study? | Administration | Units | Transfusion Date | Rel Day [1] | Concomitant Flag |
| | | Other: specify | | | | |

[1] Relative to first dose during the PK Phase.

Note: Includes patients with prior or concomitant transfusions during the PK Phase.

P=Prior (any transfusion earlier than the first dose date of study treatment).

C=Concomitant (any transfusion on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase).

Source: Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

• For the Prior/Concomitant Flag, list all that apply.

#### Repeat for:

Listing 16.2.5.3b Prior and Concomitant Transfusions (Safety Population in the Stage 2 PK Phase)

Listing 16.2.5.3c Prior and Concomitant Transfusions (Safety Population in the Extension Phase)

#### [Programming Notes for Extension Phase]

Footnote: [1] Relative to first dose during the Extension Phase. '-' Rel day before first Dose during Extension Phase, '\*' Rel day post 30-day safety window from EOT.

Note: Includes patients with prior or concomitant transfusions during the Extension Phase.

P=Prior (any transfusion started earlier than the first dose date of Extension Phase treatment).

C=Concomitant (any transfusion started on or after the initial Extension Phase treatment dosing date through EOT in Extension Phase).

Prior and concomitant transfusion completed during PK Phase only are classified as Prior transfusion during Extension Phase.

Concomitant transfusion started during PK Phase and ongoing during Extension Phase are classified as Both prior and concomitant transfusion during Extension Phase.

Listing 16.2.5.3d Prior and Concomitant Transfusions (Safety Population in the Stage 3 PK Phase)

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Listing 16.2.5.4a

Prior and Concomitant Growth Factors (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| Patient | Received growth factor within 14 | Type of | | | Administration | Prior/ |
|---|---|---|---|---|---|---|
| Number | days of first dose or during study? | Administration | Dose | Unit | Date | Concomitant Flag |
| | | Other: specify | | Other: specify | | |

Note: Includes patients with prior or concomitant growth factors during the PK Phase.

P=Prior (any growth factor earlier than the first dose date of study treatment).

C=Concomitant (any growth factor given on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase).

#### [Programming Notes]

• For the Prior/Concomitant Flag, list all that apply.

#### Repeat for:

Listing 16.2.5.4b Prior and Concomitant Growth Factors (Safety Population in the Stage 2 PK Phase)

Listing 16.2.5.4c Prior and Concomitant Growth Factors (Safety Population in the Extension Phase)

#### [Programming Notes]

Note: Includes patients with prior or concomitant growth factors during the Extension Phase.

P=Prior (any growth factors administered earlier than the first dose date of Extension Phase treatment).

C=Concomitant (any growth factors administered on or after the initial Extension Phase treatment dosing date through EOT in Extension Phase).

Prior and concomitant growth factors administered during PK Phase only are classified as Prior growth factors during Extension Phase. Concomitant growth factors administered during PK Phase and ongoing during Extension Phase are classified as Both prior and concomitant growth factors during Extension Phase.

Listing 16.2.5.4d Prior and Concomitant Growth Factors (Safety Population in the Stage 3 PK Phase)

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Listing 16.2.5.5a

Study Treatment (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET>

| | | | | | | | | | Vomit |
|---|---|---|---|---|---|---|---|---|---|
| | | | Date:Time of | Full | If No, how | | | Fast 8 hrs | within 8 |
| Patient | | | Administration | Dose | much | Reason | Bottle | prior to | hours of |
| Number | Visit | Formulation | (Rel Day [1]) | Taken? | consumed? | for Change | Number | administration? | dose? |

[1] Relative to first dose during the PK Phase.

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

### Repeat for:

Listing 16.2.5.5b Study Treatment (Safety Population in the Stage 2 PK Phase)

[For Stage 2 PK Phase]

- Modify label for Vomiting Question, 'Vomit within specified time of dose'.
- Add column for Nausea Question, 'Nausea within specified time of dose'.

|---|---|
| Protocol: XXXXX | |
| | Listing 16.2.5.5c |
| | Study Treatment (Safety Population in the Extension Phase) |
| TREATMENT: < TABLET or CAPSULE> | |

| TREATMENT: | TREATMENT: < TABLET or CAPSULE> | | | | | | |
|---|---|---|---|---|---|---|---|
| Patient<br>Number | Visit | Dose<br>Prescribed<br>(mg) | Start Date (Rel Day [1])/<br>Stop Date (Rel Day [1]) | Action Taken | Reason for<br>Modification | Bottle<br>number<br>Dispensed | Bottle Number<br>Returned |
| | | | | | Other <specify reason=""></specify> | | |

<sup>[1]</sup> Relative to first dose during the Extension Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

Protocol: XXXXX

Listing 16.2.5.5d

Study Treatment (Safety Population in the Stage 3 PK Phase)

Treatment Sequence: <FASTED/FED or <FED/FASTED>

| | | | | | | Vomit within | Fast for |
|---|---|---|---|---|---|---|---|
| | | | Date:Time of | | Fast 10 hrs | protocol | minimum of 4 |
| Patient | | Fasted or | Administration | | prior to | specified hours | hours post |
| Number | Visit | Fed State | (Rel Day [1]) | Bottle Number | administration? | from dose? | dose? |

<sup>[1]</sup> Relative to first dose during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

| TESARO, In | ic. | Confide | ential | Page 1 of x |
|---|---|---|---|---|
| Protocol: | XXXXX | | | |
| | | Listing 16 | .2.5.6b | |
| | Subsequent Ant | ti-Cancer Therapy (Safety | Population in the Stage 2 PK Phase) | |
| Treatment | Sequence: TABLET/CAPSULE or CAPS | CULE/TABLET | | |
| Patient<br>Number | Date of Subsequent Anti-Cancer<br>Administration | Relative Day [1] | | |
| Note: Incl | 1 1 | t anti-cancer therapy rec | orded for patients who do not continue to Extension | Phase. |
| | ogram: XXXXXXXXXXXXXXXXXX. Outpact Date: DDMMMYYYY, Data Cutoff | | nerated on DDMMMYYYY:HH:MM:SS | |

# Niraparib Statistical Analysis Plan Protocol No: 3000-01-004

| TESARO, In Protocol: | | Confide | ntial | Page 1 of x |
|---|---|---|---|---|
| | | Listing 16 | .2.5.6c | |
| | Subsequent An | ti-Cancer Therapy (Safety | Population in the Extension Phase) | |
| Treatment: | < TABLET or CAPSULE> | | | |
| Patient<br>Number | Date of Subsequent Anti-Cancer<br>Administration | Relative Day [1] | | |
| | | | ost 30-day safety window from EOT. orded as initiated after last dose of the Exte | ension Phase. |
| | ogram: XXXXXXXXXXXXXXXXXX. Outp<br>ct Date: DDMMMYYYY, Data Cutoff | | nerated on DDMMMYYYY:HH:MM:SS | |

# Niraparib Statistical Analysis Plan Protocol No: 3000-01-004

| TESARO, Inc.<br>Protocol: XXX | Page 1 of x | | | | |
|---|---|---|---|---|---|
| | Meal Status (Safety Population in the Stage 3 PK Phase) | | | | |
| Treatment Seq | uence: <fasted fed<="" th=""><th>or <fed fasted=""></fed></th><th></th><th></th><th></th></fasted> | or <fed fasted=""></fed> | | | |
| Patient<br>Number | Visit | Meal Start Date | Meal Start Time | Meal End Time | % of Meal Consumed |
| Source: Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY | | | | | |


| TESARO, In | | | Confi | dential | Page 1 of x |
|---|---|---|---|---|---|
| 11000001. | 7777777 | Investigator Ass | Listing 1 | .6.2.6.1c fety Population in the Extension Phase) | |
| | | investigator not | sebament of Responde (but | recy reparation in the Entendion Image, | |
| TREATMENT: | < TABLET or CA | PSULE> | | | |
| Patient<br>Number | Tumor Type | Date | Rel Day [1] | Overall Response | |
| | | | | NE: <reason></reason> | |
| [1] Relati | _ | ± ' | • | rtial Response, SD=Stable Disease, NE=Not Evaluable. before first Dose during Extension Phase, '*' Rel day | post 30-day |
| | 2 | - | out: xxxxxxxxxxxxx.rtf. G | Generated on DDMMMYYYY:HH:MM:SS | |

Protocol: XXXXX

Listing 16.2.7.1a

Adverse Events (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| | | | Start Date:Time | | | | Action | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Dosing Period/ | Adverse Event | (Rel Day [1]) | | SAE/ | | Taken on | Other | | |
| Patient | Niraparib | MedDRA Preferred Term | End Date (Rel | | Reason | | Study | Action | Relation- | |
| Number | Treatment | System Organ Class | Day [1]) | TEAE? | [2] | Severity | Treatment | Taken | ship | Outcome |
| | Period 1/<br>Capsule | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | yyyy-mm-dd [x] | Y | N | Grade 1 | | | | Recovered/<br>Resolved |
| | Period 2/<br>Tablet | XXXXXXXXXXXXXXX [P] XXXXXXXXXXXXXXXXXXXX | yyyy-mm-dd [x] | Y | N | Grade 1 | | | | Recovered/<br>Resolved |
| | PK Safety FU | | | | | | | | | |

- [1] Relative to the date of first dose in PK Phase.
- [2] Reason for SAE: 1 = Result in death; 2 = Life threatening; 3 = Result in persistent or significant disability/incapacity;
- 4 = Requires or prolongs hospitalization; 5 = Congenital abnormality/birth defect; 6 = Other medically important event.

Source: Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

Repeat for:

Listing 16.2.7.1b Adverse Events (Safety Population in the Stage 2 PK Phase)

Listing 16.2.7.1d Adverse Events (Safety Population in the Stage 3 PK Phase)

[Programming Notes]

- Stage 3: Treatment Sequence will be Fasted/Fed and Fed/Fasted.
- Stage 3: Column 2: Dosing Period/Treatment Treatment should be Niraparib FASTED or Niraparib FED.

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Listing 16.2.7.1c

Adverse Events (Safety Population in the Extension Phase)

Treatment: <TABLET or CAPSULE>, as applicable

| Patient ID = XXXXXX-XXXX | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Adverse Event | Start Date (Rel Day [1]) | | SAE/ | | | Other | | |
| MedDRA Preferred Term | End Date (Rel Day [1]) | TEAE? | Reason | | Action Taken on | Action | | |
| System Organ Class | | | [2] | Severity | Study Treatment | Taken | Relationship | Outcome |
| XXXXXXXXXXXXX | yyyy-mm-dd [x] | Y | N | Grade 1 | | | | Recovered/ |
| XXXXXXXXXXXXXXXX | yyyy-mm-dd [x] | | | | | | | Resolved |
| XXXXXXXXXXXXXXXX | | | | | | | | |
| XXXXXXXXXXXXX | yyyy-mm-dd [x] | Y | N | Grade 1 | | | | Recovered/ |
| [P]XXXXXXXXXXXXXXXXX | yyyy-mm-dd [x] | | | | | | | Resolved |
| [S]XXXXXXXXXXXXXXXX | | | | | | | | |

- [1] Relative to the date of first dose during the Extension Phase. '\*' Rel day post 30-day safety window from EOT.
- [2] Reason for SAE: 1 = Result in death; 2 = Life threatening; 3 = Result in persistent or significant disability/incapacity;
- 4 = Requires or prolongs hospitalization; 5 = Congenital abnormality/birth defect; 6 = Other medically important event.

Source: Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS
Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

Listings 16.2.7.1c and 16.2.7.2c should be mutually exclusive. Any AEs with onset during PK Phase or after, but prior to first dose of Extension Phase should be in Listing 16.2.7.2c. If the AE is ongoing from before 1st dose of Extension Phase, and the Grade is increased, it is still an ongoing AE.

There should be no records with relative days prior to first dose of Extension Phase. If an AE has onset after EOT, indicate this with '\*'.


Protocol: XXXXX

Listing 16.2.7.2c

Adverse Events Ongoing from PK Phase (Safety Population in the Extension Phase)

Treatment: <TABLET or CAPSULE>, as applicable
Patient ID = XXXXXX-XXXX

Adverse Event

Start Date (Rel Day SAE/ Other

| Adverse Event | Start Date (Rel Day | | SAE/ | | | Other | | |
|---|---|---|---|---|---|---|---|---|
| MedDRA Preferred Term | [1]) | TEAE? | Reason | | Action Taken on | Action | | |
| System Organ Class | End Date (Rel Day [1]) | | [2] | Severity | Study Treatment | Taken | Relationship | Outcome |
| XXXXXXXXXXXXX | yyyy-mm-dd [x] | Y | N | Grade 1 | | | | Recovered/ |
| xxxxxxxxxxxxxxxx | yyyy-mm-dd [x] | | | | | | | Resolved |
| xxxxxxxxxxxxxxx | | | | | | | | |
| XXXXXXXXXXXXX | yyyy-mm-dd [x] | Y | N | Grade 1 | | | | Recovered/ |
| [P]XXXXXXXXXXXXXXXX | yyyy-mm-dd [x] | | | | | | | Resolved |
| [S]XXXXXXXXXXXXXXXX | | | | | | | | |

- [1] Relative to the date of first dose during the Extension Phase. '-' Rel day before first Dose during Extension Phase, '\*' Rel day post 30-day safety window from EOT.
- [2] Reason for SAE: 1 = Result in death; 2 = Life threatening; 3 = Result in persistent or significant disability/incapacity;
- 4 = Requires or prolongs hospitalization; 5 = Congenital abnormality/birth defect; 6 = Other medically important event.

Source: Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

TESARO, Inc.

Only include AEs with date of onset during PK Phase/prior (including Extension Phase Screening/EOT for PK Phase/Safety follow-up) to first dose of Extension Phase and ongoing/resolved during Extension Phase.

Rel Day [1] should always be either zero or negative (with onset during PK Phase, Extension Screening etc.).


Protocol: XXXXX

#### Listing 16.2.8.1.1a

Hematology Results in the PK Phase (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| Patient<br>Number | Parameter (unit) | Visit | Rel Day | Sample<br>date/time | Result | Change from baseline | Normal range | Clinically<br>significant flag |
|---|---|---|---|---|---|---|---|---|
| | | | | | xx.x | XX.X | xx.x - xx.x | |

[1] Relative to the date of first dose in the PK Phase.

Scheduled and unscheduled visits through the extension screening phase or through study discontinuation for those not continuing in the Extension Phase, are included. Visits related to the extension screening phase are not included.

Source: Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]:

• If required for readability, move 'Patient Number' into Header row after 'Treatment Sequence'.

#### Repeat for:

Listing 16.2.8.1.1b Hematology Results (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.1.1c Hematology Results (Safety Population in the Extension Phase)

Listing 16.2.8.1.1d Hematology Results Through the PK End of Treatment Visit (Safety Population in the Stage 3 PK Phase)

Listing 16.2.8.1.2a Chemistry Results (Safety Population in the Stage 1 PK Phase)

Listing 16.2.8.1.2b Chemistry Results (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.1.2c Chemistry Results (Safety Population in the Extension Phase)

Listing 16.2.8.1.2d Chemistry Results Through the PK End of Treatment Visit (Safety Population in the Stage 3 PK Phase)

Listing 16.2.8.1.3a Urinalysis Results (Safety Population in the Stage 1 PK Phase)

Listing 16.2.8.1.3b Urinalysis Results (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.1.3c Urinalysis Results (Safety Population in the Extension Phase)

Listing 16.2.8.1.3d Urinalysis Results Through the PK End of Treatment Visit (Safety Population in the Stage 3 PK Phase)

[Programming Notes For Extension Phase]:

• Footnote: [1] Relative to first dose during the Extension Phase. '-' Rel day before first Dose during Extension Phase, '\*' Rel day post 30-day safety window from EOT.

|-----------------|--------------|-----------|
| illorinto, inc. | Confidencial | rage r or |

Protocol: XXXXX

Listing 16.2.8.1.4c

Liver Function Tests - Potential Hy's Law Cases (Safety Population in the Extension Phase)

TREATMENT: < TABLET or CAPSULE>

| | | | | Laboratory Analyte (result/xULN) | | | |
|---|---|---|---|---|---|---|---|
| Patient<br>Number | Visit | Sample<br>Collection Date | Day [1] | ALT (U/L) | AST (U/L) | Total Bilirubin (umol/L) | ALP (U/L) |
| | | DDMMMYYYY | | 150/3.3 | 100/2.7 | 40/2.3 | 100/0.7 |

ALP=alkaline phosphatase. ALT=alanine aminotransferase. AST=aspartate aminotransferase. ULN=upper limit of normal.

[1] Relative to first dose during the Extension Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

Include all visits for any Patients with ALT or AST >3×ULN with bilirubin >2×ULN and ALP <2×ULN at any time in Extension Phase.

Protocol: XXXXX

Listing 16.2.8.2a

Vital Signs (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| Patient<br>Number | Visit | Assessment<br>Date | Rel<br>Day<br>[1] | Height (cm) | Weight<br>(kg) | Temperature (°C) | Pulse (beats/min) | Systolic Blood<br>Pressure (mmHg) | Diastolic Blood<br>Pressure (mmHg) |
|---|---|---|---|---|---|---|---|---|---|

[1] Relative to the date of first dose in the PK Phase.

Data is listed only when the vital sign assessment was performed.

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

Repeat for:

Listing 16.2.8.2b Vital Signs (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.2c Vital Signs (Safety Population in the Extension Phase)

[Programming Notes For Extension Phase]:

- Footnote: [1] Relative to first dose during the Extension Phase. '-' Rel day before first Dose during Extension Phase, '\*' Rel day post 30-day safety window from EOT.
- Drop Height column.

Listing 16.2.8.2d Vital Signs Through the PK End of Treatment Visit (Safety Population in the Stage 3 PK Phase)

| TESARO, Inc. Protocol: XXXXX | | | | Confidential | Page 1 of x |
|---|---|---|---|---|---|
| PIOCOCOI; AAAAA | | | | Listing 16.2.8.3a | |
| | ECG Results (Safety Population in the Stage 1 PK Phase) | | | | |
| Treatment Seque CAPSULE>, as ap | | - | TABLET/CAPSULE or CAPSUI | .E/TABLET> or <stage 3:="" fasted="" fed="" or=""> or <extension:< td=""><td>TABLET or</td></extension:<></stage> | TABLET or |
| Patient Number Visit Date Rel Day [1] ECG Interpretation | | | | | |
| [1] Relative to the date of first dose in the PK Phase. NCS = Not Clinically Significant, CS = Clinically Significant. Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY | | | | | |

#### Repeat for:

Listing 16.2.8.3b ECG Results (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.3c ECG Results (Safety Population in the Extension Phase)

Listing 16.2.8.3d ECG Results (Safety Population in the Stage 3 PK Phase)

[Programming Notes For Extension Phase]:

• Footnote: [1] Relative to first dose during the Extension Phase. '-' Rel day before first Dose during Extension Phase, '\*' Rel day post 30-day safety window from EOT.

Protocol: XXXXX

Listing 16.2.8.4a

ECOG Performance Status (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| Patient | | | | |
|---------|-------|-----------------|-------------|--------------------|
| Number | Visit | Assessment Date | Rel Day [1] | Performance Status |

[1] Relative to the date of first dose in the PK Phase. Data is listed only when the ECOG Performance Status assessment was performed. ECOG = Eastern Cooperative Oncology Group:

0=Fully active, able to carry on all pre-disease performance without restriction

1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature

2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours

3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours

4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair

Source: Program: XXXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Listing 16.2.8.4b ECOG Performance Status (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.4c ECOG Performance Status (Safety Population in the Extension Phase)

[Programming Notes For Extension Phase]:

• Footnote: [1] Relative to first dose during the Extension Phase. '-' Rel day before first Dose during Extension Phase, '\*' Rel day post 30-day safety window from EOT.

Listing 16.2.8.4d ECOG Performance Status Through the PK End of Treatment Visit (Safety Population in the Stage 3 PK Phase)

|-----------------|-------------------|
| Protocol: XXXXX | |
| | Tinting 10 0 0 Fa |

Listing 16.2.8.5a

Baseline Physical Examination Findings (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| Patient<br>Number | Visit | Date Performed | Rel<br>Day [1] | Body System | Status | Abnormality Description |
|---|---|---|---|---|---|---|

[1] Relative to the date of first dose in the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Listing 16.2.8.5b Baseline Physical Examination Findings (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.5c Baseline Physical Examination Findings (Safety Population in the Extension Phase)

[Programming Notes For Extension Phase]:

Footnote: [1] Relative to first dose during the Extension Phase.

Listing 16.2.8.5d Baseline Physical Examination Findings (Safety Population in the Stage 3 PK Phase)

Protocol: XXXXX

### Listing 16.2.8.6a

Pregnancy Test (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: TABLET or CAPSULE>, as applicable

| Patient<br>Number | Visit | Was Pregnancy Test Performed? | Date of Test | Rel Day [1] | Type | Result |
|---|---|---|---|---|---|---|
| | | 2 4 | | • • • | | |

[1] Relative to the date of first dose in the PK Phase.

Scheduled and unscheduled visits through the Extension Screening Phase or through study discontinuation for those not continuing in the Extension Phase, are included. Visits related to the Extension Screening Phase are not included.

#### Repeat for:

Listing 16.2.8.6b Pregnancy Test (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.6c Pregnancy Test (Safety Population in the Extension Phase)

[Programming Notes For Extension Phase]:

Footnote: [1] Relative to first dose during the Extension Phase. '-' Rel day before first Dose during Extension Phase, '\*' Rel day post 30-day safety window from EOT.

Listing 16.2.8.6d Pregnancy Test (Safety Population in the Stage 3 PK Phase)

Protocol: XXXXX

#### Listing 16.2.9.2d

Listing of COVID-19 Assessments and Symptom Assessments for Patients with COVID-19 Adverse Events (Safety Population in the Stage 3 PK Phase)

Treatment Sequence: <Stage 3: Period 1: FASTED or FED; Period 2: FASTED or FED>

| Patient | Treatment | Adverse | AE | COVID-19 Case | COVID-19 Test<br>Performed/ Test | Assessments and | |
|---|---|---|---|---|---|---|---|
| Number | Period (State) | Event | Start Date | Diagnosis [1] | Date/ Results | Symptom Assessments | Result |
| XXXX | 1 (FASTED) | Coronavirus infection | 2020-04-16 | Suspected | Yes/<br>2020-04-17/<br>Indeterminate | Travel to Location with Community Transmission [2] | No |
| | | | | | | Visited Health Care Facility [2] | No |
| | | | | | | Contact with COVID-19 Confirmed/Probable Case [2] | Unknown |
| | | | | | | Medication Taken to Treat COVID-19 | Yes |
| | | | | | | Fever | Yes |
| | | | | | | Cough | Yes |
| | | | | | | Shortness of Breath | Yes |
| | | | | | | Sore Throat | No |
| | | | | | | Loss of Appetite | No |
| | | | | | | Nausea | No |
| | | | | | | Vomiting | No |
| | | | | | | Diarrhea | No |
| | | | | | | Abdominal Pain | No |
| | | | | | | Fatigue | No |
| | | | | | | Loss of Smell | No |
| | | | | | | Loss of Taste | No |
| | | | | | | Asymptomatic | No |
| | | | | | | Home Quarantined/Isolated | Unknown |
| | 2 (FED) | | | | | | 1 |
| Y | | | | | | | |

#### AE=Adverse event.

- [1] COVID-19 Case Diagnosis is based on WHO Definition as of DDMMMYYYYY.
- [2] Within 14 days prior to symptom onset.

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

The COVID-19 AE terms include: Asymptomatic COVID-19, Coronavirus infection, COVID-19, COVID-19 pneumonia, Suspected COVID-19. Note that the number of COVID-19 AE terms may change.

TESARO, Inc. Confidential Page 1 of x Protocol: XXXXX

Listing 16.2.9.2c

Listing of COVID-19 Assessments and Symptom Assessments for Patients with COVID-19 Adverse Events (Safety Population in the Extension Phase)

Treatment: <CAPSULE or TABLET>

| Patient<br>Number | Formulation | Adverse<br>Event | AE Start<br>Date | COVID-19 Case<br>Diagnosis [1] | COVID-19 Test Performed/ Test Date/ Results | Assessments and<br>Symptom Assessments | Result |
|---|---|---|---|---|---|---|---|
| xxxx | TABLET | Coronavirus<br>infection | 2020-04-<br>16 | Suspected | Yes/<br>2020-04-17/<br>Indeterminate | Travel to Location with Community Transmission [2] | No |
| | | | | | | Visited Health Care<br>Facility [2] | No |
| | | | | | | Contact with COVID-19 Confirmed/Probable Case [2] | Unknown |
| | | | | | | Medication Taken to Treat<br>COVID-19 | Yes |
| | | | | | | Fever | Yes |
| | | | | | | Cough | Yes |
| | | | | | | Shortness of Breath | Yes |
| | | | | | | Sore Throat | No |
| | | | | | | Loss of Appetite | No |
| | | | | | | Nausea | No |
| | | | | | | Vomiting | No |
| | | | | | | Diarrhea | No |
| | | | | | | Abdominal Pain | No |
| | | | | | | Fatigue | No |
| | | | | | | Loss of Smell | No |
| | | | | | | Loss of Taste | No |
| | | | | | | Asymptomatic | No |
| | | | | | | Home Quarantined/Isolated | Unknown |
| | CAPSULE | | | | | | |

#### AE=Adverse event.

- [1] COVID-19 Case Diagnosis is based on WHO Definition as of DDMMMYYYY.
- [2] Within 14 days prior to symptom onset.

Note: Extension Phase for all Stages of TABLET study overlapped with COVID-19 pandemic, with all Stage 3 patients commencing treatment for the Extension Phase on or after 02JUN2021 placing the AE onset during the pandemic, while last patient commenced treatment for Stages 1 and 2 on 14MAY2018 and 05DEC2019, respectively, placing their first Extension Phase treatment dose administration prior to the start of the pandemic, as defined by WHO as of 20MAR2020, with patients across all Stages ongoing until DDMMMYYYY.

Source: Program: XXXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# Signature Page for 213362 TMF-16339705 v1.0

| Reason for signing: Approved | Name: PPD Role: Author Date of signature: 12-Jul-2023 13:42:14 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: 12-Jul-2023 15:14:33 GMT+0000 |

Signature Page for TMF-16339705 v1.0

### Statistical Analysis Plan

AN OPEN-LABEL, RANDOMIZED-SEQUENCE, MULTICENTER, SINGLE-CROSSOVER STUDY TO ASSESS THE RELATIVE BIOAVAILABILITY AND BIOEQUIVALENCE OF NIRAPARIB TABLET FORMULATION COMPARED TO NIRAPARIB CAPSULE FORMULATION IN PATIENTS WITH ADVANCED SOLID TUMORS

GSK/TESARO Protocol 213362/3000-01-004

Number:

Protocol Version: 6.0 (Amendment 5)

Compound Number: GSK 3985771, MK-4827

Study Drug Name: Niraparib

Phase: Phase 1

Methodology: Open-Label, Cross-Over

Sponsor: TESARO, a Glaxo Smith Kline Company

Analysis Plan Date: 21 December 2021

Analysis Plan Version: Version 6.0

### **Confidentiality Statement**

All information contained in this document is privileged and confidential to TESARO, a wholly owned subsidiary of Glaxo Smith Kline (GSK). Any distribution, copying, or disclosure is strictly prohibited without prior written approval by TESARO.


### SPONSOR SIGNATURE PAGE

Protocol Title: AN OPEN-LABEL, RANDOMIZED-SEQUENCE,

MULTICENTER, SINGLE-CROSSOVER STUDY TO ASSESS THE RELATIVE BIOAVAILABILITY AND

BIOEQUIVALENCE OF NIRAPARIB TABLET

FORMULATION COMPARED TO NIRAPARIB CAPSULE FORMULATION IN PATIENTS WITH ADVANCED SOLID


**TUMORS** 

Protocol Number: 3000-01-004

Sponsor: TESARO, a Glaxo Smith Kline Company

980 Great West Road

Brentford

Middlesex, TW8 9GS

UK

By signing this document, I acknowledge that I have read the document and approve of the planned statistical analyses described herein. I agree that the planned statistical analyses are appropriate for this study, are in accordance with the study objectives, and are consistent with the statistical methodology described in the protocol, clinical development plan, and all applicable regulatory guidance and guidelines.

| Author: | Signature: | PPD |
|---------------------------|------------|-----|
| Alina Striha | | |
| Senior Statistician | | |
| Plus-Project Ltd. | | |
| | Date: | |
| Approver: | Signature: | |
| Izabela Malinowska | | |
| Medical Director | | |
| Glaxo Smith Kline Company | | |
| | Date: | |


# TABLE OF CONTENTS

| S | PONSC | PR SIGNATURE PAGE | 2 |
|---|--------|----------------------------------------------------|-----|
| T | ABLE | OF CONTENTS | 3 |
| T | ABLES | INCLUDED IN THE TEXT | 5 |
| F | IGURE | S INCLUDED IN THE TEXT | 5 |
| L | IST OF | ABBREVIATIONS AND DEFINITIONS OF TERMS | 6 |
| 1 | INF | ORMATION FROM THE STUDY PROTOCOL | 8 |
| | 1.1 | Introduction and Objectives | 8 |
| | 1.1. | 1 Introduction | 8 |
| | 1.1.2 | 2 Study Objectives | 8 |
| | 1.1. | Scope and Revision History | 9 |
| | 1.2 | Study Design | 12 |
| | 1.2. | 1 Synopsis of Study Design | 12 |
| | 1.2.2 | 2 Randomization Methodology | 15 |
| | 1.2. | 3 Unblinding | 16 |
| | 1.2.4 | 4 Study Procedures | 16 |
| | 1.2. | 5 Efficacy, Safety, and Pharmacokinetic parameters | 16 |
| 2 | Pati | ent Population | 16 |
| | 2.1 | Population Definitions | 16 |
| | 2.2 | Protocol Deviations. | 17 |
| 3 | GEN | NERAL STATISTICAL METHODS | 17 |
| | 3.1 | Sample Size Justification | 17 |
| | 3.2 | General Methods | 18 |
| | 3.3 | Baseline Definitions | 19 |
| | 3.4 | Methods of Pooling Data | 20 |
| | 3.5 | Adjustments for Covariates | 20 |
| | 3.6 | Multiplicity Adjustment | 20 |
| | 3.7 | Subpopulations | 20 |
| | 3.8 | Withdrawals, Drop-outs, Loss to Follow-up | 20 |
| | 3.9 | Missing Data | 20 |
| | 3.10 | Visit Windows | 21 |
| | 3.11 | Interim Analysis | 21 |
| | 3 12 | COVID-19 | 2.1 |

| 4 | STU | DY ANALYSES | 21 |
|---|-------|------------------------------------------------------------|----|
| | 4.1 | Patient Disposition | 21 |
| | 4.2 | Demographics, Baseline Characteristics and Medical History | 22 |
| | 4.3 | Investigator Assessment of Response | 23 |
| | 4.4 | Safety Evaluation | 23 |
| | 4.4.1 | Treatment Exposure and Compliance | 23 |
| | 4.4.2 | Adverse Events | 23 |
| | 4.4.3 | Laboratory Data | 26 |
| | 4.4.4 | Vital Signs and Physical Examination | 27 |
| | 4.4.5 | Electrocardiogram | 27 |
| | 4.4.6 | Prior and Concomitant Mediations | 27 |
| | 4.4.7 | Prior and Concomitant Transfusions and Growth Factors | 28 |
| | 4.4.8 | COVID-19 | 28 |
| 5 | СНА | NGES TO PLANNED ANALYSES | 29 |
| | 5.1 | Changes in v5.0 of the SAP | 29 |
| | 5.2 | Changes in v6.0 of the SAP | 29 |
| 6 | APP | ENDIX | 30 |
| | 6.1 | Planned Statistical Tables, Listings, and Figures | 30 |

| 3 T. | • • |
|---------|-------|
| Nira | narih |
| 1 111 U | pario |

# Statistical Analysis Plan


| TABLES INCLUDED IN THE TEXT | |
|---|---|
| TABLE 1 REVISION HISTORY | 11 |
| TABLE 2 NCI COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS V4.03 (CTCAE) | 27 |
| FIGURES INCLUDED IN THE TEXT | |
| FIGURE 1 STUDY DESIGN: SINGLE-CROSSOVER STUDY | 15 |


LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS


| Abbreviation | Definition |
|---|---|
| AE(s) | adverse event(s) |
| AESI | Adverse Events of Special Interest |
| ALT | alanine aminotransferase |
| ALP | alkaline phosphatase |
| AML | Acute Myeloid Leukemia |
| AST | aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| AUC | area under the plasma concentration-time curve |
| BA | bioavailability |
| BE | bioequivalence |
| BMI | body mass index |
| CI | confidence interval |
| CL/F | apparent total body clearance |
| C <sub>max</sub> | Maximum observed plasma concentration |
| CSR | clinical study report |
| CV | coefficient of variation |
| ECG | electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic case report form |
| ЕОТ | end-of-treatment |
| FE | food effect |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| LLN | lower limit of normal |
| LS mean | least-squares mean |
| CCI | |
| MDRP | Medical Data Review Plan |
| MDS | Myelodysplastic Syndromes |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCI CTCAE | National Cancer Institute Common Terminology Criteria for Adverse Events |
| PI | Package Insert |
| PK | pharmacokinetics |
| PT | preferred term |

| Abbreviation | Definition |
|------------------|------------------------------------------|
| Q <sub>1</sub> | first quartile |
| Q <sub>3</sub> | third quartile |
| QD | one time per day |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SOC | system organ class |
| t <sub>1/2</sub> | termination elimination half-life |
| TEAE | treatment-emergent adverse event |
| t <sub>max</sub> | Time to reach C <sub>max</sub> |
| US | United States |
| ULN | upper limit of normal |
| Vz/F | apparent terminal volume of distribution |
| WHO | World Health Organization |

#### 1 INFORMATION FROM THE STUDY PROTOCOL

## 1.1 Introduction and Objectives

#### 1 1 1 Introduction

The approved niraparib drug product is an immediate release hard gelatin capsule dosage form that contains 100 mg of niraparib per capsule. The labelled starting dose for niraparib is 300 mg. Facilitating this dose requires the administration of three 100 mg capsules.

It is Sponsor's intent to introduce a tablet dosage form that provides the 100 mg, 200 mg and 300 mg dose in single dose strength tablets to reduce the pill burden on the patients.

To this end, the Sponsor has developed a tablet dosage form with the specific intent to provide comparable performance to the approved capsule dosage form. The formulation and manufacturing process of the tablet were selected to produce a tablet with comparable in-vitro performance to the capsule.

This study is an open-label Phase 1 study to evaluate the relative bioavailability (BA) and bioequivalence (BE) of niraparib administered as a tablet formulation compared to the reference capsule formulation manufactured by the same process as currently marketed in the United States. Specifically, a 300 mg niraparib tablet will be compared to three (3) niraparib capsules ( $3 \times 100$  mg). In addition, this study will evaluate the effect of a high-fat meal on the pharmacokinetics (PK) of the niraparib 300 mg tablet formulation (Stage 3). The Extension Phase of this study is to enable patients enrolled in the study to continue to receive treatment with niraparib if they are tolerating it and, in the Investigator's opinion, may receive benefit.

#### 1.1.2 Study Objectives

The primary objectives of this study are as follows:

- Stage 1: To obtain preliminary assessment of the relative bioavailability of 300 mg niraparib
  administered as a tablet versus capsule formulation and to estimate the intra-subject variability of
  niraparib PK
- Stage 2: To evaluate if the tablet formulation (1  $\times$  300 mg) of niraparib is bioequivalent to the capsule formulation (3  $\times$  100 mg)
- Stage 3: To assess the effect of a high-fat meal on niraparib PK following a single 300 mg dose of the tablet formulation.

The secondary objectives of this study are as follows:

- Stage 1, Stage 2, and Stage 3: To evaluate the safety of single dose niraparib when administered as a tablet or capsule formulation in patients with advanced solid tumors
- Extension Phase: To evaluate the safety of continuously dosed niraparib in patients with advanced solid tumors.

CCI

# 1.1.3 Scope and Revision History

The exploratory objectives of this study are as follows:

A separate PK analysis plan will be written to address the PK objectives and data for this study.

This statistical analysis plan (SAP) is designed to outline the methods to be used in the analyses of non-pharmacokinetic study data. Patient populations to be used for analyses, data handling rules, statistical methods, and formats for data presentation are identified and provided. The statistical analyses and summary tabulations described in this SAP will provide the basis for the results sections of the clinical study report (CSR) for this trial.

The SAP will outline any differences in the currently planned analytical objectives relative to those planned in the study protocol.

The SAP is a living document that will be created during the trial conduct. It will be maintained throughout the lifecycle of the trial. Important changes following approval of SAP v1.0 will be tracked in this section.

The following changes have been implemented in the Appendix containing shells of the Planned Statistical Tables, Listings and Figures.

| Table/Listing<br>Number | Correction | Reason for Correction |
|---|---|---|
| Table 14.1.1D | Footnotes [2] and [3] added to the table and in the footer. | Clarification why two patients have been double counted in Screening. |
| Table 14.1.4D | Added "Missing" category to Cancer stage and Number of prior lines of therapy. | Data collected has missing information on the eCRF. |
| Table 14.3.1.1.2D | Removed "Any COVID-19 related TEAE". | Removing a duplicate entry row. |
| Table 14.3.1.14D | Removed "System Organ Class" from the table. | Line not required for the table in question as summary by Preferred Term is of interest. |
| Table 14.3.1.16D | Added footnote: "NOTE: Deaths due to progressive disease were not collected as adverse events." | Added to reflect data collection and management process and align with Stage 1 and Stage 2 programming practice. |
| Table 14.3.1.2.1.1D | Footnote added: Note: COVID-19 Case Diagnosis is based on WHO Definition as of DDMMMYYYY. | Added as per reviewer request. |
| Table 14.3.1.20D | Footnote [1] updated to: "[1] TABLET PK Phase Stage 3 opened to | Clarification of footnote explaining calendar placement of the Stage 3 |
| Table 14.3.1.21D | recruitment on DDMMMYYYY, with first patient consented on DDMMMYYYY, placing | during COVID-19 pandemic. |
| Table 14.3.1.22D | the start of the recruitment during the COVID-19 pandemic." | |

| | <ul> <li>Table titles updated to</li> <li>Table 14.3.1.20D Summary of Incidence of COVID-19 Related Adverse Events Over Time (Safety Population in the Stage 3 PK Phase)</li> <li>Table 14.3.1.21D Summary of Incidence of COVID-19 Related Adverse Events Over Time by Gender (Safety Population in the Stage 3 PK Phase)</li> <li>Table 14.3.1.22D Summary of Incidence of COVID-19 Related Adverse Events Over Time by Age Group (Safety Population in the Stage 3 PK Phase)</li> </ul> | Clarification of titles to reflect the reporting effort of COVID-19 related AE incidence rates. |
|---|---|---|
| Table 14.4.1C | Summary table of Important Protocol<br>Deviations for Open-Label Extension Phase<br>added. | Added upon request from study team for CSR reporting purposes. |
| Table 14.4.1D | Summary table of Important Protocol Deviations for the PK Phase Occurring Through End of Treatment (Safety Population in the Stage 3 PK Phase). Footnotes and corresponding references added to the table. | Added upon request from study team for CSR reporting purposes. Added upon request for clarification. |
| Listing 16.2.5.1D | Added "PK Dose 1" and "PK Dose 2" date columns to the listing. | Added columns to the shells to align Stage 3 reported outputs with those reported in Stages 1 and 2. |
| Listing 16.2.5.3D | Moved "Patient Number" into header row. Added "Rel Day [1]" column and [1] footnote: "[1] Relative to first dose during the PK Phase." | For readability purposes. Added to the shells to align Stage 3 reported outputs with those reported in Stages 1 and 2. |
| Listing 16.2.5.5D | Columns "Full Dose Taken?", "If N, how much consumed?", "Reason for Change", "Nausea within specified time of dose?" removed from the listing. | Columns removed from Stage 3 listing as not applicable, as per study design. |
| Listing 16.2.8.1.1D and associated repeat listings | Programming note added regarding location of "Patient Number" in the outputs. | Depending on spacing/information displayed, "Patient Number" may be displayed in the header row after "Treatment Sequence" in order to aid readability of the listing. |
| Listing 16.2.8.2D | Removed "Heart Rate" column. | Data collected under "Pulse" in Stage 3, added "Heart Rate" to the shells in error. |
| Listing 16.2.8.5D | Added text to footnote: "in the PK Phase" | Previously missing in error. |
| Listing 16.2.2C | Listing updated to include only "Important" protocol deviations, title updated to reflect change. | Updated upon request from study team for CSR reporting purposes. |
| Listing 16.2.2.1D | Listing updated to include only "Important" protocol deviations, title updated to reflect change. | Updated upon request from study team for CSR reporting purposes. |
| Section 1.2 | Definition of data cut has been amended. | Definition changed to reflect study reporting requirements upon request from study team. |

Table 1 Revision History

| SAP<br>version | Protocol version | eCRF<br>version | Changes from previous version |
|---|---|---|---|
| 1.0 | 2.0 | 5.0<br>(26FEB2018) | First Draft |
| 2.0 | 4.0 | 8.0<br>(12FEB2019) | <ul> <li>Major changes to this draft of the SAP include the following:</li> <li>Incorporate changes based on amended protocol.</li> <li>Modify Stage 2 analysis of AEs to accommodate the increase in washout time between period 1 and period 2 for Stage 2.</li> <li>For the Extension Phase, specify that analysis will be performed by formulation and overall to accommodate allowance of both tablet and capsule formulation in the Extension Phase.</li> <li>Define the BA/BE evaluable population and add demographic and baseline characteristic summaries for this population.</li> <li>Clarify definition of concomitant medications and add additional table for Stage 2 to analyze only medications taken during the PK collection period.</li> <li>Clarifications to mock table and listing shells (e.g., numbering, footnotes).</li> </ul> |
| 3.0 | 5.0 | 10.0<br>(31JUL2019) | <ul> <li>Major changes to this draft of the SAP include the following: <ul> <li>Incorporate changes based on amended protocol, including:</li> <li>Updated numbers of patients enrolled to account for non-evaluability.</li> <li>Specification of reasons for non-evaluability for the analysis of bioequivalence.</li> </ul> </li> <li>Focus Extension Phase laboratory summaries on select laboratory assessments hemoglobin, neutrophils, platelets, bilirubin, creatinine, AST, and ALT).</li> </ul> |
| 4.0 | 6.0 | 11.0<br>(23MAR2021) | <ul> <li>Major changes to this draft of the SAP include the following:</li> <li>Incorporate changes based on amended protocol, to address the objectives for Stage 3 of the study.</li> <li>Addition of sections relating to COVID-19 reporting.</li> </ul> |
| 5.0 | 6.0 | 11.0<br>(23MAR2021) | Primary changes to this draft associated with addition of Important Protocol Deviation table and updates to the associated listing to reporting effort. Minor updates to align Stage 1, 2 and 3 TLFs with shells, and associated update to Protocol Deviation reporting, as per the SAP. |

| SAP<br>version | Protocol version | eCRF<br>version | Changes from previous version |
|---|---|---|---|
| 6.0 | 6.0 | 11.0<br>(23MAR2021) | Primary change to this draft of the SAP is change of the data cut for reporting of final Stage 3 analysis. Minor update to footnotes of Important Protocol Deviation summary table. Minor update to Section 5 formatting. |

# 1.2 Study Design

### 1.2.1 Synopsis of Study Design

This is a multicenter, open-label study in patients with advanced solid tumors. This is a 3-stage, randomized-sequence, single-crossover study to assess the relative BA and BE of niraparib tablet formulation relative to the capsule formulation. In addition, Stage 3 of the protocol is a single cohort, randomized-sequence, 2 period, single dose, crossover study to assess effect of food on the PK of the niraparib tablet formulation.

Pharmacokinetics (PK) Phase: In Stages 1 and 2, patients will be randomized 1:1 to receive tablet formulation followed by capsule formulation or capsule formulation followed by tablet formulation. In Stage 3, patients will be randomized 1:1 to receive tablet formulation in a fasted state followed by tablet taken with a high-fat meal, or by tablet taken with a high-fat meal followed by tablet formulation taken in a fasted state.

Stage 1: Following an 8-hour fast on Day 1, patients will receive a single dose of the formulation (tablet  $[1 \times 300 \text{ mg}]$  or capsule  $[3 \times 100 \text{ mg}]$ ) followed by a 7-day (+1 day) Washout/PK period, followed by a dose of the alternate formulation also in a fasted state, followed by a 7-day (+1 day) Washout/PK period for Stage 1 of the study followed by a dose of the alternate formulation also in a fasted state, followed by a 7-day Washout/PK period. Patients receiving the tablet in the first treatment period will receive the capsules in the second treatment period and vice versa (Figure 1). Extensive PK sampling will be carried out after niraparib dosing.

Stage 2: Following an 8-hour fast on Day 1, patients will receive a single dose of the formulation (tablet  $[1 \times 300 \text{ mg}]$  or capsule  $[3 \times 100 \text{ mg}]$ ) followed by a 14-day (+/- 4 days) Washout/PK period followed by a dose of the alternate formulation also in a fasted state, followed by a 7-day Washout/PK period. Patients receiving the tablet in the first treatment period will receive the capsules in the second treatment period and vice versa (Figure 1). Extensive PK sampling will be carried out after niraparib dosing.

Stage 3: In period 1, patients will receive a single 300 mg niraparib tablet either following a 10-hour fast or directly following consumption of a high-fat meal, followed by a 14-day (+4 days) PK sampling and Washout period. In period 2, patients will be crossed over to receive a single 300 mg niraparib tablet in a fasted state or with a high-fat meal, followed by a 7-day PK sampling period. All patients will fast for a minimum of 4 hours post-dose in both periods. Patients receiving the tablet in the fasted state in the first treatment period will receive the tablet with a high-fat meal in the second treatment period and vice versa.

In the rare instance where a delay of the entire PK period 2 is needed for any reason beyond the 4 day window specified above the site must contact the Sponsor's medical monitor to discuss the patient circumstances, the Sponsor will decide if the patient can continue with PK period 2 with a delay. Similarly, should the laboratory results on Day 15 (D15) (the day of niraparib administration in PK period 2) show changes in organ function such that the original inclusion criteria for laboratory values are no longer met, or in the event of a significant change of patient's clinical status as judged by the Investigator, the site must consult with the Sponsor to discuss the patient's continued participation in PK period 2. Note that sites need not wait for the pre-dose laboratory results to begin PK period 2, but rather consult the Sponsor once the results are available as needed. In Stage 2, patients who experience emesis within 9 hours of dosing or who miss a critical PK sample (such as the last PK sample on Day 8 in each period) will be discontinued from the PK Phase and will be allowed to be screened for the Extension Phase. In Stage 3, patients who experience emesis within 10 hours of dosing will be discontinued from the PK Phase and will be allowed to be screened for the Extension Phase. Patients who miss sufficient samples to render calculation of AUC unreliable will be discontinued from the PK Phase; those that meet other criteria for continued niraparib therapy will be eligible to be screened for the Extension Phase.

For Stage 1, the PK parameters that will be estimated include area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration ( $AUC_{0-t}$ ), area under the plasma concentration-time curve from time 0 extrapolated to infinity ( $AUC_{0-\infty}$ ), apparent total body clearance (CL/F), maximum observed plasma concentration ( $C_{max}$ ), time to reach  $C_{max}$  ( $t_{max}$ ), termination elimination half-life ( $t_{1/2}$ ), apparent terminal volume of distribution (Vz/F) and BA of tablet formulation relative to the capsule formulation based on  $AUC_{0-t}$ ,  $AUC_{0-\infty}$ , and  $C_{max}$ . Relative bioavailability will be assessed based on the ratio of geometric least-squares (LS) means of the test (tablet) to reference (capsule). Additionally, the pharmacokinetics of CCI will be determined (Stage 1 only).

For Stage 2, the same PK parameters as above will be estimated. To conclude bioequivalence, the 90% confidence interval (CI) of the ratio of geometric LS means of the test (tablet) to reference (capsule) product should be within 0.800 - 1.250 (80% - 125%) for  $AUC_{0-\infty}$ ,  $AUC_{0-t}$ , and  $C_{max}$ .

For Stage 3, the same PK parameters as above will be estimated. In addition,  $t_{lag}$ , the time from administration of the dose to the first quantifiable concentration, will be determined, and  $t_{max}$  will be compared between the fed and fasted states. The relative bioavailability of the 300 mg niraparib tablet administered with a high-fat meal relative to fasted dosing will be based on the ratio of geometric LS means of  $AUC_{0-t}$ ,  $AUC_{0-\infty}$ , and  $C_{max}$ .

Additional PK parameters may be estimated (e.g., residual area), if deemed appropriate.

Extension Phase: When patients complete the PK Phase of the study (at least 7-days from the beginning of PK period 2), they may be eligible to participate in the Extension Phase following review of the Extension Phase inclusion criteria and completion of the required Extension Phase screening assessments. The starting dose of niraparib in the Extension Phase will be based on the patient's baseline actual body weight or platelet count. Patients with a baseline actual body weight of  $\geq$ 77 kg and screening platelet count of  $\geq$ 150,000/µL (obtained after completion of the PK phase, as part of Extension Phase screening) will take one 300 mg strength tablet or 3 × 100 mg tablet/capsules at each dose administration (once a day [QD]). Patients with a baseline actual body weight of  $\leq$ 77 kg or screening platelet count of  $\leq$ 150,000/µL

will take one 200 mg strength tablet or  $2 \times 100$  mg tablet/capsules at each dose administration (QD). For patients whose initial starting dose is 200 mg QD, escalation to 300 mg QD is permitted after 2 cycles of therapy if no treatment interruption or discontinuation was required during the first 2 cycles of Extension Phase therapy and after approval from the Sponsor. Additional dose modifications will not be based upon changes in the patient's actual body weight during study participation. If laboratory values at the beginning of Extension Phase are outside of the range specified in the inclusion criteria, the patient may continue to participate in the study only upon Sponsor approval with consideration for an appropriately reduced dose. Should a patient start the Extension Phase at 100 mg, consideration may be given to escalate to 200 mg after 2 cycles, therapy if no treatment interruption or discontinuation was required during the first 2 cycles of Extension Phase therapy and after approval from the Sponsor.

Patients have up to 28 days (21 days for Stage 3 only; up to 28 days may be acceptable following discussion between the Sponsor and Investigator) after completion of the PK Phase to complete the screening assessments and the Extension Phase Screening Visit.

A tumor assessment is to be performed prior to the first dose of the Extension Phase (pre-Extension Phase). The pre-Extension Phase tumor assessment need not be completed if the baseline tumor assessment was performed  $\leq$  56 days before the first dose of the Extension Phase.

The Cycle 1/Day 1 Visit can occur on the same day as the Extension Phase Screening Visit, dependent upon availability of radiographic results obtained  $\leq$  56 days of the first planned dose in the Extension Phase. If the Extension Phase Screening Visit and the Cycle 1/Day 1 Visit occur on the same day, the clinical laboratory results will be reviewed by the study personnel prior to study drug administration to ensure eligibility. At the Cycle 1/Day 1 Visit, patients will undergo safety assessments and will receive study drug supply for the duration of 1 cycle (300 mg or 200 mg tablets of niraparib for QD dosing or  $3 \times 100$  mg or  $2 \times 100$  mg tablet/capsules of niraparib for QD dosing, depending on availability). It is preferred that patients remain on the same formulation (tablet versus capsule) throughout the Extension Phase. Patients will return on the first day of every treatment cycle ( $28 \pm 7$  days) to receive study drug and for safety assessments. Visits will continue approximately every 4 weeks until treatment discontinuation. In line with the niraparib United States Package Insert (US PI), dose interruption (no longer than 28 days) will be allowed based on adverse events (AEs). In addition, dose reductions to 200 mg QD and subsequently to 100 mg QD will be allowed based on AEs (please refer to US PI). Any dose reductions differing from this must be discussed with the medical monitor. Patients can continue in the Extension Phase until the patient meets 1 of the withdrawal criteria.

End-of-treatment (EOT) and Safety Follow-up Visits: The EOT visit will occur within 7 days of the decision to discontinue study drug, for any reason, or completion of the PK Phase for patients who participate in the Extension Phase (Stage 3 only), whichever occurs first. Should the first dose of a new anti-cancer therapy occur within 14 days of the decision to discontinue study drug, all assessments required for the Safety Follow-up visit should occur at the EOT visit and this visit will be considered the Safety Follow-up visit. If the first dose of the new anti-cancer therapy occurs >14 days of the decision to discontinue study, the Safety Follow-up visit will occur 30 +7 days after the last dose of the study drug, or at the start of any new anti-cancer therapy, whichever occur first.

For Stage 3 of the PK Phase only, the data cut will occur when all patients have completed the PK Phase. Data collected up to and including PK EOT visit prior to the data cut will be presented in the FE Stage 3

PK CSR for all randomized and treated patients. Additionally, the Sponsor will include safety data related to the PK Phase, as identified up to Cycle 1/Day 1 of the Extension Phase.

Figure 1 Study Design: Single-Crossover Study



Stage 2 (completed):



Stage 1 (completed):



Abbreviations: PK = pharmacokinetics.

#### 1.2.2 Randomization Methodology

Randomization will occur centrally using an interactive voice response system/integrated web response system. In Stage 1 and Stage 2, patients will be assigned randomly in a 1:1 ratio to a dosing sequence: capsule formulation followed by tablet formulation, or vice versa. In Stage 3, patients will be assigned randomly in a 1:1 ratio to a dosing sequence: dosing after receiving a high-fat meal (fed) followed by dosing after fasting, or vice versa. The period between randomization and Cycle 1/Day 1 should be no longer than 5 calendar days.

# 1.2.3 Unblinding

Unblinding is not applicable as this is an open-label study.

## 1.2.4 Study Procedures

Refer to the latest protocol for the schedule of assessments.

#### 1.2.5 Efficacy, Safety, and Pharmacokinetic parameters

#### 1.2.5.1 Efficacy parameters

Investigator assessment of response will occur every 3-cycles while on study or per the Institution's standard practice.

#### 1.2.5.2 Safety parameters

Safety parameters to be assessed include:

- Treatment emergent adverse events (TEAE)
- Discontinuations due to AEs
- Physical examination (PE) findings
- Vital signs
- Clinical laboratory results (hematology, chemistry, urinalysis)
- Electrocardiograms (ECG)
- Use of concomitant medications.

#### 1.2.5.3 PK parameters

PK parameters and analysis methodology will be addressed in the PK analysis plan.

# 2 Patient Population

# 2.1 Population Definitions

The following patient populations will be evaluated for analyses specified in this SAP. Additional populations, relevant to the PK analysis will be defined in the PK analysis plan.

- Safety Population in the Stage 1 PK Phase: All patients who receive any amount of niraparib during the Stage 1 PK Phase of the study.
- Safety Population in the Stage 2 PK Phase: All patients who receive any amount of niraparib during the Stage 2 PK Phase of the study.
- Safety Population in the Stage 3 PK Phase: All patients who receive any amount of niraparib during the Stage 3 PK Phase of the study.
- Safety Population in the Extension Phase: All patients who receive any amount of niraparib in the Open-Label Extension Phase of the study.
- BA/BE Evaluable Population: All patients who complete both PK periods and have sufficient PK sample collection to accurately estimate PK parameters, without significant niraparib carryover (baseline concentration > 5% of C<sub>max</sub>), in both PK Periods. Patients who have significant niraparib carryover from period 1 in period 2 will be completely excluded from the BA/BE

Evaluable Population. The terminology BA Evaluable Population will be used for Stage 1 and BE Evaluable Population will be used for Stage 2.


• Food effect (FE) Evaluable Population: All patients who complete both PK periods and have sufficient PK sample collection to accurately estimate PK parameters in both periods. Patients meeting non-evaluability criteria or having significant niraparib carryover (baseline concentration >5% of C<sub>max</sub>) will be completely excluded from the FE Population.

#### 2.2 Protocol Deviations

Protocol deviations will be assessed and classified as important and/or significant per Sponsor's SOP. The Medical Data Review Plan (MDRP) prospectively identifies classification criteria for important deviations. All protocol deviations will be identified, classified and finalized prior to database lock.

A listing of protocol deviations will be provided for the Stage 1 PK Phase, Stage 2 PK Phase; for Stage 3 PK Phase and the Open-Label Extension Phase a listing of only "Important" protocol deviations will be provided.

For Stage 3 PK Phase and Open-Label Extension Phase, tables summarizing "Important" protocol deviations will be provided.

#### 3 GENERAL STATISTICAL METHODS

## 3.1 Sample Size Justification

#### Stage 1

No formal sample size calculation was performed for Stage 1. Approximately 24 patients will be enrolled in Stage 1. This sample size is considered adequate for preliminary assessment of the relative bioavailability of the tablet compared to the capsules and for estimating the intra-subject coefficient of variation, after accounting for patient drop-outs and potential carryover.

#### Stage 2

Based on estimates from Stage 1, 100 BA/BE evaluable patients are required in Stage 2. With 100 evaluable patients, assuming the intra-subject coefficient of variation (CV) is 25% and the true ratio of means is 0.89 (89%), there is at least 90% power to demonstrate the bioequivalence (bioequivalence range: 0.80 to 1.250 [80% – 125%], alpha=0.05). Power calculations were also performed under alternative assumptions for the CV and mean ratio. Assuming the CV is 30% and the true ratio of means is 0.89 (89%), with 100 evaluable patients, there is at least 82% power to demonstrate bioequivalence. Assuming the true ratio is 0.90 (90%), the power is 96% and 88% assuming CVs of 25% and 30%, respectively.

The final analysis of bioequivalence will be based on Stage 2 BA/BE evaluable patients only, with a target sample size of 100 evaluable patients. Patients may be identified as non-evaluable due to issues arising during the study conduct, such as:

• Emesis within 9 hours of dosing,

- Dosing errors,
- Patient did not fast prior to dosing,
- Missing critical PK sample on Day 8,
- Failure to complete both PK periods, and
- Significant changes to the patient medical status that would potentially affect the PK profile as determined by the Sponsor in consultation with the Investigator prior to PK data analysis.

In this patient population, approximately 170 total patients are targeted for enrollment, assuming a 35% non-evaluability rate during the study conduct, and an additional 10% non-evaluability rate during PK analysis. The non-evaluability rate arising during the study conduct will be continuously monitored by the Sponsor and the total number of enrolled patients may be adjusted accordingly with the aim to target the resulting sample size of 100 BA/BE evaluable patients.

#### Stage 3

Assuming the true ratio of means is 1 and the intra-subject CV is 20% for  $AUC_{0-t}$  and  $AUC_{0-\infty}$ , with 16 evaluable patients, there is approximately 83% probability that the 90% CI of the ratio of geometric means will be within 0.800 and 1.250 (80% - 125%). Based on the results of a FE study conducted using the capsule formulation, an effect of a high-fat meal on  $C_{max}$  is possible. The sample size of 16 patients is deemed adequate to characterize this effect.  $AUC_{0-t}$  and  $AUC_{0-\infty}$  will be the primary parameters for analysis.

The primary analysis will be based on the FE Evaluable Population as it is the most conservative approach, which maximizes the benefits of the crossover design, where each patient serves as their own control. Results for the PK Evaluable Population will also be summarized and reported for this study.

To account for non-evaluable patients, approximately 20 total patients are targeted for enrollment. The final analysis will be based on Stage 3 FE evaluable patients only. Patients may be identified as non-evaluable due to issues arising during the study conduct, such as:

- Emesis within 10 hours of dosing,
- Dosing errors,
- Patient did not follow dietary requirements prior to dose and post-dose,
- Failure to complete both PK periods, and
- Significant changes to the patient medical status that would potentially affect the PK profile as determined by the Sponsor in consultation with the Investigator prior to PK data analysis.

Patients who miss critical PK samples or miss sufficient samples to render calculation of AUC unreliable will be discontinued from the PK Phase; those that meet other criteria for continued niraparib therapy will be eligible to be screened for the Extension Phase. The non-evaluability rate arising during the study conduct will be continuously monitored by the Sponsor and the total number of enrolled patients may be adjusted accordingly with the aim to target the resulting sample size of 16 evaluable patients.

#### 3.2 General Methods

All statistical analyses will be performed using SAS statistical software v9.4 or later, unless otherwise noted. All output will be incorporated into Microsoft Word or Excel files, or Adobe Acrobat PDF files,

sorted and labeled according to the International Conference on Harmonisation (ICH) recommendations, and formatted to the appropriate page size(s).

For categorical variables, summary tabulations of the number and percentage of patients within each category of the parameter will be presented. Percentages will be based on the patients with a non-missing parameter unless missing category is presented. Percentages will be reported to one decimal place. Percentages will not be presented for zero counts.

For continuous variables, the number of patients, mean, standard deviation (SD), median, first quartile  $(Q_1)$ , third quartile  $(Q_3)$ , minimum, and maximum values will be presented. Mean, median,  $Q_1$ , and  $Q_3$  will be reported to 1 more decimal place than the raw data, while the SD will be reported to 2 more decimal places than the raw data.

All data listings that contain an evaluation date will also contain a relative study day. A unique relative study day will be calculated for the PK Phase and Extension Phase based on the first date of dosing within the study phase. Pre-treatment and on-treatment study days are numbered relative to the day of the first dose of study drug which is designated as Day 1. The preceding day is Day -1, the day before that is Day -2, etc. Post-treatment study days are numbered relative to the first dose and are designated as Day +1, Day +2, etc.

#### In addition:

- Medical history and AEs will be coded using the most up-to-date version of Medical Dictionary for Regulatory Activities (MedDRA).
- Laboratory parameter changes during the Extension Phase for selected laboratory tests will be described using shift tables, relative to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
- Concomitant medications will be coded using the latest version of the World Health Organization's (WHO) Anatomical Therapeutic Chemical (ATC) classification.
- CIs will be presented to one more decimal place than the raw data.

Summaries in the Extension Phase will be performed by formulation and overall, regardless of starting dose, unless otherwise specified. The niraparib formulation and dose at onset will be included in the listing for the Extension Phase.

All tables, figures, and listings will include footers at the bottom of the page reflecting the programs used to generate the tables, figures, and listings, and date and time of the generation of the output.

Some minor modifications may be necessary to the planned design of tables, figures, and listings to accommodate data collected during the actual study conduct.

#### 3.3 Baseline Definitions

For all analyses unless otherwise noted, baseline is defined as the most recent measurement prior to the first administration of study drug, for each phase of the study. Baseline can be the same date as first dose, given the measurement is expected prior to first dose when only date information is available.

# 3.4 Methods of Pooling Data

Data will be pooled across study sites.

# 3.5 Adjustments for Covariates

No formal statistical analyses that adjust for possible covariate effects are planned for the safety endpoints.

# 3.6 Multiplicity Adjustment

Multiplicity is not adjusted in this study.

# 3.7 Subpopulations

Not applicable.

# 3.8 Withdrawals, Drop-outs, Loss to Follow-up

Patients will not be replaced during Stage 1. During Stage 2 and Stage 3, patients who do not complete period 1 or period 2, or who are missing PK samples which render the determination of the primary PK parameters not possible, will be replaced. After evaluation, patients receiving concomitant medications which may affect the final analysis may be replaced.

# 3.9 Missing Data

In general, there will be no imputations made to accommodate missing data points. All data recorded on the eCRF will be included in data listings for the CSR.

When tabulating AE data, partial dates will be handled as follows:

- If the day of the month is missing, the onset day will be set to the first day of the month unless it is the same month and year as first study treatment. In this case, in order to conservatively report the event as treatment-emergent, the onset date will be assumed to be the date of first study treatment.
- If the onset day and month are both missing, the day and month will be assumed to be January 1, unless the event occurred in the same year as the first study treatment. In this case, the event onset will be coded to the day of first study treatment in order to conservatively report the event as treatment-emergent.
- A missing onset date will be coded as the first day of study treatment. If the resulting onset date is after a reported date of resolution, the onset date will be set equal to the date of resolution, after considering any required imputation.

Imputation of partial dates is used only to determine whether an event is treatment-emergent; data listings will present the partial date as recorded in the eCRF.

Partial start dates for prior/concomitant medication, growth factor and transfusion data will be handled in the same way as described above for adverse events. Stop dates will be imputed as follows:

- If only day of the month is missing, the end day will be set to the last day of the month.
- If end day and end month are missing, and the year is not missing, then the day and month will be set to December 31 (or date of study discontinuation/completion if earlier than December 31).

- If the stop date is completely missing, it will be set to the date of study discontinuation/completion.
- If the imputed stop date is greater than the date of study discontinuation/completion then the date will be set to the date of study discontinuation/completion.

#### 3.10 Visit Windows

By-visit summaries and analyses will be performed by nominal visit. All data will be tabulated per the evaluation visit as recorded on the eCRF even if the assessment is outside of the visit window for analysis.

# 3.11 Interim Analysis

There will be no interim analysis for this study.

#### 3.12 COVID-19

COVID-19 pandemic may impact the conduct of clinical studies. Challenges may arise from quarantines, site closures, travel limitations interruptions to the supply chain for the investigational product or other considerations if site personnel or patients become infected with COVID-19. These challenges may lead to difficulties in meeting protocol specified procedures, including administering or using the investigational product or adhering to protocol-mandated visits and laboratory/diagnostic testing.

This study was initiated by TESARO, which was subsequently acquired by GSK. Prior to the acquisition, protocol deviations were classified using TESARO definitions. The TESARO protocol deviation system was decommissioned in May 2020, and thereafter, protocol deviations were classified using GSK definitions.

All protocol deviations collected during the study will be reviewed by the TESARO (for Stage 1 and Stage 2) or GSK (for Stage 3 only) study team, as appropriate, in order to identify TESARO "Significant"/"Important" protocol deviations and GSK "Important" protocol deviations, respectively. Consistent with ICH E3 guidance, only protocol deviations identified as "Important" (GSK) are evaluated in the CSR for impact on the Stage 3 primary endpoint.

#### 4 STUDY ANALYSES

# 4.1 Patient Disposition

A by-patient data listing of patient disposition information will be presented for each phase.

For the PK Phase (Stage 1, Stage 2 and Stage 3 separately), patient disposition will be tabulated and will include the number of patients in each of the following categories:

- Patients screened
- Patients randomized
- Patients treated with each formulation (Stage 1 and 2)
- Patients treated in fed and fasted state (Stage 3)
- Patients in the safety population

- Patients completing the PK Phase
- Primary reason for discontinuation from the PK Phase
- Primary reason for discontinuation from the study, for patients who do not continue to the Extension Phase.

For the Open-Label Extension Phase, patient disposition will be tabulated and will include the number of patients in each of the following categories:

- Patients treated with at least one dose
- Patients who discontinue treatment and the reason(s) for withdrawal
- Patients who discontinue the study and the reason(s) for withdrawal.

# 4.2 Demographics, Baseline Characteristics and Medical History

Demographics, baseline characteristics, primary cancer history, and medical history information will be summarized for the PK safety population by sequence and overall (Stage 1, Stage 2 and Stage 3 separately) and for the Open-Label Extension Phase, using descriptive statistics for the safety population. No formal statistical comparisons will be performed. Demographics and baseline characteristics will also be summarized for the BA for Stage 1, BE Evaluable Population for Stage 2 and FE Evaluable population for Stage 3.

The demographic and baseline characteristics tables will include the following variables:

- Age at time of screening (years)
- Age categories (18 to <65, 65 to  $<75, \ge 75$ ; and  $\ge 65$ )
- Sex
- Race (White, Black, Asian, American Indian/Alaska Native, Native Hawaiian or other Pacific Islander, Other and Not Reported)
- Ethnicity (Hispanic or Latino, not-Hispanic or Latino, Not Reported and Unknown)
- Baseline weight (in kilograms)
- Baseline height (in centimeters)
- Baseline body mass index (BMI) (kg/m<sup>2</sup>), calculated using the patient's height and weight at screening [BMI (kg/m<sup>2</sup>) = weight (kg) / height (m)<sup>2</sup>]
- Eastern Cooperative Oncology Group (ECOG) performance status at baseline.

Primary cancer history will be summarized for the safety population and will include the following variables:

- Tumor type
- Time from first diagnosis to informed consent (years)
- Cancer stage (most recent) (Locally advanced, Metastatic)
- Number of prior lines of therapy
- Any prior radiotherapy.

Prior anti-cancer treatments will be coded using the most current version of the WHO Drug Dictionary. The number and percentage of patients reporting the use of at least one preferred term will be reported for

the safety population in the PK Phase (Stage 1, Stage 2 and Stage 3 separately) and the safety population in the Extension Phase.

Medical history will be coded using the most current version of MedDRA, and the number and percentage of patients experiencing at least one such diagnosis by MedDRA System Organ Class (SOC) and preferred term (PT) will be reported for the safety population in the PK Phase (Stage 1, Stage 2 and Stage 3 separately) and the safety population in the Extension Phase.

Demographics, baseline characteristics, primary cancer history, and medical history information for each patient will be provided in data listings.

# 4.3 Investigator Assessment of Response

Investigator assessment of response will be provided in data listings for the Extension Phase. Additional descriptive summaries of response may be performed by tumor type.

## 4.4 Safety Evaluation

### 4.4.1 Treatment Exposure and Compliance

#### PK Phase

The number and percentage of patients receiving capsules and tablets during the PK Phase (Stage 1 and Stage 2, separately) will be summarized. For Stage 3, the number of tablets received will be summarized by fed/fasted state.

A by-patient listing of the niraparib treatment data will be produced for the PK safety population.

#### **Extension Phase**

Study treatment exposure and compliance will be summarized by formulation and overall, including:

- Number and percentage of patients who initiated 1, 2, 3, 4, 5,  $\geq$ 6 treated cycles.
- Duration of treatment (months), defined as:

[last dose date - first dose date in the Extension Phase + 1] / 30.4375.

• Duration on study (months), defined as:

[last contact date - first dose date in the Extension Phase + 1] / 30.4375, where last contact date is the last visit date or date of death.

- Number of patients with at least one dose interruption.
- Number of patients with at least one dose reduction.

In addition, the starting niraparib dose for each cycle will be summarized.

A by-patient listing of the niraparib treatment data will be produced for the Open-Label Extension Phase safety population.

#### 442 Adverse Events

All AEs will be classified by SOC and PT using the most up-to-date version of MedDRA.

Per protocol, all SAEs will be collected from the signing of the ICF for this study through 90 days after the last dose of study drug (or until the start of alternate anticancer therapy, whichever occurs first, and recorded in the eCRF.

All AEs, regardless of the source of identification (e.g., physical examination, laboratory assessment, ECG, or reported by patient), will be collected and recorded in the eCRF for each patient from the time of randomization and/or treatment assignment until 30 days after the last dose of study drug.

All AEs experienced by a patient, regardless of the suspected causality, will be monitored until the AE or SAE has resolved, until AE(s) or SAE(s) have returned to baseline or normal levels, until stabilized with a satisfactory explanation for the changes observed, until the patient is lost to follow-up, or until the patient has died, starts alternate anti-cancer therapy, or until the patient withdraws consent.

For analysis, TEAEs will be defined as any AEs collected with a start date on or after the first dose of study drug. Any AEs recorded in the database that occur from the time of ICF to first dose will be listed only and not included in safety analyses. Pre-existing conditions will be recorded in the eCRF on the Medical History or appropriate page.

The severity of the toxicities will be graded according to the NCI CTCAE v4.03. Within the same MedDRA PT, only the most severe AE for each patient will be counted in tabulations by severity. Within a MedDRA SOC, patients with more than 1 MedDRA PT will be counted only once for the most severe AE reported.

The Investigator must provide a causality assessment (related or not related) regarding the relationship of the event with the study drug and/or study procedure for all AEs. In Stage 1, for analysis of the PK Phase, AEs considered related to either tablet or capsule will be considered to be related to study drug. Any AEs for which the relationship is missing (for either tablet or capsule during the Stage 1 PK Phase) will be considered as related to study treatment. During the PK Phase 2, PK Phase 3 and Extension Phase, relationship relative to niraparib will be considered. Within the same MedDRA PT, only the AE with the highest ranked relationship to treatment for each patient will be counted in tabulations by relationship to treatment. Within a MedDRA SOC, patients with more than 1 MedDRA PT will be counted only once for the AE that is most related to treatment. The imputation for a missing relationship will take place prior to determining the most related AE within a SOC or PT for a given patient.

If the start date is missing for an AE and the actual start date cannot be determined from a partial date, the AE will be considered treatment-emergent.

Adverse Events of Special Interest (AESI) for niraparib are the following:

- Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML)
- Secondary cancers (new malignancies [other than MDS or AML])
- Pneumonitis (for Stage 1 and Stage 2 only)
- Embryo-fetal toxicity (for Stage 1 and Stage 2 only).

AEs will be classified into the following time periods for analysis.

• PK Phase (for Stage 1, Stage 2 and Stage 3 separately):

- o Period 1: Any AE that begins on or after Dose 1 but prior to Dose 2.
  - For Stage 1, Period 1 will be defined as 7-days post Dose 1 for patients who do not receive Dose 2.

- For Stage 2, Period 1 will be defined as 14-days post Dose 1 for patients who do not receive Dose 2.
- o Period 2: Any AEs that begins on or after Dose 2 but prior to the end of the PK Phase as defined by 7-days post Dose 2.
- Safety Follow-Up/Extension Screening Period:
  - For patients not participating in the Extension Phase, AEs that begin after the end of the PK Phase.
  - For patients participating in the Extension Phase, AEs that begin after the end of the PK Phase until the date of first dose in the Extension Phase.
- Open-Label Extension Phase:
  - o Any AEs that start on or after the first dose in the Extension Phase.

The analyses indicated below will be performed for each of the above-mentioned phases.

A high-level overview of TEAEs will be presented in a summary table. This table will include the number and percentage of patients for the following categories:

- Any TEAE
- Any related TEAEs
- Any serious TEAEs
- Any related serious TEAEs
- Any TEAEs with CTCAE toxicity grade 3 or above
- Any related TEAEs with CTCAE toxicity grade 3 or above
- Any TEAEs leading to treatment discontinuation
- Any related TEAEs leading to treatment discontinuation
- Any TEAEs leading to dose interruption
- Any TEAEs leading to dose reduction
- Any TEAEs leading to death.

The number and percentage of patients reporting a TEAE will be summarized in the following additional AE tables. AE tabulations will be ordered in terms of decreasing frequency for SOC (alphabetically for SOCs with the same number of AEs reported), and decreasing frequency for PT within SOC (alphabetically for PTs with the same number of AEs reported within a SOC) considering the overall rate.

- TEAE by SOC and PT
- Related TEAE by SOC and PT
- Treatment emergent SAEs by SOC and PT
- Related treatment emergent SAEs by SOC and PT
- TEAE with toxicity grade 3 or above by SOC and PT
- Related TEAE with toxicity grade 3 or above by SOC and PT
- TEAEs leading to treatment discontinuation by SOC and PT
- TEAEs leading to dose interruption by SOC and PT (Extension Phase Only)

- TEAEs leading to dose reduction by SOC and PT
- TEAEs leading to death by SOC and PT
- TEAE by PT (sorted by frequency)
- TEAE by SOC, PT, and maximum toxicity grade
- Treatment emergent AESI.

For Stage 1 and Stage 2 PK Phase, primary tabulations for the PK Phase data will be provided by formulation (regardless of period), those occurring during the follow-up/extension screening and overall. In addition, the high-level overview of TEAEs and summary of TEAEs by SOC and PT will be summarized by sequence and formulation. For Stage 3 PK Phase, primary tabulations for the PK Phase data will be provided by fed/fasted state (regardless of period), and overall. In addition, the high-level overview of TEAEs and summary of TEAEs by SOC and PT will be summarized by sequence and fed/fasted state. For the Open-Label Extension Phase, data will be summarized by formulation and for all patients overall.

The following by-patient listings will be produced for the PK Phase (Stage 1, Stage 2 and Stage 3 separately) and the Open-Label Extension Phase:

- All TEAEs
- Treatment emergent SAEs
- All Deaths
- TEAEs leading to dose interruption (Extension Phase Only)
- TEAEs leading to dose reduction
- TEAEs leading to treatment discontinuation.

#### 4.4.3 Laboratory Data

Laboratory assessments for safety oversight are performed locally at each center's laboratory by means of their established methods. All laboratory values will be converted to SI units and classified as normal, low, or high based on normal ranges supplied by the local laboratories and upon employing standardization.

A by-patient listing of all laboratory data will be provided, with laboratory reference ranges and abnormal values highlighted, and including center, patient identifier, and visit for the PK Phase and the Extension Phase of the study.

For the Extension Phase, select hematology (hemoglobin, neutrophils and platelets) and chemistry (bilirubin, creatinine, aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) will be analyzed using change from baseline by visit.

For the Extension Phase, select hematology (hemoglobin, neutrophils and platelets) and chemistry tests (bilirubin, creatinine, ALT, and AST), baseline and post-baseline results will be categorized by NCI CTCAE v4.03 grade (Table 2). Shift tables will be produced by maximum post-baseline grade. Results that are considered 'normal' will be assigned a grade 0.

# Table 2 NCI Common Terminology Criteria for Adverse Events v4.03 (CTCAE) CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

### 4.4.4 Vital Signs and Physical Examination

Vital sign measurements will be presented for each patient in a data listing.

Baseline physical examination findings will be presented in a data listing. Any new or changed condition will be captured as an adverse event and will be summarized in the AE tables and listings.

#### 4.4.5 Electrocardiogram

Standard 12-lead ECGs will be performed locally for patients in the study. Any ECG findings that are assessed as clinically significant and are reported as an AE or SAE will be summarized in the AE tables and listings.

All ECG results (i.e., interpretations) for each patient will be provided in a data listing.

#### 4.4.6 Prior and Concomitant Mediations

Medications collected at Screening and during the study will be coded using the current version of the WHO Drug dictionary. Study treatment, prior anti-cancer treatments for primary cancer, transfusions and growth factors are collected and summarized separately. For each of the study phases (Stage 1 PK, Stage 2 PK, Stage 3 PK and Extension Phase), medications will be categorized as prior or concomitant using the following definitions:

• Prior medications during the PK Phase: any medications which started prior to the first dose date of study treatment during the PK Phase.

- Concomitant medications during the PK Phase: any medications being taken on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase.
  - o For PK Stage 2, concomitant medications will be further identified as those taken during the PK collection period, defined by dates of the first PK-draw to last PK-draw.

- Prior medications during the Extension Phase: any medications which started prior to the first dose date of study treatment during the Extension Phase.
- Concomitant medications during the Extension Phase: any medications on or after the first treatment dosing date in the Extension Phase through 30 days after the last dose of treatment.

Note: medications can be classified as both prior and concomitant.

Both prior medications and concomitant medications will be summarized by ATC classification drug class and WHO preferred name using the number and percentage of patients for each cohort. A patient reporting the same medication more than once will be counted only once when calculating the number and percentage of patients who received that medication in a given time category (prior or concomitant). The summary of concomitant medications will be ordered alphabetically by drug class and then by descending frequency of preferred name in total within the drug class. For drugs with the same frequency, sorting will be done alphabetically. Summaries will be based on the safety population.

For PK Stage 2, an additional summary of concomitant medications used during the PK collection period will be provided for the BE Evaluable Population.

For each phase of the study, all prior and concomitant medications will be provided in a by-patient listing sorted by patient ID number and administration date in chronological order.

#### 4.4.7 Prior and Concomitant Transfusions and Growth Factors

The number and percentage of patients receiving prior and concomitant growth factors during the PK Phase and Extension Phase will be summarized. The data will be classified as prior or concomitant using similar logic as provided in Section 4.4.6.

For each phase of the study, all prior and concomitant transfusions and growth factor use will be provided in a by-patient listing sorted by patient ID number and administration date in chronological order.

#### 4.4.8 COVID-19

The Pharmacokinetics Phase Stage 3 of the trial takes place during COVID-19 pandemic, as a result of which some of the trial procedures could be impacted in terms of missing visits and/or assessments. Missing protocol required data/visits due to COVID-19 must be noted in participant notes and recorded as a COVID-19-related protocol deviations.

A summary of the following COVID-19 assessments will be produced: case diagnosis, COVID-19 test performed, and results of the COVID-19 test.

The incidence of COVID-19 related AEs and SAEs will be summarized as part of the safety reporting summaries along with COVID-19-related as reasons for treatment discontinuation.

A listing of all patients with COVID-19 assessments and symptom assessments will be produced and will include the following:

- Treatment sequence
- Patient number
- COVID-19 case diagnosis
- COVID-19 test performed
- Result of the COVID-19 test
- Assessments and symptom assessments performed
- Results of the assessments and symptom assessments.

For PK Phase Stage 3, a separate listing defining "Important" GSK protocol deviations related to COVID-19 will be presented.

For protocol deviation reporting during the Extension Phase, a listing will be produced to present TESARO Classification of protocol deviations for patients continuing from Stage 1 and Stage 2, and GSK Classification of protocol deviations for patients continuing from Stage 3.

#### 5 CHANGES TO PLANNED ANALYSES

There is no change between the protocol-defined statistical analyses and those planned in this SAP.

# 5.1 Changes in v5.0 of the SAP

Section 2.2 has been updated to include a summary tables of Important protocol deviations for Stage 3 PK Phase and Open-Label Extension Phases, as well as clarification of associated deviation listings presenting only protocol deviations classified as "Important".

# 5.2 Changes in v6.0 of the SAP

Section 1.2 has been updated to reflect the change in PK data cut requirements for final Stage 3 analysis.

# 6 APPENDIX

# 6.1 Planned Statistical Tables, Listings, and Figures

| TABLE 14.1.1A SUBJECT DISPOSITION IN THE PK PHASE (ALL PATIENTS IN THE STAGE I PK PHASE) | 39 |
|---|---|
| TABLE 14.1.1B SUBJECT DISPOSITION IN THE PK PHASE (ALL PATIENTS IN THE STAGE 2 PK PHASE) | 40 |
| TABLE 14.1.1C SUBJECT DISPOSITION IN THE EXTENSION PHASE (ALL PATIENTS IN THE EXTENSION PHASE) | 41 |
| TABLE 14.1.1D SUBJECT DISPOSITION IN THE PK PHASE (ALL PATIENTS IN THE STAGE 3 PK PHASE) | 42 |
| TABLE 14.1.2A DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 43 |
| TABLE 14.1.2.1A DEMOGRAPHICS (BA EVALUABLE POPULATION IN THE STAGE 1 PK PHASE) | 43 |
| TABLE 14.1.2.1B DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 43 |
| TABLE 14.1.2.2B DEMOGRAPHICS (BE EVALUABLE POPULATION IN THE STAGE 2 PK PHASE) | 44 |
| TABLE 14.1.2C DEMOGRAPHICS (SAFETY POPULATION IN THE EXTENSION PHASE) | 44 |
| TABLE 14.1.2.1D DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 44 |
| TABLE 14.1.2.2D DEMOGRAPHICS (FE EVALUABLE POPULATION IN THE STAGE 3 PK PHASE) | 44 |
| TABLE 14.1.3A BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 45 |
| TABLE 14.1.3.1A BASELINE CHARACTERISTICS (BA EVALUABLE POPULATION IN THE STAGE 1 PK PHASE) | 45 |
| TABLE 14.1.3.1B BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 46 |
| TABLE 14.1.3.2B BASELINE CHARACTERISTICS (BE EVALUABLE POPULATION IN THE STAGE 2 PK PHASE) | |
| TABLE 14.1.3C BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE EXTENSION PHASE) | 46 |
| TABLE 14.1.3.1D BASELINE CHARACTERISTICS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 46 |
| TABLE 14.1.3.2D BASELINE CHARACTERISTICS (FE EVALUABLE POPULATION IN THE STAGE 3 PK PHASE) | 46 |
| TABLE 14.1.4A PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 47 |
| TABLE 14.1.4B PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 47 |
| TABLE 14.1.4C PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE EXTENSION PHASE) | 47 |
| TABLE 14.1.4D PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 47 |
| TABLE 14.1.5A PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 49 |
| TABLE 14.1.5B PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| TABLE 14.1.5C PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| TABLE 14.1.5D PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 49 |
| TABLE 14.1.6A MEDICAL HISTORY (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 50 |
| TABLE 14.1.6B MEDICAL HISTORY (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 50 |
| TABLE 14.1.6C MEDICAL HISTORY (SAFETY POPULATION IN THE EXTENSION PHASE) | 50 |
| TABLE 14.1.6D MEDICAL HISTORY (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 50 |
| TABLE 14.1.7A PRIOR MEDICATIONS BY ATC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 51 |
| TABLE 14.1.7B PRIOR MEDICATIONS BY ATC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 51 |
| TABLE 14.1.7C PRIOR MEDICATIONS BY ATC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE) | 51 |
| TABLE 14.1.7D PRIOR MEDICATIONS BY ATC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 51 |
| TABLE 14.1.8A CONCOMITANT MEDICATIONS BY ATC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHAS | SE)53 |
| TABLE 14.1.8.1B CONCOMITANT MEDICATIONS BY ATC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHA | ASE) |
| | 53 |
| TABLE 14.1.8.2B CONCOMITANT MEDICATIONS DURING THE PK COLLECTION PERIOD BY ATC AND PT (BE | |
| EVALUABLE POPULATION IN THE STAGE 2 PK PHASE). | |
| TABLE 14.1.8C CONCOMITANT MEDICATIONS BY ATC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE | E)53 |
| TABLE 14.1.8D CONCOMITANT MEDICATIONS BY ATC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHAS | |
| TABLE 14.1.9A CONCOMITANT TRANSFUSIONS AND GROWTH FACTORS (SAFETY POPULATION IN THE STAGE 1 I | PΚ |
| Phase) | 55 |

| TABLE 14.1.9B CONCOMITANT TRANSFUSIONS AND GROWTH FACTORS (SAFETY POPULATION IN THE STAGE 2 PK |
|---|
| PHASE) |
| TABLE 14.1.9C CONCOMITANT TRANSFUSIONS AND GROWTH FACTORS (SAFETY POPULATION IN THE EXTENSION |
| PHASE) |
| TABLE 14.1.9D CONCOMITANT TRANSFUSIONS AND GROWTH FACTORS (SAFETY POPULATION IN THE STAGE 3 PK |
| PHASE) |
| TABLE 14.3.1.1.1A OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS (SAFETY POPULATION IN THI |
| STAGE 1 PK PHASE)5 |
| TABLE 14.3.1.1.1B OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS (SAFETY POPULATION IN THE |
| STAGE 2 PK PHASE)5 |
| TABLE 14.3.1.1.1C OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS (SAFETY POPULATION IN THE |
| EXTENSION PHASE) |
| TABLE 14.3.1.1.1D OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS (SAFETY POPULATION IN THI |
| STAGE 3 PK PHASE) |
| TABLE 14.3.1.1.2A OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SEQUENCE AND PERIOD |
| (SAFETY POPULATION IN THE STAGE 1 PK PHASE) |
| TABLE 14.3.1.1.2B OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SEQUENCE AND PERIOD |
| (SAFETY POPULATION IN THE STAGE 2 PK PHASE) |
| TABLE 14.3.1.1.2D OVERALL SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SEQUENCE AND PERIOD |
| (SAFETY POPULATION IN THE STAGE 3 PK PHASE) |
| TABLE 14.3.1.2.1A SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION |
| IN THE STAGE 1 PK PHASE)6 |
| TABLE 14.3.1.2.1B SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION |
| IN THE STAGE 2 PK PHASE)6 |
| TABLE 14.3.1.2.1C SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION |
| IN THE OPEN-LABEL EXTENSION PHASE)6 |
| TABLE 14.3.1.2.1D SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION |
| IN THE STAGE 3 PK PHASE)6 |
| TABLE 14.3.1.2.1.1D SUMMARY OF COVID-19 RELATED ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION |
| IN THE STAGE 3 PK PHASE)6 |
| TABLE 14.3.1.2.2A SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION |
| IN THE STAGE 1 PK PHASE) 6 |
| TABLE 14.3.1.2.2B SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION |
| IN THE STAGE 2 PK PHASE)6 |
| TABLE 14.3.1.2.2D SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT (SAFETY POPULATION |
| IN THE STAGE 3 PK PHASE)6 |
| TABLE 14.3.1.3A SUMMARY OF RELATED TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) |
| 6 |
| TABLE 14.3.1.3B SUMMARY OF RELATED TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) |
| 6 |
| TABLE 14.3.1.3C SUMMARY OF RELATED TEAE BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE)6 |
| TABLE 14.3.1.3D SUMMARY OF RELATED TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) |
| 6 |
| TABLE 14.3.1.4A SUMMARY OF SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE)6 |
| TABLE 14.3.1.4B SUMMARY OF SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHASE)6 |
| TABLE 14.3.1.4C SUMMARY OF SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE).6 |
| TABLE 14.3.1.4D SUMMARY OF SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHASE)6 |
| TABLE 14.3.1.5A SUMMARY OF RELATED SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 PK |
| PHASE) |

| TABLE 14.3.1.5B SUMMARY OF RELATED SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) |
|---|
| TABLE 14.3.1.5C SUMMARY OF RELATED SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE) |
| TABLE 14.3.1.5D SUMMARY OF RELATED SERIOUS TEAE BY SOC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) |
| TABLE 14.3.1.6A SUMMARY OF TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) |
| TABLE 14.3.1.6B SUMMARY OF TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) |
| TABLE 14.3.1.6C SUMMARY OF TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE) |
| TABLE 14.3.1.6D SUMMARY OF TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) |
| TABLE 14.3.1.7A SUMMARY OF RELATED TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) |
| TABLE 14.3.1.7B SUMMARY OF RELATED TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) |
| TABLE 14.3.1.7C SUMMARY OF RELATED TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE) |
| TABLE 14.3.1.7D SUMMARY OF RELATED TEAE WITH CTCAE TOXICITY GRADE ≥3 BY SOC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) |
| TABLE 14.3.1.8A SUMMARY OF TEAE LEADING TO TREATMENT DISCONTINUATION BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) |
| TABLE 14.3.1.8B SUMMARY OF TEAE LEADING TO TREATMENT DISCONTINUATION BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) |
| TABLE 14.3.1.8C SUMMARY OF TEAE LEADING TO TREATMENT DISCONTINUATION BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE) |
| TABLE 14.3.1.8D SUMMARY OF TEAE LEADING TO TREATMENT DISCONTINUATION BY SOC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) |
| TABLE 14.3.1.9C SUMMARY OF TEAE LEADING TO TREATMENT DOSE INTERRUPTION BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE) |
| TABLE 14.3.1.10A SUMMARY OF TEAE LEADING TO TREATMENT DOSE REDUCTION BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) |
| TABLE 14.3.1.10B SUMMARY OF TEAE LEADING TO TREATMENT DOSE REDUCTION BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) |
| TABLE 14.3.1.10C SUMMARY OF TEAE LEADING TO TREATMENT DOSE REDUCTION BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE) |
| TABLE 14.3.1.10D SUMMARY OF TEAE LEADING TO TREATMENT DOSE REDUCTION BY SOC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) |
| TABLE 14.3.1.11A SUMMARY OF TEAE LEADING TO DEATH BY SOC AND PT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) |
| TABLE 14.3.1.11B SUMMARY OF TEAE LEADING TO DEATH BY SOC AND PT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) |
| TABLE 14.3.1.11C SUMMARY OF TEAE LEADING TO DEATH BY SOC AND PT (SAFETY POPULATION IN THE EXTENSION PHASE) |
| TABLE 14.3.1.11D SUMMARY OF TEAE LEADING TO DEATH BY SOC AND PT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) |

| TABLE 14.3.1.12A SUMMARY OF TREATMENT EMERGENT AESI BY SOC AND PT (SAFETY POPULATION IN THE | |
|---|---|
| Stage 1 PK Phase)6 | 57 |
| TABLE 14.3.1.12B SUMMARY OF TREATMENT EMERGENT AESI BY SOC AND PT (SAFETY POPULATION IN THE | |
| STAGE 2 PK PHASE)6 | 57 |
| TABLE 14.3.1.12C SUMMARY OF TREATMENT EMERGENT AESI BY SOC AND PT (SAFETY POPULATION IN THE | |
| Extension Phase) | 57 |
| TABLE 14.3.1.12D SUMMARY OF TREATMENT EMERGENT AESI BY SOC AND PT (SAFETY POPULATION IN THE | |
| STAGE 3 PK PHASE)6 | |
| $TABLE\ 14.3.1.13A\ SUMMARY\ OF\ TREATMENT\ EMERGENT\ ADVERSE\ EVENTS\ BY\ SOC\ AND\ PT\ AND\ CTCAE\ TOXICIT$ | |
| GRADE (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 58 |
| TABLE 14.3.1.13B SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT AND MAXIMUM | |
| TOXICITY (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 58 |
| TABLE 14.3.1.13C SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY SOC AND PT AND MAXIMUM | |
| TOXICITY (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| $TABLE\ 14.3.1.13D\ SUMMARY\ OF\ TREATMENT\ EMERGENT\ ADVERSE\ EVENTS\ BY\ SOC\ AND\ PT\ AND\ CTCAE\ TOXICIT$ | |
| GRADE (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 59 |
| TABLE 14.3.1.14A SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY PT (SAFETY POPULATION IN THE | |
| STAGE 1 PK PHASE) | 70 |
| TABLE 14.3.1.14B SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY PT (SAFETY POPULATION IN THE | |
| STAGE 2 PK PHASE) | /0 |
| TABLE 14.3.1.14C SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY PT (SAFETY POPULATION IN THE | |
| EXTENSION PHASE) | /0 |
| TABLE 14.3.1.14D SUMMARY OF TREATMENT EMERGENT ADVERSE EVENTS BY PT (SAFETY POPULATION IN THE | |
| STAGE 3 PK PHASE) | |
| TABLE 14.3.1.15A LISTING OF SERIOUS TEAES DURING PK PHASE (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | - |
| | 12 |
| TABLE 14.3.1.15B LISTING OF SERIOUS TEAES DURING THE PK PHASE (SAFETY POPULATION IN THE STAGE 2 PK | |
| PHASE) | 12 |
| TABLE 14.3.1.15C LISTING OF SERIOUS TEAES DURING THE EXTENSION PHASE (SAFETY POPULATION IN THE | |
| EXTENSION PHASE) | 12 |
| TABLE 14.3.1.15D LISTING OF SERIOUS TEAES DURING THE PK PHASE (SAFETY POPULATION IN THE STAGE 3 PK | |
| PHASE) | |
| TABLE 14.3.1.16A LISTING OF DEATHS DURING THE PK PHASE (SAFETY POPULATION IN THE STAGE 1 PK PHASE)7 | |
| TABLE 14.3.1.16B LISTING OF DEATHS DURING THE PK PHASE (SAFETY POPULATION IN THE STAGE 2 PK PHASE)7 | /2 |
| TABLE 14.3.1.16C LISTING OF DEATHS DURING THE EXTENSION PHASE (SAFETY POPULATION IN THE EXTENSION | |
| PHASE) | |
| TABLE 14.3.1.16D LISTING OF DEATHS DURING THE PK PHASE (SAFETY POPULATION IN THE STAGE 3 PK PHASE)7 | 13 |
| TABLE 14.3.1.17C LISTING OF TEAE LEADING TO DOSE INTERRUPTION DURING THE EXTENSION PHASE (SAFETY | |
| POPULATION IN THE EXTENSION PHASE) | 13 |
| TABLE 14.3.1.17D LISTING OF TEAE LEADING TO DOSE INTERRUPTION DURING THE PK PHASE (SAFETY | |
| POPULATION IN THE STAGE 3 PK PHASE) | |
| TABLE 14.3.1.18A LISTING OF TEAE LEADING TO DOSE REDUCTION DURING THE PK PHASE (SAFETY POPULATION | |
| IN THE STAGE 1 PK PHASE) | 13 |
| TABLE 14.3.1.18B LISTING OF TEAE LEADING TO DOSE REDUCTION DURING THE PK PHASE (SAFETY POPULATION | 70 |
| IN THE STAGE 2 PK PHASE) | 13 |
| TABLE 14.3.1.18C LISTING OF TEAE LEADING TO DOSE REDUCTION DURING THE EXTENSION PHASE (SAFETY | 70 |
| POPULATION IN THE EXTENSION PHASE) | |
| · | |
| IN THE STAGE 3 PK PHASE) | ) |

| TABLE 14.3.1.19A LISTING OF TEAE LEADING TO TREATMENT DISCONTINUATION DURING THE PK PHASE (SAI | |
|---|---|
| POPULATION IN THE STAGE 1 PK PHASE) | |
| TABLE 14.3.1.19B LISTING OF TEAE LEADING TO TREATMENT DISCONTINUATION DURING THE PK PHASE (SAF | ETY |
| POPULATION IN THE STAGE 2 PK PHASE) | |
| TABLE 14.3.1.19C LISTING OF TEAE LEADING TO TREATMENT DISCONTINUATION DURING THE EXTENSION PH. | ASE |
| (SAFETY POPULATION IN THE EXTENSION PHASE) | 73 |
| TABLE 14.3.1.19D LISTING OF TEAE LEADING TO TREATMENT DISCONTINUATION DURING THE PK PHASE (SAI | FETY |
| POPULATION IN THE STAGE 3 PK PHASE) | 73 |
| TABLE 14.3.1.20D SUMMARY OF INCIDENCE OF COVID-19 RELATED ADVERSE EVENTS OVER TIME (SAFETY | |
| POPULATION IN THE STAGE 3 PK PHASE) | 74 |
| TABLE 14.3.1.21D SUMMARY OF INCIDENCE OF COVID-19 RELATED ADVERSE EVENTS OVER TIME BY GENDE | R |
| (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 75 |
| TABLE 14.3.1.22D SUMMARY OF INCIDENCE OF ADVERSE EVENTS OVER TIME BY AGE GROUP (SAFETY POPULA | |
| IN THE STAGE 3 PK PHASE) | |
| TABLE 14.3.4.1A SUMMARY OF STUDY TREATMENT EXPOSURE DURING THE PK PHASE (SAFETY POPULATION I | |
| STAGE 1 PK PHASE) | |
| TABLE 14.3.4.1B SUMMARY OF STUDY TREATMENT EXPOSURE DURING THE PK PHASE (SAFETY POPULATION II | |
| STAGE 2 PK PHASE) | |
| TABLE 14.3.4.1C SUMMARY OF STUDY TREATMENT EXPOSURE DURING THE EXTENSION PHASE (SAFETY | |
| POPULATION IN THE EXTENSION PHASE) | 77 |
| TABLE 14.3.4.1D SUMMARY OF STUDY TREATMENT EXPOSURE DURING THE PK PHASE (SAFETY POPULATION I | |
| STAGE 3 PK PHASE) | |
| TABLE 14.3.4.2C SUMMARY OF NIRAPARIB DOSE BY CYCLE (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| TABLE 14.3.4.3.1C SUMMARY AND CHANGE FROM BASELINE OF SELECT HEMATOLOGY PARAMETERS BY VISIT | |
| DURING THE EXTENSION PHASE (SAFETY POPULATION IN THE EXTENSION PHASE) | 80 |
| TABLE 14.3.4.3.2C SHIFT SUMMARY OF SELECT HEMATOLOGY PARAMETERS DURING THE EXTENSION PHASE | |
| (SAFETY POPULATION IN THE EXTENSION PHASE). | 81 |
| TABLE 14.3.4.4.1C SUMMARY AND CHANGE FROM BASELINE OF SELECT CHEMISTRY PARAMETERS BY VISIT DU | |
| THE EXTENSION PHASE (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| TABLE 14.3.4.4.2C SHIFT SUMMARY OF SELECT CHEMISTRY PARAMETERS IN MAXIMUM TOXICITY GRADE DUR | |
| THE EXTENSION PHASE (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| TABLE 14.4.1C SUMMARY OF IMPORTANT PROTOCOL DEVIATIONS (SAFETY POPULATION IN THE EXTENSION PH | |
| TABLE 14.4.1D SUMMARY OF IMPORTANT PROTOCOL DEVIATIONS FOR THE PK PHASE OCCURRING THROUGH E | END OI |
| TREATMENT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.1A DISPOSITION FOR PK PHASE (ALL PATIENTS ENROLLED IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.1B DISPOSITION FOR PK PHASE (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.1C DISPOSITION FOR OPEN-LABEL EXTENSION PHASE (ALL PATIENTS ENROLLED FOR THE EXTENSION PHASE) | |
| Phase) | |
| LISTING 16.2.1D DISPOSITION FOR PK PHASE (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.1.2A REASONS FOR SCREEN FAILURE (PATIENTS WHO FAILED SCREENING IN THE STAGE 1 PK PHA | |
| LISTING 16.2.1.2B REASONS FOR SCREEN FAILURE (PATIENTS WHO FAILED SCREENING IN THE STAGE 2 PK PHA | |
| LISTING 16.2.1.2D REASONS FOR SCREEN FAILURE (PATIENTS WHO FAILED SCREENING IN THE STAGE 3 PK PHA | |
| LISTING 16.2.2A PROTOCOL DEVIATIONS FOR THE PK PHASE (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.2B PROTOCOL DEVIATION FOR THE PK PHASE (SAFETY POPULATION IN THE STAGE 2 PK PHASE). | |
| LISTING 16.2.2C IMPORTANT PROTOCOL DEVIATIONS FOR THE OPEN-LABEL EXTENSION PHASE (SAFETY | |
| POPULATION FOR OPEN-LABEL EXTENSION PHASE) | 80 |
| LISTING 16.2.2.1D IMPORTANT PROTOCOL DEVIATIONS FOR THE PK PHASE OCCURRING THROUGH END OF | |
| TREATMENT (SAFETY POPUL ATION FOR STAGE 3 PK PHASE) | 9( |

| LISTING 16.2.2.2D GSK PROTOCOL DEVIATIONS RELATED TO COVID-19 (SAFETY POPULATION FOR STAGE 3 | PK |
|---|---|
| Phase) | 91 |
| LISTING 16.2.3A STUDY POPULATIONS FOR THE PK PHASE (ALL PATIENTS ENROLLED IN THE STAGE 1 PK PHA | ASE)92 |
| LISTING 16.2.3B STUDY POPULATIONS FOR THE PK PHASE (ALL PATIENTS SCREENED IN THE STAGE 2 PK PHA | SE)92 |
| LISTING 16.2.3C STUDY POPULATIONS FOR THE OPEN-LABEL EXTENSION PHASE (ALL PATIENTS ENROLLED IN | N THE |
| EXTENSION PHASE) | 93 |
| LISTING 16.2.3D STUDY POPULATIONS FOR THE PK PHASE (ALL PATIENTS ENROLLED IN THE STAGE 3 PK PHA | ASE)94 |
| LISTING 16.2.4.1A DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 95 |
| LISTING 16.2.4.1B DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 95 |
| LISTING 16.2.4.1C DEMOGRAPHICS (SAFETY POPULATION IN THE EXTENSION PHASE) | 95 |
| LISTING 16.2.4.1D DEMOGRAPHICS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 95 |
| LISTING 16.2.4.2A MEDICAL HISTORY (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 96 |
| LISTING 16.2.4.2B MEDICAL HISTORY (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 96 |
| LISTING 16.2.4.2C MEDICAL HISTORY (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.4.2D MEDICAL HISTORY (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.4.3A PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.4.3B PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.4.3C PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.4.3D PRIOR ANTI-CANCER TREATMENT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.4.4A PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.4.4B PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.4.4C PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.4.4D PRIMARY CANCER HISTORY (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.4.5A PRIOR/CONCOMITANT RADIOTHERAPY (SAFETY POPULATION IN THE STAGE 1 PK PHASE). | |
| LISTING 16.2.4.5B PRIOR/CONCOMITANT RADIOTHERAPY (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.4.5C PRIOR/CONCOMITANT RADIOTHERAPY (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.4.5D PRIOR/CONCOMITANT RADIOTHERAPY (SAFETY POPULATION IN THE STAGE 3 PK PHASE). | |
| LISTING 16.2.5.1B PRIOR AND CONCOMITANT MEDICATIONS (SAFETY POPULATION IN THE STAGE 2 PK PHASE | |
| LISTING 16.2.5.1C PRIOR AND CONCOMITANT MEDICATIONS (SAFETY POPULATION IN THE EXTENSION PHASE | * |
| LISTING 16.2.5.1D PRIOR AND CONCOMITANT MEDICATIONS (SAFETY POPULATION IN THE STAGE 3 PK PHASI | * |
| LISTING 16.2.5.2A PRIOR/CONCOMITANT PROCEDURES DURING PK PHASE (SAFETY POPULATION IN THE STAGE | |
| Phase) | |
| LISTING 16.2.5.2B PRIOR/CONCOMITANT PROCEDURES DURING THE PK PHASE (SAFETY POPULATION IN THE | STAGE 2 |
| PK PHASE) | |
| LISTING 16.2.5.2C PRIOR/CONCOMITANT PROCEDURES DURING THE EXTENSION PHASE (SAFETY POPULATION | |
| EXTENSION PHASE) | |
| LISTING 16.2.5.2D PRIOR/CONCOMITANT PROCEDURES DURING THE PK PHASE (SAFETY POPULATION IN THE | |
| 3 PK PHASE) | |
| LISTING 16.2.5.3A PRIOR AND CONCOMITANT TRANSFUSIONS (SAFETY POPULATION IN THE STAGE 1 PK PHAS | |
| LISTING 16.2.5.3B PRIOR AND CONCOMITANT TRANSFUSIONS (SAFETY POPULATION IN THE STAGE 2 PK PHAS | |
| LISTING 16.2.5.3C PRIOR AND CONCOMITANT TRANSFUSIONS (SAFETY POPULATION IN THE EXTENSION PHASE | |
| LISTING 16.2.5.3D PRIOR AND CONCOMITANT TRANSFUSIONS (SAFETY POPULATION IN THE STAGE 3 PK PHAS | * |
| LISTING 16.2.5.4A PRIOR AND CONCOMITANT GROWTH FACTORS (SAFETY POPULATION IN THE STAGE 1 PK P | |
| LISTING 16.2.5.4B PRIOR AND CONCOMITANT GROWTH FACTORS (SAFETY POPULATION IN THE STAGE 2 PK P | |
| LISTING 16.2.5.4C PRIOR AND CONCOMITANT GROWTH FACTORS (SAFETY POPULATION IN THE EXTENSION PI | |
| | · |

| LISTING 16.2.5.4D PRIOR AND CONCOMITANT GROWTH FACTORS (SAFETY POPULATION IN THE STAGE 3 PK PHASI | |
|---|---|
| LISTING 16.2.5.5A STUDY TREATMENT (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.5.5B STUDY TREATMENT (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.5.5C STUDY TREATMENT (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.5.5D STUDY TREATMENT (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.5.6B SUBSEQUENT ANTI-CANCER THERAPY (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.5.6C SUBSEQUENT ANTI-CANCER THERAPY (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.5.6D MEAL STATUS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| $LISTING~16.2.6.1C~Investigator~Assessment~of~Response~(Safety~Population~in~the~Extension~Phase) \dots \\$ | 110 |
| LISTING 16.2.7.1A ADVERSE EVENTS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.7.1B ADVERSE EVENTS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 111 |
| LISTING 16.2.7.1C ADVERSE EVENTS (SAFETY POPULATION IN THE EXTENSION PHASE) | 111 |
| LISTING 16.2.7.1D ADVERSE EVENTS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 111 |
| LISTING 16.2.8.1.1A HEMATOLOGY RESULTS IN THE PK PHASE (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 112 |
| LISTING 16.2.8.1.1B HEMATOLOGY RESULTS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 112 |
| LISTING 16.2.8.1.1C HEMATOLOGY RESULTS (SAFETY POPULATION IN THE EXTENSION PHASE) | 112 |
| LISTING 16.2.8.1.1D HEMATOLOGY RESULTS THROUGH THE PK END OF TREATMENT VISIT (SAFETY POPULATION | IN |
| THE STAGE 3 PK PHASE) | 112 |
| LISTING 16.2.8.1.2A CHEMISTRY RESULTS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 112 |
| LISTING 16.2.8.1.2B CHEMISTRY RESULTS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.8.1.2C CHEMISTRY RESULTS (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.8.1.2D CHEMISTRY RESULTS THROUGH THE PK END OF TREATMENT VISIT (SAFETY POPULATION IN | |
| THE STAGE 3 PK PHASE) | |
| LISTING 16.2.8.1.3A URINALYSIS RESULTS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.8.1.3B URINALYSIS RESULTS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.8.1.3C URINALYSIS RESULTS (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.8.1.3D URINALYSIS RESULTS THROUGH THE PK END OF TREATMENT VISIT (SAFETY POPULATION IN | |
| THE STAGE 3 PK PHASE) | |
| LISTING 16.2.8.1.4C LIVER FUNCTION TESTS – POTENTIAL HY'S LAW CASES (SAFETY POPULATION IN THE | |
| EXTENSION PHASE) | 113 |
| LISTING 16.2.8.2A VITAL SIGNS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.8.2B VITAL SIGNS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.8.2C VITAL SIGNS (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.8.2D VITAL SIGNS THROUGH THE PK END OF TREATMENT VISIT (SAFETY POPULATION IN THE STAGI | |
| PK PHASE). | |
| LISTING 16.2.8.3A ECG RESULTS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.8.3B ECG RESULTS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.8.3C ECG RESULTS (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.8.3D ECG RESULTS (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | |
| LISTING 16.2.8.4A ECOG PERFORMANCE STATUS (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | |
| LISTING 16.2.8.4B ECOG PERFORMANCE STATUS (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | |
| LISTING 16.2.8.4C ECOG PERFORMANCE STATUS (SAFETY POPULATION IN THE EXTENSION PHASE) | |
| LISTING 16.2.8.4D ECOG PERFORMANCE STATUS THROUGH THE PK END OF TREATMENT VISIT (SAFETY | 110 |
| POPULATION IN THE STAGE 3 PK PHASE) | 116 |
| LISTING 16.2.8.5A BASELINE PHYSICAL EXAMINATION FINDINGS (SAFETY POPULATION IN THE STAGE 1 PK PHASE | |
| EISTING TO.2.6.3A DASELINE I ITTSICAL LAAWINATION I INDINGS (SAFETT TOTOLATION IN THE STAGE I TK I HASE | - |
| LISTING 16.2.8.5B BASELINE PHYSICAL EXAMINATION FINDINGS (SAFETY POPULATION IN THE STAGE 2 PK PHASE | |
| EISTING 10.2.6.3D DASELINE I ITTSICAL EXAMINATION I INDINGS (GALETT I OF CLATION IN THE STAGE 2 I K I HASE | |

| LISTING 16.2.8.5C BASELINE PHYSICAL EXAMINATION FINDINGS (SAFETY POPULATION IN THE EXTENSION P | HASE) |
|---|---|
| | 117 |
| LISTING 16.2.8.5D BASELINE PHYSICAL EXAMINATION FINDINGS (SAFETY POPULATION IN THE STAGE 3 PK | Phase) |
| | 117 |
| LISTING 16.2.8.6A PREGNANCY TEST (SAFETY POPULATION IN THE STAGE 1 PK PHASE) | 118 |
| LISTING 16.2.8.6B PREGNANCY TEST (SAFETY POPULATION IN THE STAGE 2 PK PHASE) | 118 |
| LISTING 16.2.8.6C PREGNANCY TEST (SAFETY POPULATION IN THE EXTENSION PHASE) | 118 |
| LISTING 16.2.8.6D PREGNANCY TEST (SAFETY POPULATION IN THE STAGE 3 PK PHASE) | 118 |
| LISTING 16.2.9.2D LISTING OF COVID-19 ASSESSMENTS AND SYMPTOM ASSESSMENTS FOR PATIENTS WITH | COVID- |
| 19 Adverse Events (Safety Population in the Stage 3 PK Phase) | 119 |

# **TABLES**

#### General guidelines:

Tables will be provided for the Stage 1 PK Phase, Stage 2 PK Phase, Stage 3 PK Phase and the Open-Label Extension Phase.

For the PK Phase (Stage 1, Stage 2 and Stage 3):

- Treatment=Sequence and Overall, in general. For PK and AE data, please see mock tables.
- Population=Safety Population in Stage 1 PK (Stage 2 PK or Stage 3 PK) Phase, unless otherwise specified.
- PK Phase Data:
  - o For patients who do not continue to Extension Phase, PK Phase is any data collected.
  - o For patients who do continue to Extension Phase,
    - AEs prior to first dose in Extension Phase
    - Prior meds/procedures/etc. prior to first dose in PK Phase
    - Concomitant meds meds prior to first dose in Extension Phase.
- Assessments (Labs, ECGs, Vitals, ECOG, PE, etc.) use visit to identify data.

#### For the Extension Phase:

- Treatment=Niraparib Tablet or Capsule (regardless of starting dose); Summarize by Tablet; Capsule; Overall, unless otherwise specified.
- Population=Safety Population in the Open-Label Extension Phase (i.e., those who receive at least 1 dose), unless otherwise specified.
- Extension Phase Data:
  - o For patients who do not continue to Extension Phase, there is no Extension Phase data.
  - o For patients who do continue to Extension Phase,
    - AEs on or after first dose in Extension Phase
    - Prior meds/procedures/etc. prior to first dose in Extension Phase
    - Concomitant meds meds on or after the first dose in Extension Phase
    - Assessments (Labs, ECGs, Vitals, ECOG, PE, etc.) use visit to identify data.

Sort order: All AE tabulations, unless otherwise specified, will be ordered in terms of decreasing frequency for SOC (alphabetically for SOCs with the same number of AEs reported), and decreasing frequency for PT within SOC (alphabetically for PTs with the same number of AEs reported within a SOC) considering the overall rate.


Protocol No: XXXXX

#### Table 14.1.1A

Subject Disposition in the PK Phase (All Patients in the Stage 1 PK Phase)

| Parameter | Statistic | Sequence<br>TABLET/CAPSULE | Sequence<br>CAPSULE/TABLET | Overall |
|---|---|---|---|---|
| Number of Patients | | | | |
| Screened | n | | | XX |
| Randomized | n | Х | Х | Х |
| Received Tablet | n | Х | Х | Х |
| Received Capsule | n | Х | Х | Х |
| Received Both Tablet and Capsule | n | Х | Х | Х |
| PK Phase Safety Population | n | Х | Х | Х |
| Completed PK Phase | n | X | Х | X |
| Discontinuation from PK Phase | n | X | X | X |
| Reason1 | n | х | х | Х |
| Reason2 | n | Х | Х | X |
| Participate in Extension Phase | n | X | X | X |
| Discontinuation from Study Prior to Entering the Extension Phase | | | | |
| Reason1 | n | XX | XX | XX |
| Reason2 | n | XX | XX | XX |

Source: Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

Only include DC from study for those patients who do not enter the Extension Phase.

Table 14.1.1B

Subject Disposition in the PK Phase (All Patients in the Stage 2 PK Phase)

| Parameter | Statistic | Sequence<br>TABLET/CAPSULE | Sequence<br>CAPSULE/TABLET | Overall |
|---|---|---|---|---|
| Number of Patients | | | | |
| Screened | n | | | XX |
| Randomized | n | X | Х | X |
| Not Treated | n | Х | Х | X |
| Received Tablet | n | Х | Х | X |
| Received Capsule | n | X | Х | X |
| Received Both Tablet and Capsule | n | Х | Х | X |
| PK Phase Safety Population | n | X | Х | X |
| Completed PK Phase | n | X | Х | X |
| Discontinuation from PK Phase [1] | n | X | Х | X |
| Reason 1 | n | X | Х | X |
| Reason 2 | n | X | Х | X |
| Participate in Extension Phase | n | Х | Х | X |
| Discontinuation from Study Prior to Entering the Extension Phase | | | • | |
| Reason 1 | n | XX | XX | XX |
| Reason 2 | n | xx | XX | XX |

[1] Includes patients in the Safety Population (i.e., treated patients) only.

Source: Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

[Programming Notes]


Only include DC from study for those patients who do not enter the Extension Phase.

TESARO Inc. Confidential Page 1 of x Protocol No: XXXXX

Table 14.1.1C

Subject Disposition in the Extension Phase (All Patients in the Extension Phase)

| Parameter | Statistic | Niraparib | Niraparib | Niraparib |
|---|---|---|---|---|
| | | Tablet | Capsule | Overall |
| Number of Patients | | | | |
| Dosed | n | xx | XX | XX |
| Discontinued Treatment After Receiving at Least 1 Dose | n | XX | XX | XX |
| Reason 1 | n | XX | XX | XX |
| Reason 2 | n | XX | XX | XX |
| Discontinued Study | n | XX | XX | XX |
| Reason 1 | n | XX | XX | XX |
| Reason 2 | n | XX | XX | XX |

Source: Listing XXXXXXXXX, Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


Table 14.1.1D

Subject Disposition in the PK Phase (All Patients in the Stage 3 PK Phase)

| Parameter | Statistic | Sequence<br>NIRAPARIB TABLET<br>FASTED/FED | Sequence<br>NIRAPARIB TABLET<br>FED/FASTED | OVERALL |
|---|---|---|---|---|
| Number of Patients | | | | |
| Screened [1] | n | | | XX |
| Randomized | n | Х | Х | Х |
| Not Treated | n | Х | Х | Х |
| Received Tablet in Fasted State | n | Х | Х | Х |
| Received Tablet in Fed State | n | Х | Х | Х |
| Received Tablet in Both Fasted and Fed State | n | Х | Х | Х |
| PK Phase Safety Population | n | Х | х | X |
| Completed PK Phase | n | х | х | X |
| Discontinuation from PK Phase [2] | n | Х | Х | Х |
| Reason 1 | n | Х | Х | Х |
| Reason 2 | n | х | х | X |
| Participate in Extension Phase | n | х | х | X |
| Discontinuation from Study Prior to Entering the Extension Phase | | | | |
| Reason 1 | n | xx | xx | XX |
| Reason 2 | n | xx | xx | XX |

<sup>[1]</sup> Patient xxxxxx-xxxx (Screen Failure ID: XXi) and xxxxxx-xxxx (Screen Failure ID: YYi) re-screened and reconsented after screen failure are counted twice in Screening.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Note]

XXi/YYi is ID that was SF.

Programming, please note footnote references changed order in the shell and footer.

<sup>[2]</sup> Includes patients in the Safety Population (i.e., treated patients) only.

TESARO Inc. Confidential Page 1 of x Protocol No: XXXXX

Table 14.1.2A

Demographics (Safety Population in the Stage 1 PK Phase)

| Parameter | Statistic | Sequence<br>TABLET/CAPSULE | Sequence<br>CAPSULE/TABLET | OVERALL |
|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) |
| Age (yrs) | n | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | XX.X |
| | Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| Age Group | | | | |
| 18 -< 65 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 65 -< 75 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ≥ 75 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sex | | | | |
| Male | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race | | | | |
| White | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| African American | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| American Indian or Alaska Native | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Native Hawaiian or other Pacific Islander | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity | | | | |
| Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Table 14.1.2.1A Demographics (BA Evaluable Population in the Stage 1 PK Phase)

Table 14.1.2.1B Demographics (Safety Population in the Stage 2 PK Phase)
Table 14.1.2.2B Demographics (BE Evaluable Population in the Stage 2 PK Phase)

Table 14.1.2C Demographics (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for Tablet; Capsule; Overall Table 14.1.2.1D Demographics (Safety Population in the Stage 3 PK Phase)

Table 14.1.2.2D Demographics (FE Evaluable Population in the Stage 3 PK Phase)

• Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL.


# Table 14.1.3A

Baseline Characteristics (Safety Population in the Stage 1 PK Phase)

| Parameter | Statistic | Sequence | Sequence | |
|---|---|---|---|---|
| | | TABLET/CAPSULE | CAPSULE/TABLET | OVERALL |
| | | (N=xx) | (N=xx) | (N=xx) |
| Weight (kg) | n | xx | xx | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| II a de alba de de acceptante de la companya della companya de la companya della | | | | |
| Height (cm) | n<br>Maria (GD) | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X |
| | Min, Max | xx, xx | XX, XX | XX, XX |
| BMI (kg/m <sup>2</sup> ) | n | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| ECOC Danfarmana Chahua | <u>_</u> | | | |
| ECOG Performance Status | (0) | / | ( | / |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ± | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

ECOG = Eastern Cooperative Oncology Group:

0=Fully active, able to carry on all pre-disease performance without restriction

1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature

2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours

3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours

4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair

Source: Program: XXXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Table 14.1.3.1A Baseline Characteristics (BA Evaluable Population in the Stage 1 PK Phase)

Table 14.1.3.1B Baseline Characteristics (Safety Population in the Stage 2 PK Phase)

Table 14.1.3.2B Baseline Characteristics (BE Evaluable Population in the Stage 2 PK Phase)

Table 14.1.3C Baseline Characteristics (Safety Population in the Extension Phase)

- Summarize Extension Phase Data with columns for Tablet; Capsule; Overall Table 14.1.3.1D Baseline Characteristics (Safety Population in the Stage 3 PK Phase)
- Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL Table 14.1.3.2D Baseline Characteristics (FE Evaluable Population in the Stage 3 PK Phase)
  - Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL

### Table 14.1.4A

Primary Cancer History (Safety Population in the Stage 1 PK Phase)

| Parameter | Statistic | Sequence | Sequence | |
|---|---|---|---|---|
| | | TABLET/CAPSULE | CAPSULE/TABLET | OVERALL |
| | | (N=xx) | (N=xx) | (N=xx) |
| Tumor Type | | | | |
| Xxxxxxx | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Xxxxxxx | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Xxxxxxxx | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time from first diagnosis to informed consent (years) | n | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x |
| | Min, Max | XX, XX | XX, XX | xx, xx |
| Cancer Stage (most recent) | | | | |
| Locally advanced | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Metastatic | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of prior lines of therapy | | | | |
| 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=6 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any prior radiotherapy | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Table 14.1.4B Primary Cancer History (Safety Population in the Stage 2 PK Phase)

Table 14.1.4C Primary Cancer History (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for Tablet; Capsule; Overall Table 14.1.4D Primary Cancer History (Safety Population in the Stage 3 PK Phase)

• Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL


Table 14.1.5A

Prior Anti-Cancer Treatment (Safety Population in the Stage 1 PK Phase)

| Preferred Term | Statistic | Sequence<br>TABLET/CAPSULE<br>(N=xx) | Sequence<br>CAPSULE/TABLET<br>(N=xx) | OVERALL<br>(N=xx) |
|---|---|---|---|---|
| Agent 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Agent 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Agent 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# [Programming Notes]

Sort by decreasing frequency in the OVERALL column.

#### Repeat for:

Table 14.1.5B Prior Anti-Cancer Treatment (Safety Population in the Stage 2 PK Phase)

Table 14.1.5C Prior Anti-Cancer Treatment (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for Tablet; Capsule; Overall

Table 14.1.5D Prior Anti-Cancer Treatment (Safety Population in the Stage 3 PK Phase)

• Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED AND OVERALL.

Table 14.1.6A

Medical History (Safety Population in the Stage 1 PK Phase)

| System Organ Class | Statistic | Sequence | Sequence | |
|--------------------|-----------|----------------|----------------|-----------|
| Preferred Term | | TABLET/CAPSULE | CAPSULE/TABLET | OVERALL |
| | | (N=xx) | (N=xx) | (N=xx) |
| Any condition | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (웅) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

[Programming Notes]

Sort alphabetically by SOC/PT.

#### Repeat for:

Table 14.1.6B Medical History (Safety Population in the Stage 2 PK Phase)

Table 14.1.6C Medical History (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for Tablet; Capsule; Overall.

Table 14.1.6D Medical History (Safety Population in the Stage 3 PK Phase)

• Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL

Table 14.1.7A

Prior Medications by ATC and PT (Safety Population in the Stage 1 PK Phase)

| ATC (Level 3) | Statistic | Sequence | Sequence | |
|---|---|---|---|---|
| Preferred Term | | TABLET/CAPSULE | CAPSULE/TABLET | OVERALL |
| | | (N=xx) | (N=xx) | (N=xx) |
| Any prior medication | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Prior medications are any medications with a start date earlier than the first dose date of study treatment and are coded using WHO Drug Dictionary version YYYYMM. Study treatment, prior anti-cancer treatments for primary cancer, transfusions and growth factors are not included.

## [Programming Notes]

Sort alphabetically by ATC3 and Preferred Term. If there are uncoded terms due to no ATC level 3 term not being available, add footnote for uncoded term: [1] ATC level 3 term is not available through WHO Drug Dictionary.

#### Repeat for:

Table 14.1.7B Prior Medications by ATC and PT (Safety Population in the Stage 2 PK Phase)

Table 14.1.7C Prior Medications by ATC and PT (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for Tablet; Capsule; Overall

### [Programming Notes]

- Footnote Extension Phase: Prior medications are any medications, other than study treatments and pre-medications for study treatment, with a start date earlier than the first dose date of study treatment during the Extension Phase and are coded using WHO Drug Dictionary version YYYYMM.
- Prior anti-cancer treatments for primary cancer are not included.

Table 14.1.7D Prior Medications by ATC and PT (Safety Population in the Stage 3 PK Phase)

• Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL


Table 14.1.8A

Concomitant Medications by ATC and PT (Safety Population in the Stage 1 PK Phase)

| ATC (Level 3) | Statistic | Sequence | Sequence | |
|---|---|---|---|---|
| Preferred Term | | TABLET/CAPSULE | CAPSULE/TABLET | OVERALL |
| | | (N=xx) | (N=xx) | (N=xx) |
| Any concomitant medication | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Concomitant medications are any medications being taken on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase. They are coded using WHO Drug Dictionary version YYYYMM.

#### [Programming Notes]

Sort alphabetically by ATC3 and Preferred Term. If there are uncoded terms due to no ATC level 3 term not being available, add footnote for uncoded term: [1] ATC level 3 term is not available through WHO Drug Dictionary.

## Repeat for:

Table 14.1.8.1B Concomitant Medications by ATC and PT (Safety Population in the Stage 2 PK Phase)

Table 14.1.8.2B Concomitant Medications During the PK Collection Period by ATC and PT (BE Evaluable Population in the Stage 2 PK Phase)

• Footnote: Concomitant medications during the PK collection period are any concomitant medications taken between the first PK-draw until the last PK-draw. They are coded using WHO Drug Dictionary version YYYYMM.

Table 14.1.8C Concomitant Medications by ATC and PT (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for Tablet; Capsule; Overall

### [Programming Notes]

• Footnote - Extension Phase: Concomitant medications are any medications being taken on or after the initial study treatment dosing date during the Extension Phase through 30 days after the last dose. They are coded using WHO Drug Dictionary version YYYYMM.

Table 14.1.8D Concomitant Medications by ATC and PT (Safety Population in the Stage 3 PK Phase)

- Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL
- Footnote Stage 3: Concomitant medications are any medications being taken on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase. They are coded using WHO Drug Dictionary version YYYYMM.


Table 14.1.9A

Concomitant Transfusions and Growth Factors (Safety Population in the Stage 1 PK Phase)

| Parameter | Statistic | Sequence<br>TABLET/CAPSULE<br>(N=xx) | Sequence<br>CAPSULE/TABLET<br>(N=xx) | OVERALL<br>(N=xx) |
|---|---|---|---|---|
| Any Concomitant Transfusions | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Red Blood Cells | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Platelet | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Concomitant Growth Factors | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| G-CSF | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GM-CSF | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Recombinant Erythropoietin | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Concomitant transfusions or growth factors are any transfusion or growth factor given on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose for those not continuing into the Extension Phase.

## Repeat for:

Table 14.1.9B Concomitant Transfusions and Growth Factors (Safety Population in the Stage 2 PK Phase)

Table 14.1.9C Concomitant Transfusions and Growth Factors (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for Tablet; Capsule; Overall

#### [Programming Notes]

• Footnote - Extension Phase: Concomitant transfusions or growth factors are any transfusion or growth factor given on or after the initial study treatment dosing date during the Extension Phase through 30 days after the last dose.

Table 14.1.9D Concomitant Transfusions and Growth Factors (Safety Population in the Stage 3 PK Phase)

- Summarize Stage 3 data by Sequence with columns for NIRAPARIB TABLET FASTED/FED, NIRAPARIB TABLET FED/FASTED and OVERALL
- Footnote Stage 3: Concomitant transfusions or growth factors are any transfusion or growth factor given on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose for those not continuing into the Extension Phase.

Table 14.3.1.1.1A

Overall Summary of Treatment Emergent Adverse Events (Safety Population in the Stage 1 PK Phase)

| | TABLET [1] | CAPSULE [2] | FU/Ext Screening | Total [4] |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | [3] (N=xx) | (N=xx) |
| Any Treatment Emergent Adverse Event (TEAE) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Reduction | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib capsules.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxrtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

## Repeat for:

Table 14.3.1.1.1B Overall Summary of Treatment Emergent Adverse Events (Safety Population in the Stage 2 PK Phase)

Table 14.3.1.1.1C Overall Summary of Treatment Emergent Adverse Events (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for Tablet; Capsule; Overall

# [Programming Notes]

• Sort order: All AE tabulations, unless otherwise specified, will be ordered in terms of decreasing frequency for SOC (alphabetically for SOCs with the same number of AEs reported), and decreasing frequency for PT within SOC (alphabetically for PTs with the same number of AEs reported within a SOC) considering the overall rate.


### Table 14.3.1.1.1D

Overall Summary of Treatment Emergent Adverse Events (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB | NIRAPARIB | FU/Ext | |
|---|---|---|---|---|
| | TABLET FASTED [1] | TABLET FED [2] | Screening [3] | Total [4] |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any Treatment Emergent Adverse Event (TEAE) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Reduction | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any COVID-19 related TEAE Leading to Treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinuation | | | | |
| | | · | | |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

<sup>[3]</sup> For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.

<sup>[4]</sup> Includes TEAEs occurring at any time during the PK Phase.


### Table 14.3.1.1.2A

Overall Summary of Treatment Emergent Adverse Events by Sequence and Period (Safety Population in the Stage 1 PK Phase)

| | | Sequence | | | Sequence | |
|---|---|---|---|---|---|---|
| | | TABLET/CAPSULE | | | CAPSULE/TABLET | |
| | | (N=xx) | | | (N=xx) | |
| | TABLET | CAPSULE | FU/Ext | CAPSULE | TABLET | FU/Ext |
| | Period 1 | Period 2 | Screening | Period 1 | Period 2 | Screening |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any Treatment Emergent Adverse Event (TEAE) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Reduction | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE Leading to Treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinuation | | | | | | |
| Any TEAE Leading to Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# Repeat for:

Table 14.3.1.1.2B Overall Summary of Treatment Emergent Adverse Events by Sequence and Period (Safety Population in the Stage 2 PK Phase)


### Table 14.3.1.1.2D

Overall Summary of Treatment Emergent Adverse Events by Sequence and Period (Safety Population in the Stage 3 PK Phase)

| | | Sequence | | | Sequence | |
|---|---|---|---|---|---|---|
| | NIRAPA | RIB TABLET FAS' | red/fed | NIRAI | PARIB TABLET FED/F | ASTED |
| | | (N=xx) | | | (N=xx) | |
| | NIRAPARIB | NIRAPARIB | | NIRAPARIB | | |
| | TABLET | TABLET | | TABLET | NIRAPARIB | |
| | FASTED | FED | FU/Ext | FED | TABLET FASTED | FU/Ext |
| | Period 1 | Period 2 | Screening | Period 1 | Period 2 | Screening |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any Treatment Emergent Adverse Event (TEAE) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE with CTCAE Toxicity Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE with CTCAE Toxicity Grade ≥ | | | | | | |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Reduction | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE leading to Dose Interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Related TEAE Leading to Treatment | | | | | | |
| Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any TEAE Leading to Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any COVID-19 related TEAE Leading to | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment Discontinuation | | | | | | |

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


### Table 14.3.1.2.1A

Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 1 PK Phase)

| System Organ Class<br>Preferred Term | TABLET [1] (N=xx) | CAPSULE [2]<br>(N=xx) | FU/Ext Screening [3] (N=xx) | Total [4] (N=xx) |
|---|---|---|---|---|
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib capsules.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

For all tables of adverse events by SOC and PT, sort SOCs by descending overall frequency of events reported. Within each SOC, sort PTs by descending overall frequency of events reported.

Table 14.3.1.2.1B Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 2 PK Phase)


Table 14.3.1.2.1C

Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Open-Label Extension Phase)

| | Niraparib | Niraparib | Niraparib |
|--------------------|-----------|-----------|-----------|
| System Organ Class | TABLET | CAPSULE | OVERALL |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 50C2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing XXXXXXXXX, Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# [Programming Notes]

For all tables of adverse events by SOC and PT, sort SOCs by descending overall frequency of events reported. Within each SOC, sort PTs by descending overall frequency of events reported.

Table 14.3.1.2.1D

Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB | NIRAPARIB | FU/Ext | |
|---|---|---|---|---|
| System Organ Class | TABLET FASTED [1] | TABLET FED [2] | Screening [3] | Total [4] |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]


For all tables of adverse events by SOC and PT, sort SOCs by descending overall frequency of events reported. Within each SOC, sort PTs by descending overall frequency of events reported.

Table 14.3.1.2.1.1D

Summary of COVID-19 related Adverse Events by SOC and PT (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB | NIRAPARIB | FU/Ext | |
|---|---|---|---|---|
| System Organ Class | TABLET FASTED [1] | TABLET FED [2] | Screening [3] | Total [4] |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any COVID-19 related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: COVID-19 Case Diagnosis is based on WHO Definition as of DDMMMYYYY.

- [1] Includes COVID-19 related TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes COVID-19 related TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes COVID-19 related TEAEs occurring at any time during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]


For all tables of adverse events by SOC and PT, sort SOCs by descending overall frequency of events reported. Within each SOC, sort PTs by descending overall frequency of events reported.

Select only COVID-19 related TEAEs.


Table 14.3.1.2.2A

Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 1 PK Phase)

| | | Sequence | | | Sequence | |
|---|---|---|---|---|---|---|
| | | TABLET/CAPSULE | | | CAPSULE/TABLET | |
| | | (N=xx) | | | (N=xx) | |
| | TABLET | CAPSULE | FU/Ext | CAPSULE | TABLET | FU/Ext |
| System Organ Class | Period 1 | Period 2 | Screening | Period 1 | Period 2 | Screening |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# [Programming Notes]

For tables of adverse events by SOC and PT by sequence and period, sort alphabetically by SOCs and PTs.

Table 14.3.1.2.2B Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 2 PK Phase)


Table 14.3.1.2.2D

Summary of Treatment Emergent Adverse Events by SOC and PT (Safety Population in the Stage 3 PK Phase)

| | | Sequence | | Sequence | | |
|---|---|---|---|---|---|---|
| | NIRAPA | ARIB TABLET FAST | ED/FED | NIRAP. | NIRAPARIB TABLET FED/FASTED | |
| | | (N=xx) | | | (N=xx) | |
| | NIRAPARIB | NIRAPARIB | | NIRAPARIB | NIRAPARIB | |
| | TABLET FASTED | TABLET FED | FU/Ext | TABLET FASTED | TABLET FED | FU/Ext |
| System Organ Class | Period 1 | Period 2 | Screening | Period 1 | Period 2 | Screening |
| Preferred Term | (N=xx) | (N=xx) (N=xx) (N=xx) (N=xx) | | (N=xx) | | |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

[Programming Notes]

For tables of adverse events by SOC and PT by sequence and period, sort alphabetically by SOCs and PTs.

```
Using Mock Shell (Table 14.3.1.2.1A, Table 14.3.1.2.1B, Table 14.3.1.2.1C, Table 14.3.1.2.1D)
Repeat for:
Table 14.3.1.3A Summary of Related TEAE by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.3B Summary of Related TEAE by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.3C Summary of Related TEAE by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.3D Summary of Related TEAE by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.4A Summary of Serious TEAE by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.4B Summary of Serious TEAE by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.4C Summary of Serious TEAE by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.4D Summary of Serious TEAE by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.5A Summary of Related Serious TEAE by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.5B Summary of Related Serious TEAE by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.5C Summary of Related Serious TEAE by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.5D Summary of Related Serious TEAE by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.6A Summary of TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.6B Summary of TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.6C Summary of TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.6D Summary of TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.7A Summary of Related TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.7B Summary of Related TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 2 PK Phase)
Table 14.3.1.7C Summary of Related TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Extension Phase)
Table 14.3.1.7D Summary of Related TEAE with CTCAE Toxicity Grade ≥3 by SOC and PT (Safety Population in the Stage 3 PK Phase)
Table 14.3.1.8A Summary of TEAE Leading to Treatment Discontinuation by SOC and PT (Safety Population in the Stage 1 PK Phase)
Table 14.3.1.8B Summary of TEAE Leading to Treatment Discontinuation by SOC and PT (Safety Population in the Stage 2 PK Phase)
```


| Table 14.3.1.8C Summary of TEAE Leading to Treatment Discontinuation by SOC and PT (Safety Population in the Extension Phase) |
|---|
| Table 14.3.1.8D Summary of TEAE Leading to Treatment Discontinuation by SOC and PT (Safety Population in the Stage 3 PK Phase) |
| Table 14.3.1.9C Summary of TEAE Leading to Treatment Dose Interruption by SOC and PT (Safety Population in the Extension Phase) |
| Table 14.3.1.10A Summary of TEAE Leading to Treatment Dose Reduction by SOC and PT (Safety Population in the Stage 1 PK Phase) |
| Table 14.3.1.10B Summary of TEAE Leading to Treatment Dose Reduction by SOC and PT (Safety Population in the Stage 2 PK Phase) |
| Table 14.3.1.10C Summary of TEAE Leading to Treatment Dose Reduction by SOC and PT (Safety Population in the Extension Phase) |
| Table 14.3.1.10D Summary of TEAE Leading to Treatment Dose Reduction by SOC and PT (Safety Population in the Stage 3 PK Phase) |
| Table 14.3.1.11A Summary of TEAE Leading to Death by SOC and PT (Safety Population in the Stage 1 PK Phase) |
| Table 14.3.1.11B Summary of TEAE Leading to Death by SOC and PT (Safety Population in the Stage 2 PK Phase) |
| Table 14.3.1.11C Summary of TEAE Leading to Death by SOC and PT (Safety Population in the Extension Phase) |
| Table 14.3.1.11D Summary of TEAE Leading to Death by SOC and PT (Safety Population in the Stage 3 PK Phase) |
| Table 14.3.1.12A Summary of Treatment Emergent AESI by SOC and PT (Safety Population in the Stage 1 PK Phase) |
| Table 14.3.1.12B Summary of Treatment Emergent AESI by SOC and PT (Safety Population in the Stage 2 PK Phase) |
| Table 14.3.1.12C Summary of Treatment Emergent AESI by SOC and PT (Safety Population in the Extension Phase) |
| Table 14.3.1.12D Summary of Treatment Emergent AESI by SOC and PT (Safety Population in the Stage 3 PK Phase) |

Protocol No: XXXX

Table 14.3.1.13A

Summary of Treatment Emergent Adverse Events by SOC and PT and CTCAE Toxicity Grade (Safety Population in the Stage 1 PK Phase)

| | | | FU/Ext | |
|--------------------|------------|-------------|---------------|-----------|
| System Organ Class | TABLET [1] | CAPSULE [2] | Screening [3] | Total [4] |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Grade 1 | | | | |
| • | | | | |
| Grade 5 | | | | |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Grade 1 | | | | |
| • | | | | |
| Grade 5 | | | | |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Grade 1 | | | | |
| • | | | | |
| Grade 5 | | | | |
| •••• | | | | |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib capsules.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

#### Repeat for:

Table 14.3.1.13B Summary of Treatment Emergent Adverse Events by SOC and PT and Maximum Toxicity (Safety Population in the Stage 2 PK Phase)

Table 14.3.1.13C Summary of Treatment Emergent Adverse Events by SOC and PT and Maximum Toxicity (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for Tablet; Capsule; Overall

### [Programming Notes]

For all tables of adverse events by SOC and PT, sort SOCs by descending overall frequency of events reported. Within each SOC, sort PTs by descending overall frequency of events reported. Within each PT, sort by presented maximum toxicity grade.

Protocol No: XXXX

Table 14.3.1.13D

Summary of Treatment Emergent Adverse Events by SOC and PT and CTCAE Toxicity Grade (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB | NIRAPARIB | FU/Ext | |
|---|---|---|---|---|
| System Organ Class | TABLET FASTED [1] | TABLET FED [2] | Screening [3] | Total [4] |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| • | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| Grade 5 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| • | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| Grade 5 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| • | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| Grade 5 | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

|--------------------|--------------|-------------|

Table 14.3.1.14A

Summary of Treatment Emergent Adverse Events by PT (Safety Population in the Stage 1 PK Phase)

| | TABLET [1] | CAPSULE [2] | FU/Ext Screening [3] | Total [4] |
|----------------|------------|-------------|----------------------|-----------|
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib capsules.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

 $\texttt{Source: Program: XXXXXXXXXXXXXXXXXXX}. \ \ \texttt{Output: xxxxxxxxxxxxxxxxx.rtf.} \ \ \texttt{Generated on DDMMMYYYY:HH:MM:SS}$ 

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# Repeat for:

Table 14.3.1.14B Summary of Treatment Emergent Adverse Events by PT (Safety Population in the Stage 2 PK Phase)

Table 14.3.1.14C Summary of Treatment Emergent Adverse Events by PT (Safety Population in the Extension Phase)

• Summarize Extension Phase Data with columns for Tablet; Capsule; Overall

# [Programming Notes]

Sort PTs by descending overall frequency of events reported.


Table 14.3.1.14D

Summary of Treatment Emergent Adverse Events by PT (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB | NIRAPARIB | FU/Ext | |
|---|---|---|---|---|
| Preferred Term | | | · · | Total [4] |
| 110101100 101 | (N=xx) | ABLET FASTED [1] TABLET FED [2] Screening [3] (N=xx) (N=xx) (N=xx) xx (xx.x) | (N=xx) | |
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | | | | |

- [1] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes TEAEs with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.
- [3] For patients not participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase through the End of Study. For patients participating in the Extension Phase, includes TEAEs that began after the end of the PK Phase until the date of first dose in the Extension Phase.
- [4] Includes TEAEs occurring at any time during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


### Table 14.3.1.15A

Listing of Serious TEAEs During PK Phase (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| | | | Start | Stop | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Date | Date | | | | | | | |
| | | | Time/ | Time | | | | | | | |
| | Dosing Period/ | Adverse Event | (Rel | (Rel | | SAE/ | | Action Taken | Other | | |
| Patient | Niraparib | [P]MedDRA Preferred Term | Day | Day | | Reason | | on Study | Action | Relationship | |
| Number | Treatment | [S]System Organ Class | [1]) | [1]) | TEAE? | [2] | Severity | Treatment[3] | Taken | [3] | Outcome |
| | Period 1/ | XXXXXXXXXXXXX | уууу- | уууу- | Y | N | Grade 1 | T: NA | | T: NA | Recovered/ |
| | Capsule | [P]XXXXXXXXXXXXXXXXXX | mm-dd | mm-dd | | | | C: Dose Not | | C: Related | Resolved |
| | | [S]XXXXXXXXXXXXXXXXXX | hh:mm | [x] | | | | Changed | | | |
| | | | [x] | | | | | | | | |
| | Period 2/ | XXXXXXXXXXXXXX | уууу- | уууу- | Y | N | Grade 1 | T: Dose Not | | T: Related | Recovered/ |
| | Tablet | [P]XXXXXXXXXXXXXXXXXX | mm-dd | mm-dd | | | | Changed | | C: NA | Resolved |
| | | [S]XXXXXXXXXXXXXXXXXX | hh:mm | [x] | | | | C: NA | | | |
| | | | [x] | | | | | | | | |
| | PK Safety FU | | | | | | | | | | |

- [1] Relative to the date of first dose in PK Phase.
- [2] Reason for SAE: 1 = Result in death; 2 = Life threatening; 3 = Result in persistent or significant disability/incapacity; 4 = Requires or prolongs hospitalization; 5 = Congenital abnormality/birth defect; 6 = Other medically important event.
- [3] T=Tablet; C=Capsule.

Source: Program: XXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxxrtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

# [Programming notes]

Please add time to Start Date column for PK Phase Stage 2 and Extension Phase.

#### Repeat for:

Table 14.3.1.15B Listing of Serious TEAEs During the PK Phase (Safety Population in the Stage 2 PK Phase)

Table 14.3.1.15C Listing of Serious TEAEs During the Extension Phase (Safety Population in the Extension Phase)

Table 14.3.1.15D Listing of Serious TEAEs During the PK Phase (Safety Population in the Stage 3 PK Phase)

Table 14.3.1.16A Listing of Deaths During the PK Phase (Safety Population in the Stage 1 PK Phase)

Table 14.3.1.16B Listing of Deaths During the PK Phase (Safety Population in the Stage 2 PK Phase)


Table 14.3.1.16C Listing of Deaths During the Extension Phase (Safety Population in the Extension Phase)

Table 14.3.1.16D Listing of Deaths During the PK Phase (Safety Population in the Stage 3 PK Phase)

- Footnote: 'NOTE: Deaths due to progressive disease were not collected as adverse events.'
- Table 14.3.1.17C Listing of TEAE Leading to Dose Interruption During the Extension Phase (Safety Population in the Extension Phase)
- Table 14.3.1.17D Listing of TEAE Leading to Dose Interruption During the PK Phase (Safety Population in the Stage 3 PK Phase)
- Table 14.3.1.18A Listing of TEAE Leading to Dose Reduction During the PK Phase (Safety Population in the Stage 1 PK Phase)
- Table 14.3.1.18B Listing of TEAE Leading to Dose Reduction During the PK Phase (Safety Population in the Stage 2 PK Phase)
- Table 14.3.1.18C Listing of TEAE Leading to Dose Reduction During the Extension Phase (Safety Population in the Extension Phase)
- Table 14.3.1.18D Listing of TEAE Leading to Dose Reduction During the PK Phase (Safety Population in the Stage 3 PK Phase)
- Table 14.3.1.19A Listing of TEAE Leading to Treatment Discontinuation During the PK Phase (Safety Population in the Stage 1 PK Phase)
- Table 14.3.1.19B Listing of TEAE Leading to Treatment Discontinuation During the PK Phase (Safety Population in the Stage 2 PK Phase)
- Table 14.3.1.19C Listing of TEAE Leading to Treatment Discontinuation During the Extension Phase (Safety Population in the Extension Phase)

Table 14.3.1.19D Listing of TEAE Leading to Treatment Discontinuation During the PK Phase (Safety Population in the Stage 3 PK Phase)

#### [Programming Notes]

- Stage 3: Treatment Sequence will be NIRAPARIB TABLET FASTED/FED and NIRAPARIB TABLET FED/FASTED.
- Stage 3: Column 2: Dosing Period/Treatment Treatment should be NIRAPARIB FASTED or NIRAPARIB FED.
- Stage 3: Treatment discontinuation during PK phase add column to record if discontinuation was due to COVID-19 ["COVID-19 Reason" with Options "COVID-19 infection" or "Issues rel. to COVID-19 pandemic"].
- Extension Phase: Replace column for Dosing Period/Treatment with Treatment and Starting Dose.
- Extension Phase: Do not need time with start/stop dates.
- Extension Phase: Footnote: [1] Relative to first dose during the Extension Phase.
- Extension Phase: Add column for Dose at Onset of AE.


Table 14.3.1.20D

Summary of Incidence of COVID-19 Related Adverse Events Over Time (Safety Population in the Stage 3 PK Phase)

| | | NIRAPARIB | NIRAPARIB |
|---|---|---|---|
| | | TABLET FASTED | TABLET FED |
| | Period during COVID-19 | (N=xx) | (N=xx) |
| | Pandemic [1] | n/Patients at Risk (%) | n/Patients at Risk (%) |
| Any COVID-19 Related AE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| _ | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Any COVID-19 Related SAE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Any COVID-19 Related Grade ≥3 AE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |

<sup>[1]</sup> TABLET PK Phase Stage 3 opened to recruitment on DDMMMYYYY, with first patient consented on DDMMMYYYY, placing the start of the recruitment during the COVID-19 pandemic.

Source: Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


Table 14.3.1.21D

Summary of Incidence of COVID-19 Related Adverse Events Over Time by Gender (Safety Population in the Stage 3 PK Phase)

Report on separate page for each: <Gender: Male, Female>

| | Period during COVID-19 | NIRAPARIB<br>TABLET FASTED<br>(N=xx) | NIRAPARIB<br>TABLET FED<br>(N=xx) |
|---|---|---|---|
| | Pandemic [1] | n/Patients at Risk (%) | n/Patients at Risk (%) |
| Any COVID-19 Related AE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Any COVID-19 Related SAE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| Any COVID-19 Related Grade ≥3 AE | Period 1 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |
| | Period 2 | xx/xxx (xx.x%) | xx/xxx (xx.x%) |

<sup>[1]</sup> TABLET PK Phase Stage 3 opened to recruitment on DDMMMYYYY, with first patient consented on DDMMMYYYY, placing the start of the recruitment during the COVID-19 pandemic.

#### Repeat for:

Table 14.3.1.22D Summary of Incidence of Adverse Events Over Time by Age Group (Safety Population in the Stage 3 PK Phase)

• Use the FDAAA age groups <=18, 18-64, >=65

Table 14.3.4.1A

Summary of Study Treatment Exposure During the PK Phase (Safety Population in the Stage 1 PK Phase)

| | Statistic | Sequence<br>TABLET/CAPSULE<br>(N=xx) | Sequence<br>CAPSULE/TABLET<br>(N=xx) | OVERALL<br>(N=xx) |
|---|---|---|---|---|
| # of 100 mg Capsules Received | | | | |
| 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| # of 300 mg Tablets Received | | | | |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

Repeat for:

Table 14.3.4.1B Summary of Study Treatment Exposure During the PK Phase (Safety Population in the Stage 2 PK Phase)


Table 14.3.4.1C

Summary of Study Treatment Exposure During the Extension Phase (Safety Population in the Extension Phase)

| | | Niraparib | Niraparib | Niraparib |
|---|---|---|---|---|
| | | TABLET | CAPSULE | OVERALL |
| Parameters | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Number of Cycles | | | | |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| • • • | | | • • • | |
| ≥ 6 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Duration of Treatment (months) | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | XX.X |
| | Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Duration on Study (months) | n | xx | xx | XX |
| - | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | xx.x |
| | Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Min, Max | xx, xx | XX, XX | xx, xx |
| Total Number of Patients with dose interruption | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total Number of Patients with dose reduction | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total Number of Patients with dose re-escalation | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing XXXXXXXXX, Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

|--------------------|--------------|-------------|

Table 14.3.4.1D

Summary of Study Treatment Exposure During the PK Phase (Safety Population in the Stage 3 PK Phase)

| | Statistic | NIRAPARIB | NIRAPARIB | |
|------------------------------|-----------|-----------|-----------|-----------|
| | | FASTED | FED | OVERALL |
| | | (N=XX) | (N=XX) | (N=xx) |
| # of 300 mg Tablets Received | | | | |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


Table 14.3.4.2C

Summary of Niraparib Dose by Cycle (Safety Population in the Extension Phase)

| Cycle | Starting<br>Niraparib<br>Dose (mg) | Statistic | Niraparib<br>TABLET | Niraparib<br>CAPSULE | Niraparib<br>OVERALL |
|---|---|---|---|---|---|
| 1 | 300<br>200<br>100 | N<br>n (%)<br>n (%)<br>n (%) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| 2 | 300<br>200<br>100 | N<br>n (%)<br>n (%)<br>n (%) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| 3 | 300<br>200<br>100 | N<br>n (%)<br>n (%)<br>n (%) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xxx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| • | | | | | |

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

TESARO Inc. Confidential Page 1 of x Protocol No: XXXXX

#### Table 14.3.4.3.1C

Summary and Change from Baseline of Select Hematology Parameters by Visit During the Extension Phase (Safety Population in the Extension Phase)

| | | | NIRAPARIB TABLE | T (N=xx) | NIRAPARIB CAPSU | LE (N=xx) | NIRAPARIB OVERA | LL (N=xx) |
|---|---|---|---|---|---|---|---|---|
| arameter | Visit | Statistic | Actual | Change | Actual | Change | Actual | Change |
| arameter | Baseline | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | |
| | Cycle 1<br>- Day 8 | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| | Cycle 1<br>- Day 15 | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| | Cycle 1<br>- Day 22 | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| | Cycle 2<br>- Day 1 | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| | | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |
| | EOT | n (missing) Mean (SD) Median Q1, Q3 Min, Max | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx | xx (xx)<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx, xx |

Source: Listing XXXXXXXXX, Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxxxrtf. Generated on DDMMMYYYY:HH:MM:St Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


Table 14.3.4.3.2C

Shift Summary of Select Hematology Parameters During the Extension Phase (Safety Population in the Extension Phase)

| Treatment Group Post-Baseline Maximum CTCAE Grade | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Niraparib | Laboratory | Baseline | Statistic | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Missing |
| Tablet | Test | CTCAE Grade | | | | | | | |
| | xxxxx | Grade 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Grade 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Grade 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Grade 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Grade 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Missing | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xxxxx | | | | | | | | |

Source: Listing XXXXXXXXX, Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

Include Tablet, Capsule and Overall

#### Repeat for:

Table 14.3.4.4.1C Summary and Change from Baseline of Select Chemistry Parameters by Visit During the Extension Phase (Safety Population in the Extension Phase)

Table 14.3.4.4.2C Shift Summary of Select Chemistry Parameters in Maximum Toxicity Grade During the Extension Phase (Safety Population in the Extension Phase)

Table 14.3.4.4.1D


Summary of COVID-19 Assessments for Patients with Suspected, Probable or Confirmed COVID-19 Case Diagnosis (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB TABLET | NIRAPARIB TABLET |
|-------------------------------|------------------|------------------|
| | FASTED | FED |
| Assessment | (N=XX) | (N=XX) |
| COVID-19 Case Diagnosis [1] | xx (xx.x%) | xx (xx.x%) |
| Confirmed | xx (xx.x%) | xx (xx.x%) |
| Probable | xx (xx.x%) | xx (xx.x%) |
| Suspected | xx (xx.x%) | xx (xx.x%) |
| COVID-19 Test Performed [2] | | |
| n | XX | xx |
| No | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Yes | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Result from the COVID-19 Test | | |
| n | XX | XX |
| Negative | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Positive | xx/xx (xx.x%) | xx/xx (xx.x%) |
| Indeterminate | xx/xx (xx.x%) | xx/xx (xx.x%) |

<sup>[1]</sup> COVID-19 Case Diagnosis is based on WHO Definition as of DDMMMYYYY.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


<sup>[2]</sup> COVID-19 Test Performed is only captured for patients with a COVID-19 Case Diagnosis.


Table 14.4.1C

Summary of Important Protocol Deviations (Safety Population in the Extension Phase)

| | NIRAPARIB | NIRAPARIB | |
|-----------------------------------|-----------|-----------|-----------|
| | TABLET | CAPSULE | TOTAL |
| Category/Coded Term | (N=XX) | (N=XX) | (N=XX) |
| Any important protocol deviations | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| CATEGORY 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| SUBCATEGORY 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| SUBCATEGORY 2 | xx (xx%) | xx (xx%) | xx (xx%) |
| CATEGORY 2 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| SUBCATEGORY 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| SUBCATEGORY 2 | xx (xx%) | xx (xx%) | xx (xx%) |
| | | • | • |

#### [Programming Notes]:

- Include only IMPORTANT protocol deviations.
- <Category 1...> represents ADDV.DVCAT. <Subcategory 1...> represents ADDV.DVDECOD.
- Sort Categories in descending order according to overall counts, if ties are present, present alphabetically.

Table 14.4.1D

Summary of Important Protocol Deviations for the PK Phase Occurring Through End of Treatment (Safety Population in the Stage 3 PK Phase)

| | NIRAPARIB TABLET | NIRAPARIB TABLET | |
|---|---|---|---|
| | FASTED [1] | FED [2] | TOTAL [3] |
| Category/Coded Term | (N=XX) | (N=XX) | (N=XX) |
| Any important protocol deviations | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| CATEGORY 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| SUBCATEGORY 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| SUBCATEGORY 2 | xx (xx%) | xx (xx%) | xx (xx%) |
| CATEGORY 2 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| SUBCATEGORY 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| SUBCATEGORY 2 | xx (xx%) | xx (xx%) | xx (xx%) |

- [1] Includes protocol deviations with onset date in Period 1 or Period 2 where patient received niraparib tablet in fasted state.
- [2] Includes protocol deviations with onset date in Period 1 or Period 2 where patient received niraparib tablet in fed state.
- [3] Includes protocol deviations occurring at any time during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]:


- Include only IMPORTANT protocol deviations.
- <Category 1...> represents ADDV.DVCAT. <Subcategory 1...> represents ADDV.DVDECOD.
- Sort Categories in descending order according to overall counts, if ties are present, present alphabetically.


# **LISTINGS**

### General guidelines:

Listings are separated for the PK Phase (Stage 1, Stage 2 and Stage 3 separately) and the Open)-Label Extension Phase.

#### For the PK Phase:

- Treatment=Sequence (for Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET; for Stage 3: NIRAPARIB TABLET FASTED/FED or NIRAPARIB TABLET FED/FASTED).
- Population=Safety Population in the PK Phase (i.e., those who receive at least 1 dose), unless otherwise specified.
- Include all data assessments relative to the PK Phase.
  - o For patients who do not continue to the Extension Phase, include all EOT/Safety FU data. Also include Extension Phase Screening for those patients who DO not proceed to the Extension Phase.
- Relative day: With respect to first date of dosing in PK period.

### For the Extension Phase:

- Treatment=Niraparib Tablet; Niraparib Capsule.
- Population=Safety Population in the Open-Label Extension Phase (i.e., those who receive at least 1 dose), unless otherwise specified.
- Include all assessments relative to the Extension Phase.
  - o Any assessment specific to Extension Phase, including Screening Data.
- Relative day: With respect to first date of dosing in Extension Phase.


Listing 16.2.1A

Disposition for PK Phase (All Patients Enrolled in the Stage 1 PK Phase)

Treatment: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| Patient | Date of Last | Date of | Reason for | Date of | Reason for | Date of | Date of | Protocol |
|---|---|---|---|---|---|---|---|---|
| Number | Niraparib Dose | Discontinuation | Discontinuation | Discontinuation | Discontinuation | Death | Progression | Version |
| | During PK Phase | From PK Phase | from PK Phase | from Study (Rel | from Study | (Rel | (Rel Day) | |
| | (Rel Day) | (Rel Day) | | Day) | | Day) | | |
| | | | Other: specify | | | | | |
| | | | Completion | | | | | |

Relative Day calculated relative to first dose in PK Phase.

Only study discontinuations, disease progressions and deaths that occur during PK phase (i.e., before 1st dose of extension or prior to discontinuing the study for patients not entering the Extension Phase) are listed.

#### [Programming Notes - PK Phase]

• Include only data that falls before first-dose Open-Label Extension Phase, i.e., for those patients who DC study and do not continue in the Open-Label Extension Phase.

#### Repeat for:

Listing 16.2.1B Disposition for PK Phase (Safety Population in the Stage 2 PK Phase)

Listing 16.2.1C Disposition for Open-Label Extension Phase (All Patients Enrolled for the Extension Phase)

Listing 16.2.1D Disposition for PK Phase (Safety Population in the Stage 3 PK Phase)

[Programming Notes - Extension Phase]

- Change 'PK Phase' to 'Open-Label Extension' Phase in respective columns.
- Treatment: Niraparib Tablet or Niraparib Capsule.
- Footnote: Relative Day calculated relative to first dose in Extension Phase.


| TESARO Inc. Protocol No: XXXXX | | Confidential | Page 1 of x |
|---|---|---|---|
| FIOCOCOI NO. AAAAA | | | |
| | Reasons for Screen Fa | ailure (Patients who Failed Screening in the Stage 1 PK Phase) | |
| Treatment Sequence: <s0< th=""><th>CREEN FAILURE&gt;</th><th></th><th></th></s0<> | CREEN FAILURE> | | |
| Patient | | | |
| Number | Protocol Version | Inclusion/Exclusion Criteria Not Met | |
| xxxxxx-xxxx | Version 1.0 (original) | INPXX: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | |
| | • | | |
| xxxxxx-xxxx | Version 1.0 (original) | EXPXX: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | |
| <u> </u> | XXXXXXXXXXXXXX Output: MMMYYYY, Data Cutoff Dat | xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS | |

#### Repeat for:

Listing 16.2.1.2B Reasons for Screen Failure (Patients who Failed Screening in the Stage 2 PK Phase)

Listing 16.2.1.2D Reasons for Screen Failure (Patients who Failed Screening in the Stage 3 PK Phase)

| TESARO Inc. | TESARO Inc. Confidential | | | |
|---|---|---|---|---|
| Protocol No: | Protocol No: XXXXX Listing 16.2.2A Protocol Deviations for the PK Phase (Safety Population in the Stage 1 PK Phase) | | | |
| Treatment: < | Stage 1 & 2 | : TABLET/CAPSULE or CAPSULE/TABLET> | | |
| Patient<br>Number | Visit | Protocol Deviation Category | Protocol Deviation Severity | Description of Protocol Deviation |
| Source: Progr | am: XXXXXX | XXXXXXXXXXXXX Output: xxxxxxxxxxx.rtf. | Generated on DDMMMYYYY:HH:MM:S | 3 |

#### [Programming Notes]

• Include only data that falls before first-dose Open-Label Extension Phase (i.e., for those patients who DC study and do not continue in the Open-Label Extension Phase)

#### Repeat for:

Listing 16.2.2B Protocol Deviation for the PK Phase (Safety Population in the Stage 2 PK Phase)


Listing 16.2.2C

Important Protocol Deviations for the Open-Label Extension Phase (Safety Population for Open-Label Extension Phase)

Treatment: <Extension (Stages 1 & 2): NIRAPARIB TABLET or NIRAPARIB CAPSULE; Extension (Stage 3): NIRAPARIB TABLET>

| Patient | | Protocol Deviation | Protocol Deviation | Description of | TESARO | GSK |
|---|---|---|---|---|---|---|
| | | | | <u> </u> | | |
| Number | Visit | Category | Severity | Protocol Deviation | Classification [1] | Classification [2] |
| | | | | | < <significant <="" td=""><td>&lt;<important non-<="" td=""></important></td></significant> | < <important non-<="" td=""></important> |
| | | | | | IMPORTANT>> | IMPORTANT>> |

<sup>[1]</sup> For Stages 1 & 2, protocol deviation classification is done based on TESARO Protocol Deviation Management System only. GSK Classification will remain blank.

#### [Programming notes]

For Stage 3 Extension Phase, patients will receive NIRAPARIB TABLET formulation only.

For Stages 1 and 2 reporting, only TESARO Classifications will be populated, for Stage 3 - only GSK Classification will be populated.

Only include protocol deviation classed as Important.


<sup>[2]</sup> For Stage 3, protocol deviation classification is done based on GSK Protocol Deviation Management System only. TESARO Classification will remain blank.

|---|---|---|---|---|---|
| Importa | ant Protoco | l Deviations for the PK Phase | Listing 16.2.2.1D Occurring Through End of Trea | tment (Safety Population for Stage 3 PK | Phase) |
| Treatment: < | NIRAPARIB | FASTED or NIRAPARIB FED> | | | |
| Patient<br>Number | Visit | Protocol Deviation Category | Protocol Deviation Severity | Description of Protocol Deviation | |
| | • | XXXXXXXXXXXXXXX Output: xxxxx<br>MMMYYYY, Data Cutoff Date: D | | MMMYYYY:HH:MM:SS | |

### [Programming notes]:

• Only include protocol deviation classed as Important.


Listing 16.2.2.2D

GSK Protocol Deviations related to COVID-19 (Safety Population for Stage 3 PK Phase)

Treatment: <NIRAPARIB FASTED or NIRAPARIB FED>

| Patient | | | | |
|---|---|---|---|---|
| Number | Deviation Category | Description of Deviation | GSK Classification | Date |
| | | | <pre><important not-important=""></important></pre> | |

Note: \* Patients with probable, suspected or confirmed COVID-19. Note: This listing only includes COVID-19 related protocol deviations.

Source: Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


| TESARO Inc. | | Confidential | Pa | age 1 of x |
|---|---|---|---|---|
| | | Listing 16.2.3A | | |
| | Study Populations for the F | PK Phase (All Patients Enrolled in the Sta | age 1 PK Phase) | |
| Treatment: <t< td=""><td>ABLET/CAPSULE or CAPSULE/TABLET or SCRE</td><td>EN FAILURE&gt;</td><td></td><td></td></t<> | ABLET/CAPSULE or CAPSULE/TABLET or SCRE | EN FAILURE> | | |
| Patient | PK Phase Safety | Informed Consent Date | Randomization Date | |
| Number | (SAF) Population | | | |
| | Y | | | |
| _ | am: XXXXXXXXXXXXXXXXXX Output: xxxxx<br>Date: DDMMMYYYY, Data Cutoff Date: D | xxxxxxx.rtf. Generated on DDMMMYYYY:HH:M | M:SS | |

### Repeat for:

Listing 16.2.3B Study Populations for the PK Phase (All Patients Screened in the Stage 2 PK Phase)

ullet For Stage 2 PK, add column for BE Evaluable Population (Y/N).

| TESARO Inc. | | | Confidential | | | | <br>Page 1 o | fх |
|---|---|---|---|---|---|---|---|---|
| Protocol No: XXXXX | | т | isting 16.2.3C | | | | | |
| St | udy Populations for the | Open-Label Extens | ion Phase (All Patients | s Enrolled in the Ex | tension Phas | se) | | |
| Treatment: <nirapar< td=""><td>RIB TABLET or NIRAPARIB</td><td>CAPSULE&gt;</td><td></td><td></td><td></td><td></td><td></td><td></td></nirapar<> | RIB TABLET or NIRAPARIB | CAPSULE> | | | | | | |
| | Extension Phase | | | | | | | |
| Patient | Safety (SAF) | | | | | | | |
| Number | Population | | | | | | | |
| | Y | | | | | | | |
| Source: Program: > | XXXXXXXXXXXXXXXXXX Out | put: xxxxxxxxxxx. | rtf. Generated on DDMN | MMYYYY:HH:MM:SS | | | | |
| Data Extract Date: | DDMMMYYYY, Data Cutof | f Date: DDMMMYYYY | | | | | | |


|---|---|---|---|---|
| | | Listing 16.2.3 | | |
| | Study Populations | for the PK Phase (All Patients | Enrolled in the Stage 3 PK Ph | ase) |
| Treatment: <f< td=""><td>ASTED/FED or FED/FASTED or SCR</td><td>EEN FAILURE&gt;</td><td></td><td></td></f<> | ASTED/FED or FED/FASTED or SCR | EEN FAILURE> | | |
| Patient | PK Phase | FE Population | Informed Consent Date | Randomization Date |
| Number | Safety (SAF) Population | | | |
| | Y | Y | | |
| | | N | | |

Source: Program: XXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY


#### Listing 16.2.4.1A

Demographics (Safety Population in the Stage 1 PK Phase)

Study Treatment: <Stage 1 & 2: NOT DOSED or TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: NOT DOSED or FASTED/FED or FED/FASTED> or

<Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| /EXCEILS I | OII. NIINAI | . AIVID IA | DLEI OI NIKAFAKI | D CALOUDE, | as applicable | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Patient | Age | Sex | Child-Bearing | Ethnicity | Race | Height | Weight | BMI | ECOG Performance |
| Number | (yrs) | | Potential | | | (cm) | (kg) | (kg/m²) | Status |
| | | | | | Other: specify | | | | |

ECOG = Eastern Cooperative Oncology Group: 0=Fully active, able to carry on all pre-disease performance without restriction 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature 2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair

#### Repeat for:

Listing 16.2.4.1B Demographics (Safety Population in the Stage 2 PK Phase)

Listing 16.2.4.1C Demographics (Safety Population in the Extension Phase)

Listing 16.2.4.1D Demographics (Safety Population in the Stage 3 PK Phase)


Listing 16.2.4.2A

Medical History (Safety Population in the Stage 1 PK Phase)

PK Phase Treatment: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| | System Organ Class | | | |
|---------|----------------------------|-------|--------------|-----------|
| Patient | Preferred Term | Start | Ongoing at | |
| Number | Medical Condition or Event | Date | Study Start? | Stop Date |

Includes only patients with major medical conditions.

Note: MedDRA version XX.X.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Listing 16.2.4.2B Medical History (Safety Population in the Stage 2 PK Phase)

Listing 16.2.4.2C Medical History (Safety Population in the Extension Phase)

Listing 16.2.4.2D Medical History (Safety Population in the Stage 3 PK Phase)

#### [Programming notes]

• For Stage 3, the latest available MedDRA version is to be used.


Listing 16.2.4.3A

Prior Anti-Cancer Treatment (Safety Population in the Stage 1 PK Phase)

Treatment: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| Patient | Regimen | -Verbatim Term | | |
|---|---|---|---|---|
| Number | Number | Preferred Term | Reason for Administration | Best Response |
| | | | Other: specify | |

#### Repeat for:

Listing 16.2.4.3B Prior Anti-Cancer Treatment (Safety Population in the Stage 2 PK Phase)

Listing 16.2.4.3C Prior Anti-Cancer Treatment (Safety Population in the Extension Phase)

Listing 16.2.4.3D Prior Anti-Cancer Treatment (Safety Population in the Stage 3 PK Phase)


Listing 16.2.4.4A

Primary Cancer History (Safety Population in the Stage 1 PK Phase)

Treatment: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| Patient | | Date of First | | Number of Prior Lines |
|---|---|---|---|---|
| Number | Tumor Type | Diagnosis | Cancer Stage (Most Recent) | of Therapy |
| | <pre><other: specify=""></other:></pre> | | | |

#### Repeat for:

Listing 16.2.4.4B Primary Cancer History (Safety Population in the Stage 2 PK Phase)

Listing 16.2.4.4C Primary Cancer History (Safety Population in the Extension Phase)

Listing 16.2.4.4D Primary Cancer History (Safety Population in the Stage 3 PK Phase)


#### Listing 16.2.4.5A

Prior/Concomitant Radiotherapy (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| TADDET OF MITCHINED C. | mbodd, as appricable | | | | |
|---|---|---|---|---|---|
| Patient | | | | | Prior/ |
| Number | Site or Region | Date Started | Date Stopped | Total Grays | Concomitant Flag |

Note: Includes patients with prior or concomitant radiotherapy with respect to the PK Phase.

P=Prior (radiotherapy with start date earlier than the first dose date of study treatment)

C=Concomitant (radiotherapy occurring on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase).

Source: Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxrtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Listing 16.2.4.5B Prior/Concomitant Radiotherapy (Safety Population in the Stage 2 PK Phase)

Listing 16.2.4.5C Prior/Concomitant Radiotherapy (Safety Population in the Extension Phase)

Listing 16.2.4.5D Prior/Concomitant Radiotherapy (Safety Population in the Stage 3 PK Phase)


Listing 16.2.5.1A

Prior and Concomitant Medications (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

Patient Number = xxxxxx-xxxx

| ATC/<br>Preferred<br>Term/<br>Verbatim | Dogo por | Dogo | Eroguana | Indica | Route of<br>Administr | Start/ | | Prior/<br>Concomitant | | |
|---|---|---|---|---|---|---|---|---|---|---|
| verbatim | Dose per | Dose | Frequenc | Indica | Administr | Start/ | | Concomitant | | |
| Term | Administration | Unit | У | tion | ation | Stop Date | Ongoing | Flag | PK Dose 1 | PK Dose 2 |
| | | | | | | | | | YYYY-MM-DD | YYYY-MM-DD |

Note: Includes patients with prior or concomitant medications taken during the PK Phase. P=Prior medication only; C=Concomitant medication only; B=Both prior and concomitant medications.

Source: Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

- For the Prior/Concomitant Flag, list all that apply.
- If ATC3 not available, use a footnote [1] ATC level 3 term is not available through WHO Drug Dictionary.

#### Repeat for:

Listing 16.2.5.1B Prior and Concomitant Medications (Safety Population in the Stage 2 PK Phase)

Listing 16.2.5.1C Prior and Concomitant Medications (Safety Population in the Extension Phase)

Listing 16.2.5.1D Prior and Concomitant Medications (Safety Population in the Stage 3 PK Phase)


Listing 16.2.5.2A

Prior/Concomitant Procedures During PK Phase (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| Patient | Procedure | Rel Day | | | | | Prior/Concomitant |
|---|---|---|---|---|---|---|---|
| Number | Date | [1] | Procedure | Results/Findings | AE/SAE? | Indication | Flag |
| XXXXX-XXXX | | | | | | | |

[1] Relative to first dose during the PK Phase.

Note: Includes patients with prior or concomitant procedures during the PK Phase.

P=Prior (any procedure earlier than the first dose date of study treatment).

C=Concomitant (any procedure on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase).

Source: Program: XXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for

Listing 16.2.5.2B Prior/Concomitant Procedures During the PK Phase (Safety Population in the Stage 2 PK Phase)

Listing 16.2.5.2C Prior/Concomitant Procedures During the Extension Phase (Safety Population in the Extension Phase)

[Programming Notes for Extension Phase]

• Footnote: [1] Relative to first dose during the Extension Phase.

Listing 16.2.5.2D Prior/Concomitant Procedures During the PK Phase (Safety Population in the Stage 3 PK Phase)


Listing 16.2.5.3A

Prior and Concomitant Transfusions (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| | Received Transfusion | | | | | |
|---|---|---|---|---|---|---|
| Patient | within 14 days of first | Type of | | | | Prior/ |
| Number | dose or during study? | Administration | Units | Transfusion Date | Rel Day [1] | Concomitant Flag |
| | | Other: specify | | | | |

[1] Relative to first dose during the PK Phase.

Note: Includes patients with prior or concomitant transfusions during the PK Phase.

P=Prior (any transfusion earlier than the first dose date of study treatment).

C=Concomitant (any transfusion on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase).

#### [Programming Notes]

• For the Prior/Concomitant Flag, list all that apply.

#### Repeat for:

Listing 16.2.5.3B Prior and Concomitant Transfusions (Safety Population in the Stage 2 PK Phase)

Listing 16.2.5.3C Prior and Concomitant Transfusions (Safety Population in the Extension Phase)

Listing 16.2.5.3D Prior and Concomitant Transfusions (Safety Population in the Stage 3 PK Phase)


#### Listing 16.2.5.4A

Prior and Concomitant Growth Factors (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| Patient | Received growth factor within 14 | Type of | | | Administration | Prior/ |
|---|---|---|---|---|---|---|
| Number | days of first dose or during study? | Administration | Dose | Unit | Date | Concomitant Flag |
| | | Other: specify | | Other: specify | | |

Note: Includes patients with prior or concomitant growth factors during the PK Phase.

P=Prior (any growth factor earlier than the first dose date of study treatment).

C=Concomitant (any growth factor given on or after the initial study treatment dosing date through either the first dose of the Extension Phase or through 30 days after the last dose, for those not continuing into the Extension Phase).

Source: Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxrtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]

• For the Prior/Concomitant Flag, list all that apply.

#### Repeat for:

Listing 16.2.5.4B Prior and Concomitant Growth Factors (Safety Population in the Stage 2 PK Phase)

Listing 16.2.5.4C Prior and Concomitant Growth Factors (Safety Population in the Extension Phase)

Listing 16.2.5.4D Prior and Concomitant Growth Factors (Safety Population in the Stage 3 PK Phase)

TESARO Inc. Confidential Page 1 of x Protocol No: XXXXX

Listing 16.2.5.5A

Study Treatment (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET>

| | | | | | | | | | Vomit |
|---|---|---|---|---|---|---|---|---|---|
| | | | Date:Time of | Full | If No, how | | | Fast 8 hrs | within 8 |
| Patient | | | Administration | Dose | much | Reason | Bottle | prior to | hours of |
| Number | Visit | Formulation | (Rel Day [1]) | Taken? | consumed? | for Change | Number | administration? | dose? |

[1] Relative to first dose during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxxrtf. Generated on DDMMMYYYY: HH: MM: SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Listing 16.2.5.5B Study Treatment (Safety Population in the Stage 2 PK Phase)

[For Stage 2 PK Phase]

- Modify label for Vomiting Question, 'Vomit within specified time of dose'.
- Add column for Nausea Question, 'Nausea within specified time of dose'.

| TESARO Inc. Confidential Pa | age 1 | of | Ē | Х | 7 |
|-----------------------------|-------|----|---|---|---|
|-----------------------------|-------|----|---|---|---|


Listing 16.2.5.5C

Study Treatment (Safety Population in the Extension Phase)

TREATMENT: <NIRAPARIB TABLET or NIRAPARIB CAPSULE>

| 11(111111111111111111111111111111111111 | ALLEMAN AND A | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Patient<br>Number | Visit | Dose<br>Prescribed<br>(mg) | Start Date<br>(Rel Day [1])/<br>Stop Date (Rel<br>Day [1]) | Was Full<br>Dose<br>Taken? | Action Taken | Reason for<br>Modification | Bottle<br>number<br>Dispensed | Bottle<br>Number<br>Returned | Tablets<br>Remaining |
| | | | | No | | Other <specify reason=""></specify> | | | |

[1] Relative to first dose during the Extension Phase.

Source: Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

TESARO Inc. Confidential Page 1 of x Protocol No: XXXXX

Listing 16.2.5.5D

Study Treatment (Safety Population in the Stage 3 PK Phase)

Treatment Sequence: <FASTED/FED or <FED/FASTED>

| Patient<br>Number | Visit | Fasted or<br>Fed State | Date:Time of Administration (Rel Day [1]) | Bottle Number | Fast 10 hrs prior to administration? | Vomit within protocol specified hours from dose? | Fast for minimum of 4 hours post dose? |
|---|---|---|---|---|---|---|---|

[1] Relative to first dose during the PK Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

| TESARO Inc<br>Protocol N | | Confide | ential | Page 1 of x |
|---|---|---|---|---|
| Listing 16.2.5.6B Subsequent Anti-Cancer Therapy (Safety Population in the Stage 2 PK Phase) | | | | |
| Treatment | Sequence: TABLET/CAPSULE or CAPS | SULE/TABLET | | |
| Patient<br>Number | Date of Subsequent Anti-Cancer<br>Administration | Relative Day [1] | | |
| | ve to first dose during the PK Ph<br>udes only patients with subsequer | | orded for patients who do not continue to Extens | sion Phase. |
| | ogram: XXXXXXXXXXXXXXXXXX. Outp<br>ct Date: DDMMMYYYY, Data Cutoff | | nerated on DDMMMYYYY:HH:MM:SS | |

| TESARO Inc<br>Protocol No | | Confide | ential | Page 1 of x |
|---|---|---|---|---|
| 11000001 1. | | Listing 16<br>ti-Cancer Therapy (Safety | .2.5.6C Population in the Extension Phase) | |
| Treatment: | <pre><niraparib niraparib<="" or="" pre="" tablet=""></niraparib></pre> | CAPSULE> | | |
| Patient<br>Number | Date of Subsequent Anti-Cancer<br>Administration | Relative Day [1] | | |
| | ve to first dose during the Extenudes only patients with subsequen | | orded. | |
| | ogram: XXXXXXXXXXXXXXXXXX. Outp<br>ct Date: DDMMMYYYY, Data Cutoff | | nerated on DDMMMYYYY:HH:MM:SS | |

| TESARO Inc.<br>Protocol No: | VVVVV | | Confidential | | Page 1 of x |
|---|---|---|---|---|---|
| PIOCOCOI NO: | Listing 16.2.5.6D<br>Meal Status (Safety Population in the Stage 3 PK Phase) | | | | |
| Treatment Seq | uence: <fasted fed<="" th=""><th>or <fed fasted=""></fed></th><th></th><th></th><th></th></fasted> | or <fed fasted=""></fed> | | | |
| Patient<br>Number | Visit | Meal Start Date | Meal Start Time | Meal End Time | % of Meal Consumed |
| _ | | XXXX. Output: xxxxxxxxxxxx.<br>Data Cutoff Date: DDMMMYYYY | | YYYY:HH:MM:SS | |


| TESARO Inc | | | | Confidential | | Page 1 of x |
|---|---|---|---|---|---|---|
| Listing 16.2.6.1C<br>Investigator Assessment of Response (Safety Population in the Extension Phase) | | | | | | |
| TREATMENT: | <nirapari< td=""><td>B TABLET or N</td><td>IRAPARIB CAPSU</td><td>LE&gt;</td><td></td><td></td><td></td><td></td><td></td></nirapari<> | B TABLET or N | IRAPARIB CAPSU | LE> | | |
| Patient<br>Number | Visit | Date | Date Rel Day [1] Overall Response | | | |
| | | | | NE: <reason></reason> | | |
| | [1] Relative to first dose during the Extension Phase. Source: Program: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | |
| | _ | | ta Cutoff Date | | - | |


#### Listing 16.2.7.1A

Adverse Events (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| | | | Start Date:Time | | | | Action | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Dosing Period/ | Adverse Event | (Rel Day [1]) | | SAE/ | | Taken on | Other | | |
| Patient | Niraparib | MedDRA Preferred Term | End Date (Rel | | Reason | | Study | Action | Relation- | |
| Number | Treatment | System Organ Class | Day [1]) | TEAE? | [2] | Severity | Treatment | Taken | ship | Outcome |
| | Period 1/<br>Capsule | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | yyyy-mm-dd [x] | Y | N | Grade 1 | | | | Recovered/<br>Resolved |
| | Period 2/<br>Tablet | XXXXXXXXXXXXXXX<br>[P]XXXXXXXXXXXXXXXXXX<br>[S]XXXXXXXXXXXXXXXXX | yyyy-mm-dd [x] | Y | N | Grade 1 | | | | Recovered/<br>Resolved |
| | PK Safety FU | | | | | | | | | |

- [1] Relative to the date of first dose in PK Phase.
- [2] Reason for SAE: 1 = Result in death; 2 = Life threatening; 3 = Result in persistent or significant disability/incapacity;
- 4 = Requires or prolongs hospitalization; 5 = Congenital abnormality/birth defect; 6 = Other medically important event.

Source: Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Listing 16.2.7.1B Adverse Events (Safety Population in the Stage 2 PK Phase)

#### [Add time for start date]

Listing 16.2.7.1C Adverse Events (Safety Population in the Extension Phase)

Listing 16.2.7.1D Adverse Events (Safety Population in the Stage 3 PK Phase)

#### [Programming Notes]

- Stage 3: Treatment Sequence will be Fasted/Fed and Fed/Fasted.
- Stage 3: Column 2: Dosing Period/Treatment Treatment should be Niraparib FASTED or Niraparib FED.
- Extension Phase: Do not need column for Dosing Period/Treatment.
- Extension Phase: Do not need time with start/stop dates.
- Extension Phase: Footnote: [1] Relative to first dose during the Extension Phase.
- $\bullet$  Extension Phase: Add column for Dose at Onset of AE.


#### Listing 16.2.8.1.1A

Hematology Results in the PK Phase (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| Patient<br>Number | Parameter (unit) | Visit | Rel Day | Sample<br>date/time | Result | Change from baseline | Normal range | Out of range flag | Clinically significant flag |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | XX.X | XX.X | xx.x - xx.x | | |

[1] Relative to the date of first dose in the PK Phase.

Scheduled and unscheduled visits through the extension screening phase or through study discontinuation for those not continuing in the Extension Phase, are included. Visits related to the extension screening phase are not included.

Source: Program: XXXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### [Programming Notes]:

• If required for readability, move 'Patient Number' into Header row after 'Treatment Sequence'.

#### Repeat for:

Listing 16.2.8.1.1B Hematology Results (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.1.1C Hematology Results (Safety Population in the Extension Phase)

Listing 16.2.8.1.1D Hematology Results Through the PK End of Treatment Visit (Safety Population in the Stage 3 PK Phase)

Listing 16.2.8.1.2A Chemistry Results (Safety Population in the Stage 1 PK Phase)

Listing 16.2.8.1.2B Chemistry Results (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.1.2C Chemistry Results (Safety Population in the Extension Phase)

Listing 16.2.8.1.2D Chemistry Results Through the PK End of Treatment Visit (Safety Population in the Stage 3 PK Phase)

Listing 16.2.8.1.3A Urinalysis Results (Safety Population in the Stage 1 PK Phase)

Listing 16.2.8.1.3B Urinalysis Results (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.1.3C Urinalysis Results (Safety Population in the Extension Phase)

[Programming Notes For Extension Phase Tables]:

• Footnote: [1] Relative to first dose during the Extension Phase.

Listing 16.2.8.1.3D Urinalysis Results Through the PK End of Treatment Visit (Safety Population in the Stage 3 PK Phase)

| TESARO Inc. | | |
|-------------|--------------|-------------|
| | Confidential | Page 1 of x |


Listing 16.2.8.1.4C

Liver Function Tests - Potential Hy's Law Cases (Safety Population in the Extension Phase)

TREATMENT: <NIRAPARIB TABLET or NIRAPARIB CAPSULE>

| | | | | Laboratory Analyte (result/xULN) | | | |
|---|---|---|---|---|---|---|---|
| Patient<br>Number | Visit | Sample<br>Collection Date | Day [1] | ALT (U/L) | AST (U/L) | Total Bilirubin (umol/L) | ALP (U/L) |
| | | DDMMMYYYY | | 150/3.3 | 100/2.7 | 40/2.3 | 100/0.7 |

ALP=alkaline phosphatase. ALT=alanine aminotransferase. AST=aspartate aminotransferase. ULN=upper limit of normal.

[1] Relative to first dose during the Extension Phase.

Source: Program: XXXXXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

[Programming Notes]

Include all visits for any Patients with ALT or AST >3×ULN with bilirubin >2×ULN and ALP <2×ULN at any time in Extension Phase.


Listing 16.2.8.2A

Vital Signs (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| Patient<br>Number | Visit | Assessment<br>Date | Rel<br>Day<br>[1] | Height (cm) | Weight (kg) | Temperature (°C) | Pulse (beats/min) | Systolic Blood<br>Pressure (mmHg) | Diastolic Blood<br>Pressure (mmHg) |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | · | | | |

[1] Relative to the date of first dose in the PK Phase. Data is listed only when the vital sign assessment was performed.

Source: Program: XXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Listing 16.2.8.2B Vital Signs (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.2C Vital Signs (Safety Population in the Extension Phase)

[Programming Notes For Extension Phase Tables]:

• Footnote: [1] Relative to first dose during the Extension Phase

Listing 16.2.8.2D Vital Signs Through the PK End of Treatment Visit (Safety Population in the Stage 3 PK Phase)

| TESARO Inc.<br>Protocol No: XX | vvv | | | Confidential | Page 1 of x |
|---|---|---|---|---|---|
| FIOCOCOI NO. AA | AAA | | | Listing 16.2.8.3A | |
| | | | ECG Results (Safety | Population in the Stage 1 PK Phase) | |
| Treatment Seque<br>TABLET or NIRAP | | - | | E/TABLET> or <stage 3:="" fasted="" fed="" or=""> or <extension:< td=""><td>NIRAPARIB</td></extension:<></stage> | NIRAPARIB |
| Patient<br>Number | Visit | Date | Rel Day [1] | ECG Interpretation | |
| | | | dose in the PK Phase.<br>CS = Clinically Signific | eant. | |
| _ | | | XX. Output: xxxxxxxxxxx<br>ta Cutoff Date: DDMMMYY | xx.rtf. Generated on DDMMMYYYY:HH:MM:SS | |

#### Repeat for:

Listing 16.2.8.3B ECG Results (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.3C ECG Results (Safety Population in the Extension Phase)

Listing 16.2.8.3D ECG Results (Safety Population in the Stage 3 PK Phase)

[Programming Notes For Extension Phase Tables]:

• Footnote: [1] Relative to first dose during the Extension Phase

| ESARO Inc. | Confidential | Page 1 of x |
|------------|--------------|-------------|
|------------|--------------|-------------|


#### Listing 16.2.8.4A

ECOG Performance Status (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| Patient | | | | |
|---------|-------|-----------------|-------------|--------------------|
| Number | Visit | Assessment Date | Rel Day [1] | Performance Status |

[1] Relative to the date of first dose in the PK Phase. Data is listed only when the ECOG Performance Status assessment was performed. ECOG = Eastern Cooperative Oncology Group:

0=Fully active, able to carry on all pre-disease performance without restriction

1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature

2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours

3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours

4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair

Source: Program: XXXXXXXXXXXXXXXXXX. Output: xxxxxxxxxxx.rtf. Generated on DDMMMYYYYY:HH:MM:SS

Data Extract Date: DDMMMYYYY, Data Cutoff Date: DDMMMYYYY

#### Repeat for:

Listing 16.2.8.4B ECOG Performance Status (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.4C ECOG Performance Status (Safety Population in the Extension Phase)

[Programming Notes For Extension Phase Tables]:

• Footnote: [1] Relative to first dose during the Extension Phase

Listing 16.2.8.4D ECOG Performance Status Through the PK End of Treatment Visit (Safety Population in the Stage 3 PK Phase)

| TESARO Inc. Protocol No: XXXXX | | Confidential Pa | | | | |
|---|---|---|---|---|---|---|
| Protocol No: | ***** | Listing 16.2.8.5A | | | | |
| | | Baseline Physical Exam | mination Findin | gs (Safety Populati | on in the Stag | e 1 PK Phase) |
| - | | ge 1 & 2: TABLET/CAPSUI<br>ULE>, as applicable | LE or CAPSULE/TA | ABLET> or <stage 3:<="" td=""><td>FASTED/FED or</td><td>FED/FASTED&gt; or <extension: niraparib<="" td=""></extension:></td></stage> | FASTED/FED or | FED/FASTED> or <extension: niraparib<="" td=""></extension:> |
| Patient<br>Number | Visit | Date Performed | Rel<br>Day [1] | Body System | Status | Abnormality Description |
| Source: Progr | am: XXXXXX | of first dose in the F<br>XXXXXXXXXXXXXX Output:<br>MYYYY, Data Cutoff Dat | xxxxxxxxxxx.rt | f. Generated on Di | MMMYYYY:HH:MM: | ss |

#### Repeat for:

Listing 16.2.8.5B Baseline Physical Examination Findings (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.5C Baseline Physical Examination Findings (Safety Population in the Extension Phase)

Listing 16.2.8.5D Baseline Physical Examination Findings (Safety Population in the Stage 3 PK Phase)

[Programming Notes For Extension Phase Tables]:

• Footnote: [1] Relative to first dose during the Extension Phase.


Listing 16.2.8.6A

Pregnancy Test (Safety Population in the Stage 1 PK Phase)

Treatment Sequence: <Stage 1 & 2: TABLET/CAPSULE or CAPSULE/TABLET> or <Stage 3: FASTED/FED or FED/FASTED> or <Extension: NIRAPARIB TABLET or NIRAPARIB CAPSULE>, as applicable

| Patient | | Was | | | | |
|---|---|---|---|---|---|---|
| Number | Visit | Pregnancy Test Performed? | Date of Test | Rel Day [1] | Туре | Result |

[1] Relative to the date of first dose in the PK Phase.

Scheduled and unscheduled visits through the Extension Screening Phase or through study discontinuation for those not continuing in the Extension Phase, are included. Visits related to the Extension Screening Phase are not included.

#### Repeat for:

Listing 16.2.8.6B Pregnancy Test (Safety Population in the Stage 2 PK Phase)

Listing 16.2.8.6C Pregnancy Test (Safety Population in the Extension Phase)

[Programming Notes For Extension Phase Tables]:

• Footnote: [1] Relative to first dose during the Extension Phase

Listing 16.2.8.6D Pregnancy Test (Safety Population in the Stage 3 PK Phase)


Listing 16.2.9.2D

Listing of COVID-19 Assessments and Symptom Assessments for Patients with COVID-19 Adverse Events (Safety Population in the Stage 3 PK Phase)

Treatment Sequence: <Stage 3: Period 1: FASTED or FED; Period 2: FASTED or FED>

| Patient<br>Number | Treatment<br>Period (State) | Adverse<br>Event | AE<br>Start Date | COVID-19 Case<br>Diagnosis [1] | COVID-19 Test Performed/ Test Date/ Results | Assessments and<br>Symptom Assessments | Result |
|---|---|---|---|---|---|---|---|
| xxxx | 1 (FASTED) | Coronavirus infection | 2020-04-16 | Suspected | Yes/<br>2020-04-17/<br>Indeterminate | Travel to Location with Community Transmission [2] | No |
| | | | | | | Visited Health Care Facility [2] | No |
| | | | | | | Contact with COVID-19<br>Confirmed/Probable Case [2] | Unknown |
| | | | | | | Medication Taken to Treat COVID-19 | Yes |
| | | | | | | Fever | Yes |
| | | | | | | Cough | Yes |
| | | | | | | Shortness of Breath | Yes |
| | | | | | | Sore Throat | No |
| | | | | | | Loss of Appetite | No |
| | | | | | | Nausea | No |
| | | | | | | Vomiting | No |
| | | | | | | Diarrhea | No |
| | | | | | | Abdominal Pain | No |
| | | | | | | Fatigue | No |
| | | | | | | Loss of Smell | No |
| | | | | | | Loss of Taste | No |
| | | | | | | Asymptomatic | No |
| | | | | | | Home Quarantined/Isolated | Unknown |
| | 2 (FED) | | | | | | |

#### AE=Adverse event.

- [1] COVID-19 Case Diagnosis is based on WHO Definition as of DDMMMYYYYY.
- [2] Within 14 days prior to symptom onset.

#### [Programming Notes]

The COVID-19 AE terms include: Asymptomatic COVID-19, Coronavirus infection, COVID-19, COVID-19 pneumonia, Suspected COVID-19. Note that the number of COVID-19 AE terms may change.